CLINICAL TRIAL: NCT02212457
Title: A Phase 2b, Randomized, Controlled, Observer-Blind, Multi-Center Study Assessing the Immunogenicity and Safety of GSK Meningococcal ABCWY Vaccine Administered at Different Schedules Compared to GSK Meningococcal Group B Vaccine, in Healthy Adolescents
Brief Title: Trial to Assess Immunogenicity and Safety of GlaxoSmithKline (GSK) Biologicals' Meningococcal ABCWY Vaccine as Compared to Meningococcal B Vaccine in Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: 205215; V102_15 (Other: Novartis); 2013-002451-15 (EudraCT Number)
Record Dates: First submitted 2014-08-06; First posted 2014-08-08 (Estimated); Results first posted 2017-07-21 (Actual); Last update posted 2019-06-27 (Actual); Status verified 2019-06

CONDITIONS: Infections, Meningococcal
MeSH Terms: conditions — Meningococcal Infections | interventions — 4CMenB vaccine; Hepatitis A Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (6):
- rMenB_0_2 Group (Experimental): Subjects received two injections of Bexsero vaccine at Visit Month 0 and Visit Month 2, Havrix vaccine at Visit Month 6 and Visit Month 12 and saline placebo at Visit Month 1.
  Interventions: Biological: Bexsero; Other: Saline Placebo; Biological: Havrix
- ABCWY_ 0_2 Group (Experimental): Subjects received MenABCWY vaccine at Visit Month 0 and Visit Month 2, Havrix vaccine at Visit Month 6 and Visit Month 12 and saline placebo at Visit Month 1.
  Interventions: Other: Saline Placebo; Biological: Havrix; Biological: MenABCWY
- ABCWY_0_1 Group (Experimental): Subjects received MenABCWY vaccine at Visit Month 0 and Visit Month 1, Havrix vaccine at Visit Month 2 and Visit Month 12 and saline placebo at Visit Month 6.
  Interventions: Other: Saline Placebo; Biological: Havrix; Biological: MenABCWY
- ABCWY_0_6 Group (Experimental): Subjects received MenABCWY vaccine at Visit Month 0 and Visit Month 6, Havrix vaccine at Visit Month 1 and Visit Month 12 and saline placebo at Visit Month 2.
  Interventions: Other: Saline Placebo; Biological: Havrix; Biological: MenABCWY
- ABCWY_0_11 Group (Experimental): Subjects received MenABCWY vaccine at Visit Month 1 and Visit Month 12, Havrix vaccine at Visit Month 0 and Visit Month 6 and saline placebo at Visit Month 2.
  Interventions: Other: Saline Placebo; Biological: Havrix; Biological: MenABCWY
- ABCWY_0_2_6 Group (Experimental): Subjects received MenABCWY vaccine at Visit Month 0, Visit Month 2 and Visit Month 6 and Havrix vaccine at Visit Month 1 and Visit Month 12.
  Interventions: Biological: Havrix; Biological: MenABCWY

INTERVENTIONS:
Biological: Bexsero — Two doses administered intramuscularly into the deltoid area at Months 0 and 2 in rMenB_0_2 Group.
  Arms: rMenB_0_2 Group
Other: Saline Placebo — One dose administered intramusculary in the deltoid muscle at Month 1 in ABCWY_ 0_2 Group and rMenB_0_2 Group, Month 2 in ABCWY_0_6 Group and ABCWY_0_11 Group and Month 6 in ABCWY_0_1 Group.
  Arms: ABCWY_ 0_2 Group; ABCWY_0_1 Group; ABCWY_0_11 Group; ABCWY_0_6 Group; rMenB_0_2 Group
Biological: Havrix — Two doses administered in the deltoid muscle at Month 2 and 12 in ABCWY_0_1 Group, Month 1 and 12 in Group ABCWY_0_6 Group and ABCWY_0_2_6 Group , Month 0 and 6 in ABCWY_0_11 Group and Month 6 and 12 in ABCWY_ 0_2 Group and rMenB_0_2 Group.
Biological: MenABCWY — Two to three doses administered in the deltoid muscle at Month 0 and 1 in ABCWY_0_1 Group, Month 0 and 6 in ABCWY_0_6 Group, Month 1 and 12 in ABCWY_0_11 Group, Month 0, 2 and 6 in ABCWY_0_2_6 Group, Month 0 and 2 in ABCWY_ 0_2 Group and rMenB_0_2 Group.
  Arms: ABCWY_ 0_2 Group; ABCWY_0_1 Group; ABCWY_0_11 Group; ABCWY_0_2_6 Group; ABCWY_0_6 Group

SUMMARY:
The main purposes for conducting the study are firstly to assess immunological non-inferiority of the MenABCWY vaccine, administered according to 0, 2 month schedule to healthy adolescents 10 to 18 years of age, to those of the licensed rMenB+OMV vaccine (Bexsero™) in terms of hSBA GMTs at one month after the second vaccination, secondly to give the flexibility for the national vaccination program by showing the safety and immunogenicity of MenABCWY administrated according to four different vaccination schedules and additionally to evaluate a potential benefit of the 3-dose vaccination series.

ELIGIBILITY:
Inclusion Criteria:

1. Adolecents from 10-18 yearsof age, generally in good health, and available for all study visits, and who/whose legally acceptable representative has given written informed consent at the time of enrollment.
2. Individuals of who the investigator believes can and will comply with the requirements of the protocol (e.g. use of an eDiary, return for follow-up visits, available for phone contacts).
3. Female subjects of childbearing potential must have a negative urine preganancy test.

Exclusion Criteria:

1. Serious, acute, or chronic illness. Previous or suspected disease caused by N. meningitidis. Previous immunization with any menincococcal or Hepatitis A vaccines.
2. Exposure to individuals with clicically proven meningococcal disease or clinical bacterial meningitis without further microbiologic characteriszation.

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1063 (Actual)
Dates: Start 2014-08-21 (Actual); Primary Completion 2015-05-22 (Actual); Study Completion 2016-03-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (30):
- United States (13):
  - GSK Investigational Site, Jonesboro, Arkansas
  - GSK Investigational Site, Hialeah, Florida
  - GSK Investigational Site, Melbourne, Florida
  - GSK Investigational Site, Augusta, Kansas
  - GSK Investigational Site, Niles, Michigan
  - GSK Investigational Site, Saint Paul, Minnesota
  - GSK Investigational Site, Bellevue, Nebraska
  - GSK Investigational Site, Omaha, Nebraska
  - GSK Investigational Site, Binghamton, New York
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Dayton, Ohio
  - GSK Investigational Site, Charleston, South Carolina
  - GSK Investigational Site, Mt. Pleasant, South Carolina
- Finland (10):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vantaa
- Poland (7):
  - GSK Investigational Site, Dębica
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Lodz
  - GSK Investigational Site, Osielsko
  - GSK Investigational Site, Siemianowice Śląskie
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wroclaw

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 32 centers from Finland, Poland and United States.
Pre-assignment Details: All subjects were included in the trial.
Period: Overall Study
Arm/Group | rMenB_0_2 Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group | ABCWY_0_2_6 Group
Started | 228 | 232 | 157 | 134 | 152 | 160
Completed | 209 | 211 | 141 | 123 | 137 | 147
Not Completed | 19 | 21 | 16 | 11 | 15 | 13
Not completed — Adverse Event | 1 | 2 | 2 | 2 | 0 | 1
Not completed — Withdrawal by Subject | 8 | 10 | 8 | 6 | 5 | 4
Not completed — Lost to Follow-up | 6 | 7 | 4 | 1 | 8 | 4
Not completed — Protocol Violation | 2 | 1 | 0 | 1 | 2 | 3
Not completed — Other | 2 | 1 | 2 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | rMenB_0_2 Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group | ABCWY_0_2_6 Group | Total
Number analyzed (Participants) | 228 | 232 | 157 | 134 | 152 | 160 | 1063
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.5 (3.09) | 14.2 (3.17) | 14.4 (3.01) | 14.4 (3.06) | 14.5 (3.1) | 14.3 (3.16) | 14.4 (3.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 130 | 119 | 101 | 76 | 89 | 96 | 611
  Male | 98 | 113 | 56 | 58 | 63 | 64 | 452

OUTCOME MEASURES:

1. Primary Outcome: Human Serum Bactericidal Assay (hSBA) Geometric Mean Titers (GMTs) Against N. Meningitidis Serogroup B Test Strains When Administered According to 0_2 Month Schedule.
Description: The non-inferiority of the Meningococcal (groups A, C, W and Y) oligosaccharide diphtheria CRM-197 conjugate combined with meningococcal (group B) multicomponent recombinant (MenABCWY) vaccine to Meningococcal (group B) multicomponent recombinant adsorbed (Bexsero) vaccine, administered according to 0, 2 month schedule, as measured by hSBA GMTs against N.meningitidis serogroup B test strains at 1 month after the last meningococcal vaccination, is reported. The test strains assessed were Meningitis B NZ98/254 Ab, Meningitis B M14459 Ab, Meningitis B M07-0241084 Ab and Meningitis B 96217 Ab. This outcome measure was evaluated in the rMenB_0_2 and ABCWY_ 0_2 Groups.
Time Frame: At baseline (Month 0) and 1 month after the last meningococcal vaccination (Month 3)
Population: Analysis was done on Per Protocol Set (PPS)-Month 3, which included all screened subjects who received a study vaccination, provided evaluable serum samples at pre- & post-vaccination, with results available for at least 1 serogroup B test strain & who was not excluded due to protocol deviations/other reasons defined before unblinding/analysis
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ABCWY_ 0_2 Group | rMenB_0_2 Group
Number analyzed (Participants) | 158 | 150
Titers
  M14459 strain (Month 0): number analyzed (Participants) | 155 | 147
  M14459 strain (Month 0) | 1.28 [1.07 to 1.53] | 1.31 [1.09 to 1.57]
  M14459 strain (Month 3) | 11.64 [8.61 to 16] | 15.78 [12 to 22]
  M07-0241084 strain (Month 0): number analyzed (Participants) | 151 | 148
  M07-0241084 strain (Month 0) | 2.12 [1.60 to 2.82] | 2.16 [1.61 to 2.89]
  M07-0241084 strain (Month 3): number analyzed (Participants) | 154 | 150
  M07-0241084 strain (Month 3) | 8.19 [6.31 to 11] | 11.56 [8.86 to 15]
  96217 strain (Month 0): number analyzed (Participants) | 152 | 143
  96217 strain (Month 0) | 2.93 [2.13 to 4.03] | 2.36 [1.70 to 3.28]
  96217 strain (Month 3): number analyzed (Participants) | 156 | 149
  96217 strain (Month 3) | 150.82 [118 to 192] | 229.29 [179 to 294]
  NZ98/254 strain (Month 0): number analyzed (Participants) | 154 | 147
  NZ98/254 strain (Month 0) | 1.27 [1.06 to 1.53] | 1.15 [0.95 to 1.39]
  NZ98/254 strain (Month 3): number analyzed (Participants) | 157 | 150
  NZ98/254 strain (Month 3) | 11.95 [9.10 to 16] | 24.31 [18 to 32]
Statistical Analysis 1: Comparison: ABCWY_ 0_2 Group vs rMenB_0_2 Group; Non-inferiority response against N. meningitidis serogroup B test strain M14459 of the MenABCWY vaccine to that of the Bexsero vaccine, administered according to 0, 2 month schedule; Test type: Non-Inferiority or Equivalence — Non-inferiority was concluded when, at 1 month after the second meningococcal vaccination (Visit Month 3), the lower limit of the two-sided 95% confidence interval for the between-group ratios of GMTs (ABCWY_0_2 versus rMenB_0_2) was greater than 0.5 for each of the four serogroup B test strains; ANCOVA; Geometric Mean Ratio = 0.74, 95% CI 2-sided [0.53 to 1.02]
Statistical Analysis 2: Comparison: ABCWY_ 0_2 Group vs rMenB_0_2 Group; Non-inferiority response against N. meningitidis serogroup B test strain M07-0241084 of the MenABCWY vaccine to that of the Bexsero vaccine, administered according to 0, 2 month schedule; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Geometric Mean Ratio = 0.71, 95% CI 2-sided [0.54 to 0.94]
Statistical Analysis 3: Comparison: ABCWY_ 0_2 Group vs rMenB_0_2 Group; Non-inferiority response against N. meningitidis serogroup B test strain 96217 of the MenABCWY vaccine to that of the Bexsero vaccine, administered according to 0, 2 month schedule; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Geometric Mean Ratio = 0.66, 95% CI 2-sided [0.51 to 0.85]
Statistical Analysis 4: Comparison: ABCWY_ 0_2 Group vs rMenB_0_2 Group; Non-inferiority response against N. meningitidis serogroup B test strain NZ98/254 of the MenABCWY vaccine to that of the Bexsero vaccine, administered according to 0, 2 month schedule; Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; ANCOVA; Geometric Mean Ratio = 0.49, 95% CI 2-sided [0.37 to 0.66]

2. Secondary Outcome: hSBA GMTs Against N. Meningitidis Serogroups A, C, W and Y and Serogroup B Test Strains When Administered According to 0_2_6 Month and 0_2 Month Schedule.
Description: The immunogenicity of MenABCWY vaccine, administered according to 0, 2, 6 months schedule was compared with those administered according to 0, 2 months schedule, as measured by hSBA GMTs against N. meningitidis serogroup B test strains and serogroups A,C, W and Y at 1 month after the last meningococcal vaccination. The B test strains assessed were Meningitis B NZ98/254 Ab, Meningitis B M14459 Ab, Meningitis B M07-0241084 Ab and Meningitis B 96217 Ab. This outcome measure was evaluated in the ABCWY_ 0_2 and ABCWY_0_2_6 Groups. 1 month post last meningococcal vaccination corresponds to Month 3 for ABCWY_0_2 Group and Month 7 for ABCWY_0_2_6 Group.
Time Frame: At baseline (Month 0) and 1 month after the last meningococcal vaccination (Month 3 for ABCWY_ 0_2 Group and Month 7 for ABCWY_0_2_6 Group)
Population: Analysis was done on the FAS-1 month after the last meningococcal vaccination.All subjects in All Enrolled Set who received a study meningococcal vaccination & provided evaluable serum samples at pre- & at one month after the last meningococcal vaccination whose result is available for at least one A,C,W,or Y serogroup or serogroup B test strain.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ABCWY_ 0_2 Group | ABCWY_0_2_6 Group
Number analyzed (Participants) | 213 | 151
Titers
  M14459 strain (Month 0): number analyzed (Participants) | 207 | 151
  M14459 strain (Month 0) | 1.21 [1.07 to 1.37] | 1.12 [0.98 to 1.28]
  M14459 strain (Month 3/Month 7): number analyzed (Participants) | 211 | 151
  M14459 strain (Month 3/Month 7) | 12.17 [9.60 to 15] | 27.09 [21 to 35]
  M07-0241084 strain (Month 0): number analyzed (Participants) | 201 | 145
  M07-0241084 strain (Month 0) | 2.36 [1.85 to 3.01] | 2.05 [1.58 to 2.67]
  M07-0241084 strain (Month 3/Month 7): number analyzed (Participants) | 206 | 148
  M07-0241084 strain (Month 3/Month 7) | 8.91 [7.10 to 11] | 18.03 [14 to 23]
  96217 strain (Month 0): number analyzed (Participants) | 205 | 146
  96217 strain (Month 0) | 2.31 [1.75 to 3.06] | 2.28 [1.68 to 3.07]
  96217 strain (Month 3/Month7): number analyzed (Participants) | 210 | 150
  96217 strain (Month 3/Month7) | 174.27 [142 to 215] | 298.76 [239 to 374]
  NZ98/254 strain (Month 0): number analyzed (Participants) | 208 | 151
  NZ98/254 strain (Month 0) | 1.24 [1.09 to 1.41] | 1.07 [0.93 to 1.23]
  NZ98/254 strain (Month 3/Month7): number analyzed (Participants) | 212 | 151
  NZ98/254 strain (Month 3/Month7) | 12.57 [9.81 to 16] | 17.55 [13 to 23]
  A human serogroup (Month 0): number analyzed (Participants) | 206 | 146
  A human serogroup (Month 0) | 1.19 [1.04 to 1.36] | 1.10 [0.95 to 1.27]
  A human serogroup (Month 3/Month7): number analyzed (Participants) | 211 | 147
  A human serogroup (Month 3/Month7) | 66.73 [54 to 83] | 125.45 [99 to 159]
  C human serogroup (Month 0): number analyzed (Participants) | 206 | 145
  C human serogroup (Month 0) | 3.59 [2.85 to 4.53] | 3.19 [2.48 to 4.10]
  C human serogroup (Month 3/Month7): number analyzed (Participants) | 212 | 149
  C human serogroup (Month 3/Month7) | 158.8 [127 to 199] | 376.44 [295 to 481]
  W human serogroup (Month 0): number analyzed (Participants) | 198 | 138
  W human serogroup (Month 0) | 5.20 [3.56 to 7.59] | 4.64 [3.05 to 7.05]
  W human serogroup (Month 3/Month7): number analyzed (Participants) | 208 | 140
  W human serogroup (Month 3/Month7) | 206.62 [175 to 244] | 295.9 [246 to 356]
  Y human serogroup (Month 0): number analyzed (Participants) | 202 | 150
  Y human serogroup (Month 0) | 1.33 [1.10 to 1.60] | 1.26 [1.03 to 1.55]
  Y human serogroup (Month 3/Month7): number analyzed (Participants) | 213 | 150
  Y human serogroup (Month 3/Month7) | 79.84 [62 to 103] | 163.69 [124 to 216]

3. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥LLQ Against N. Meningitidis Serogroups A, C, W and y and Serogroup B Test Strains When Administered According to 0_2_6 Month and 0_2 Month Schedule.
Description: The immunogenicity of MenABCWY vaccine, administered according to 0, 2, 6 month schedule, was compared with those, administered according to 0, 2 month schedule, as measured by the percentages of subjects with hSBA titers ≥ LLQ against N. meningitidis serogroup B test strains at 1 month after the last meningococcal vaccination.
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | ABCWY_ 0_2 Group | ABCWY_0_2_6 Group
Number analyzed (Participants) | 213 | 151
Percentages of subjects
  NZ98/254 strain (Month 0): number analyzed (Participants) | 208 | 151
  NZ98/254 strain (Month 0) | 6 [3.37 to 10.45] | 2 [0.41 to 5.70]
  NZ98/254 strain (Month 3/7): number analyzed (Participants) | 212 | 151
  NZ98/254 strain (Month 3/7) | 63 [55.85 to 69.26] | 74 [65.72 to 80.35]
  M14459 strain (Month 0): number analyzed (Participants) | 207 | 151
  M14459 strain (Month 0) | 5 [2.68 to 9.31] | 2 [0.41 to 5.70]
  M14459 strain (Month 3/Month 7): number analyzed (Participants) | 211 | 151
  M14459 strain (Month 3/Month 7) | 70 [63.48 to 76.23] | 89 [83.36 to 93.82]
  M07-0241084 strain (Month 0): number analyzed (Participants) | 201 | 145
  M07-0241084 strain (Month 0) | 18 [13.30 to 24.47] | 18 [12.06 to 25.16]
  M07-0241084 strain (Month 3/7): number analyzed (Participants) | 206 | 148
  M07-0241084 strain (Month 3/7) | 49 [41.54 to 55.59] | 72 [64.35 to 79.33]
  96217 strain (Month 0): number analyzed (Participants) | 205 | 144
  96217 strain (Month 0) | 28 [22.24 to 34.99] | 27 [20.02 to 35.11]
  96217 strain (Month 3/7): number analyzed (Participants) | 210 | 150
  96217 strain (Month 3/7) | 97 [93.25 to 98.65] | 99 [96.34 to 99.98]
  Serogroup A (Month 0): number analyzed (Participants) | 206 | 146
  Serogroup A (Month 0) | 3 [1.08 to 6.23] | 1 [0.02 to 3.76]
  Serogroup A (Month 3/7): number analyzed (Participants) | 211 | 147
  Serogroup A (Month 3/7) | 88 [83.01 to 92.18] | 95 [89.56 to 97.62]
  Serogroup C (Month 0): number analyzed (Participants) | 206 | 145
  Serogroup C (Month 0) | 44 [37.28 to 51.24] | 41 [32.62 to 49.15]
  Serogroup C (Month 3/7): number analyzed (Participants) | 212 | 149
  Serogroup C (Month 3/7) | 99 [96.63 to 99.89] | 100 [97.55 to 100]
  Serogroup W (Month 0): number analyzed (Participants) | 198 | 138
  Serogroup W (Month 0) | 27 [21.20 to 34.04] | 22 [15.17 to 29.56]
  Serogroup W (Month 3/7): number analyzed (Participants) | 208 | 140
  Serogroup W (Month 3/7) | 97 [93.19 to 98.64] | 99 [96.08 to 99.98]
  Serogroup Y (Month 0): number analyzed (Participants) | 202 | 150
  Serogroup Y (Month 0) | 9 [5.37 to 13.72] | 6 [2.78 to 11.08]
  Serogroup Y (Month 3/7): number analyzed (Participants) | 213 | 150
  Serogroup Y (Month 3/7) | 92 [86.97 to 94.91] | 97 [93.31 to 99.27]

4. Secondary Outcome: hSBA GMTs Against Each of N. Meningitidis Serogroups A, C, W and Y and Serogroup B Test Strains When Administered According to 0_1 Month, 0_2 Month, 0_6 Month and 0, 11 Month Schedule.
Description: The immunogenicity of MenABCWY vaccine, administered according to 0, 2 months schedule, was compared with those, administered according to 0, 1 month, 0, 6 month and 0, 11 month schedules as measured by hSBA GMTs against N. meningitidis serogroups A, C, W and Y and serogroup B test strains at 1 month after the second meningococcal vaccination.
Time Frame: At 1 Month after the last vaccination (Month 2 for ABCWY_0_1 Group, Month 3 for ABCWY_0_2 Group, Month 7 for ABCWY_0_6 Group and Month 13 for ABCWY_0_11 Group)
Population: Analysis was done on the FAS- 1 month after last meningococcal vaccination, which included all screened subjects who provided informed consent, received a study vaccination & provided evaluable serum samples at 1 month after last vaccination whose results were available for atleast 1 serogroup or B strain
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group
Number analyzed (Participants) | 213 | 143 | 123 | 133
Titers
  NZ98/254 strain: number analyzed (Participants) | 212 | 142 | 121 | 131
  NZ98/254 strain | 12.32 [9.82 to 15] | 6.33 [4.86 to 8.23] | 13.64 [10 to 18] | 15.87 [12 to 21]
  M14459 strain: number analyzed (Participants) | 211 | 140 | 122 | 133
  M14459 strain | 12.72 [10 to 16] | 9.19 [7.11 to 12] | 26.48 [20 to 35] | 29.57 [23 to 39]
  M07-0241084 strain: number analyzed (Participants) | 206 | 140 | 123 | 131
  M07-0241084 strain | 9.15 [7.52 to 11] | 6.59 [5.25 to 8.27] | 15.04 [12 to 19] | 16.22 [13 to 21]
  96217 strain: number analyzed (Participants) | 210 | 143 | 121 | 133
  96217 strain | 165.47 [133 to 206] | 117.28 [91 to 151] | 237.89 [182 to 310] | 244.97 [189 to 317]
  A human serogroup: number analyzed (Participants) | 211 | 142 | 123 | 133
  A human serogroup | 69.61 [56 to 87] | 79.87 [62 to 103] | 140.76 [108 to 184] | 162.76 [126 to 211]
  C human serogroup: number analyzed (Participants) | 212 | 142 | 123 | 131
  C human serogroup | 162.57 [132 to 201] | 145.73 [114 to 186] | 225.00 [174 to 290] | 292.61 [227 to 376]
  W human serogroup: number analyzed (Participants) | 208 | 143 | 123 | 131
  W human serogroup | 215.72 [182 to 256] | 197.69 [162 to 241] | 376.03 [306 to 462] | 531.79 [434 to 652]
  Y human serogroup: number analyzed (Participants) | 213 | 142 | 123 | 132
  Y human serogroup | 71.66 [55 to 93] | 57.45 [42 to 78] | 120.76 [88 to 166] | 209.53 [153 to 286]

5. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ Lower Limit of Quantitation (LLQ) Against N. Meningitidis Serogroup B Test Strains When Administered According to 0_2 Month Schedule.
Description: A sufficient immune response following Bexsero vaccine, administered according to 0, 2 month schedule, as measured by the percentage of subjects with hSBA titers ≥ Lower Limit of Quantitation (LLQ) against N. meningitidis serogroup B test strains at 1 month after the last meningococcal vaccination, was to be demonstrated. Criterion: the immune response was to be considered sufficient if the lower limit of the two-sided 95% CI for the percentage of subjects with hSBA titers ≥ LLQ was greater than 75% for each of the four serogroup B test strains. The test strains assessed were Meningitis B NZ98/254 Ab, Meningitis B M14459 Ab, Meningitis B M07-0241084 Ab and Meningitis B 96217 Ab.
Time Frame: At baseline (Month 0) and 1 month after the last meningococcal vaccination (Month 3)
Population: Analysis was done on Full Analysis Set(FAS)- 1 month post meningococcal vaccination. Subjects in All Enrolled Set who received a study meningococcal vaccination & provided evaluable serum samples at pre- & at 1 month post last meningococcal vaccination whose result is available for at least one A,C,W or Y serogroup or serogroup B test strain.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB_0_2 Group | ABCWY_ 0_2 Group
Number analyzed (Participants) | 188 | 185
Percentages of subjects
  NZ98/254 strain - month 0 (LLQ = 8.2) | 7 [3.73 to 11.53] | 6 [3.40 to 11.06]
  NZ98/254 strain - month 3 (LLQ = 8.2) | 88 [82.82 to 92.52] | 61 [53.65 to 68.15]
  M14459 strain - month 0 (LLQ = 8.0): number analyzed (Participants) | 184 | 179
  M14459 strain - month 0 (LLQ = 8.0) | 7 [3.41 to 11.11] | 5 [2.32 to 9.33]
  M14459 strain - month 3 (LLQ = 8.0): number analyzed (Participants) | 184 | 179
  M14459 strain - month 3 (LLQ = 8.0) | 82 [75.75 to 87.32] | 68 [60.21 to 74.39]
  M07-0241084 strain - month 0 (LLQ = 8.9): number analyzed (Participants) | 188 | 176
  M07-0241084 strain - month 0 (LLQ = 8.9) | 21 [15.19 to 27.25] | 18 [12.78 to 24.69]
  M07-0241084 strain - month 3 (LLQ = 8.9): number analyzed (Participants) | 188 | 176
  M07-0241084 strain - month 3 (LLQ = 8.9) | 66 [59.26 to 73.19] | 47 [39.60 to 54.81]
  96217 strain - month 0 (LLQ = 8.6): number analyzed (Participants) | 186 | 178
  96217 strain - month 0 (LLQ = 8.6) | 23 [17.26 to 29.85] | 29 [22.14 to 35.89]
  96217 strain - month 3 (LLQ = 8.6): number analyzed (Participants) | 186 | 178
  96217 strain - month 3 (LLQ = 8.6) | 99 [97.04 to 99.99] | 97 [92.81 to 98.75]

6. Secondary Outcome: hSBA GMTs Against N. Meningitidis Serogroups A, C, W and Y and Serogroup B Test Strains When Administered According to 0_2_6 Month and 0_6 Month Schedule.
Description: The immunogenicity of MenABCWY vaccine, administered according to 0, 2, 6 months schedule was compared with those administered according to 0, 6 months schedule, as measured by hSBA GMTs against N. meningitidis serogroups A, C, W and Y and serogroup B test strains at 1 month after the last meningococcal vaccination.
Time Frame: At 1 month after last vaccination (Month 7)
Population: Analysis was done on the FAS- 1 month after last meningococcal vaccination, which included all screened subjects who provided informed consent, received a study vaccination & provided evaluable serum samples at 1 month after last vaccination whose results were available for atleast 1 serogroup or B strains
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | ABCWY_0_6 Group | ABCWY_0_2_6 Group
Number analyzed (Participants) | 123 | 151
Titers
  NZ98/254 strain: number analyzed (Participants) | 121 | 151
  NZ98/254 strain | 13.62 [9.98 to 19] | 17.13 [13 to 23]
  M14459 strain: number analyzed (Participants) | 122 | 151
  M14459 strain | 27.82 [21 to 36] | 29.27 [23 to 37]
  M07-0241084 strain: number analyzed (Participants) | 123 | 148
  M07-0241084 strain | 17.43 [13 to 23] | 20.92 [16 to 27]
  96217 strain: number analyzed (Participants) | 121 | 150
  96217 strain | 240.13 [186 to 310] | 291.63 [232 to 367]
  Serogroup A: number analyzed (Participants) | 123 | 147
  Serogroup A | 140.14 [107 to 184] | 128.75 [101 to 164]
  Serogroup C: number analyzed (Participants) | 123 | 149
  Serogroup C | 246.48 [191 to 318] | 413.60 [328 to 522]
  Serogroup W: number analyzed (Participants) | 123 | 140
  Serogroup W | 341.90 [283 to 413] | 282.74 [237 to 338]
  Serogroup Y: number analyzed (Participants) | 123 | 150
  Serogroup Y | 123.96 [91 to 169] | 151.36 [115 to 200]

7. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ Lower Limit of Quantitation (LLQ) Against Serogroups A, C, W and Y and Serogroup B Test Strains When Administered According to 0_2_6 Month and 0_6 Month Schedule.
Description: The immunogenicity of MenABCWY vaccine, administered according to 0, 2, 6 month schedule, was compared with those, administered according to 0, 6 month schedule, as measured by the percentages of subjects with hSBA titers ≥ LLQ against serogroups A, C, W and Y and serogroup B test strains at 1 month after the last meningococcal vaccination.
Time Frame: At baseline (Month 0) and 1 month after the last meningococcal vaccination (Month 7)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | ABCWY_0_6 Group | ABCWY_0_2_6 Group
Number analyzed (Participants) | 123 | 151
Percentages of subjects
  NZ98/254 strain - month 0 (LLQ=8.2): number analyzed (Participants) | 120 | 151
  NZ98/254 strain - month 0 (LLQ=8.2) | 5 [1.86 to 10.57] | 2 [0.41 to 5.70]
  NZ98/254 strain - month 7 (LLQ=8.2): number analyzed (Participants) | 121 | 151
  NZ98/254 strain - month 7 (LLQ=8.2) | 64 [55.25 to 72.95] | 74 [65.72 to 80.35]
  M14459 strain - month 0 (LLQ=8.0): number analyzed (Participants) | 121 | 151
  M14459 strain - month 0 (LLQ=8.0) | 5 [1.84 to 10.48] | 2 [0.41 to 5.70]
  M14459 strain - month 7 (LLQ=8.0): number analyzed (Participants) | 122 | 151
  M14459 strain - month 7 (LLQ=8.0) | 87 [79.58 to 92.31] | 89 [83.36 to 93.82]
  M07-0241084 strain - month 0 (LLQ=8.9): number analyzed (Participants) | 122 | 145
  M07-0241084 strain - month 0 (LLQ=8.9) | 14 [8.33 to 21.37] | 18 [12.06 to 25.16]
  M07-0241084 strain - month 7 (LLQ=8.9): number analyzed (Participants) | 123 | 148
  M07-0241084 strain - month 7 (LLQ=8.9) | 66 [56.76 to 74.16] | 72 [64.35 to 79.33]
  96217 strain - month 0 (LLQ=8.6): number analyzed (Participants) | 119 | 144
  96217 strain - month 0 (LLQ=8.6) | 27 [19.18 to 35.79] | 27 [20.02 to 35.11]
  996217 strain - month 7 (LLQ=8.6): number analyzed (Participants) | 121 | 150
  996217 strain - month 7 (LLQ=8.6) | 98 [92.93 to 99.49] | 99 [96.34 to 99.98]
  A human serogroup - month 0 (LLQ=22.7): number analyzed (Participants) | 118 | 146
  A human serogroup - month 0 (LLQ=22.7) | 2 [0.21 to 5.99] | 1 [0.02 to 3.76]
  A human serogroup - month 7 (LLQ=22.7): number analyzed (Participants) | 123 | 147
  A human serogroup - month 7 (LLQ=22.7) | 94 [88.63 to 97.68] | 95 [89.56 to 97.62]
  C human serogroup - month 0 (LLQ=5.2): number analyzed (Participants) | 122 | 145
  C human serogroup - month 0 (LLQ=5.2) | 42 [32.94 to 51.07] | 41 [32.62 to 49.15]
  C human serogroup - month 7 (LLQ=5.2): number analyzed (Participants) | 123 | 149
  C human serogroup - month 7 (LLQ=5.2) | 99 [95.55 to 99.98] | 100 [97.55 to 100]
  W human serogroup - month 0 (LLQ=39.6): number analyzed (Participants) | 119 | 138
  W human serogroup - month 0 (LLQ=39.6) | 20 [13.37 to 28.51] | 22 [15.17 to 29.56]
  W human serogroup -month 7 (LLQ=39.6): number analyzed (Participants) | 123 | 140
  W human serogroup -month 7 (LLQ=39.6) | 99 [95.55 to 99.98] | 99 [96.08 to 99.98]
  Y human serogroup - month 0 (LLQ=14.7): number analyzed (Participants) | 120 | 150
  Y human serogroup - month 0 (LLQ=14.7) | 7 [2.92 to 12.71] | 6 [2.78 to 11.08]
  Y human serogroup - month 7 (LLQ=14.7): number analyzed (Participants) | 123 | 150
  Y human serogroup - month 7 (LLQ=14.7) | 94 [88.63 to 97.68] | 97 [93.31 to 99.27]

8. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥ LLQ Against N. Meningitidis Serogroups A, C, W and Y and Serogroup B Test Strains When Administered According to 0_1 Month, 0_2 Month, 0_6 Month and 0_11 Month Schedule.
Description: The immunogenicity of MenABCWY vaccine, administered according to 0, 2 month schedule, was compared with those, administered according to 0, 1 month, 0, 6 month and 0, 11 month schedules, as measured by the percentages of subjects with hSBA titers ≥ LLQ against N. meningitidis serogroups A, C, W and Y and serogroup B test strains at 1 month after the second meningococcal vaccination.
Time Frame: At 1 month after second vaccination (Month 2 for ABCWY_0_1 Group, Month 3 for ABCWY_0_2 Group , Month 7 for ABCWY_0_6 Group and Month 13 for ABCWY_0_11 Group)
Population: as for outcome 4
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group
Number analyzed (Participants) | 213 | 143 | 123 | 133
Percentages of subjects
  NZ98/254 strain (LLQ=8.2): number analyzed (Participants) | 212 | 142 | 121 | 131
  NZ98/254 strain (LLQ=8.2) | 63 [55.85 to 69.26] | 44 [35.36 to 52.23] | 64 [55.25 to 72.95] | 73 [64.85 to 80.63]
  M14459 strain (LLQ=8.0): number analyzed (Participants) | 211 | 140 | 122 | 133
  M14459 strain (LLQ=8.0) | 70 [63.48 to 76.23] | 62 [53.56 to 70.20] | 87 [79.58 to 92.31] | 89 [82.08 to 93.55]
  M07-0241084 strain (LLQ=8.9): number analyzed (Participants) | 206 | 140 | 123 | 131
  M07-0241084 strain (LLQ=8.9) | 49 [41.54 to 55.59] | 40 [31.82 to 48.61] | 66 [56.76 to 74.16] | 69 [60.82 to 77.21]
  96217 strain (LLQ=8.6): number analyzed (Participants) | 210 | 143 | 121 | 133
  96217 strain (LLQ=8.6) | 97 [93.25 to 98.65] | 97 [92.99 to 99.23] | 98 [92.93 to 99.49] | 98 [93.55 to 99.53]
  Serogroup A (LLQ=22.7): number analyzed (Participants) | 211 | 142 | 123 | 133
  Serogroup A (LLQ=22.7) | 88 [83.01 to 92.18] | 92 [85.70 to 95.56] | 94 [88.63 to 97.68] | 94 [88.49 to 97.37]
  Serogroup C (LLQ=5.2): number analyzed (Participants) | 212 | 142 | 123 | 131
  Serogroup C (LLQ=5.2) | 99 [96.63 to 99.89] | 100 [97.44 to 100] | 99 [95.55 to 99.99] | 100 [97.22 to 100]
  Serogroup W (LLQ=39.6): number analyzed (Participants) | 208 | 143 | 123 | 131
  Serogroup W (LLQ=39.6) | 97 [93.19 to 98.64] | 96 [91.09 to 98.44] | 99 [95.55 to 99.98] | 98 [93.45 to 99.53]
  Serogroup Y (LLQ=14.7): number analyzed (Participants) | 213 | 142 | 123 | 132
  Serogroup Y (LLQ=14.7) | 92 [86.97 to 94.91] | 85 [78.29 to 90.61] | 94 [88.63 to 97.68] | 97 [92.42 to 99.17]

9. Secondary Outcome: hSBA GMTs Against Serogroups A, C, W and Y and Serogroup B Test Strains at All the Relevant Time Points for All Schedules.
Description: The kinetic of immune response (at Months 0, 2, 3, 7 and 13) following different vaccination schedules as measured by the adjusted hSBA GMTs against serogroups A,C, W and Y and serogroup B test strains was assessed.
Time Frame: At Month 0, Month 2, Month 3, Month 7 and Month 13
Population: Analysis was done on the FAS Month 13 which included all screened subjects who received a study vaccination & provided evaluable serum samples at month 0 and atleast from month 2 to 13 and provided results for atleast one serogroup or serogroup B test strain.
Measure: Geometric Mean (95% Confidence Interval); unit: Titers
Arm/Group | rMenB_0_2 Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group | ABCWY_0_2_6 Group
Number analyzed (Participants) | 188 | 185 | 122 | 114 | 128 | 137
Titers
  NZ98/254 strain (Month 0): number analyzed (Participants) | 188 | 185 | 120 | 112 | 126 | 134
  NZ98/254 strain (Month 0) | 1.22 [1.08 to 1.38] | 1.22 [1.08 to 1.38] | 1.21 [1.04 to 1.40] | 1.13 [0.97 to 1.31] | 1.12 [0.97 to 1.29] | 1.06 [0.93 to 1.22]
  NZ98/254 strain (Month 2): number analyzed (Participants) | 188 | 185 | 120 | 112 | 126 | 134
  NZ98/254 strain (Month 2) | 2.67 [2.14 to 3.34] | 2.27 [1.82 to 2.84] | 6.50 [4.98 to 8.48] | 1.92 [1.46 to 2.51] | 3.87 [2.98 to 5.01] | 2.20 [1.71 to 2.82]
  NZ98/254 strain (Month 3): number analyzed (Participants) | 188 | 185 | 120 | 112 | 126 | 134
  NZ98/254 strain (Month 3) | 27.17 [22 to 34] | 11.46 [9.28 to 14] | 3.15 [2.44 to 4.05] | 1.69 [1.31 to 2.19] | 2.38 [1.86 to 3.05] | 12.80 [10 to 16]
  NZ98/254 strain (Month 7): number analyzed (Participants) | 188 | 185 | 120 | 112 | 126 | 134
  NZ98/254 strain (Month 7) | 3.00 [2.44 to 3.67] | 2.41 [1.97 to 2.95] | 1.88 [1.47 to 2.40] | 14.30 [11 to 18] | 1.75 [1.38 to 2.22] | 18.24 [14 to 23]
  NZ98/254 strain (Month 13): number analyzed (Participants) | 188 | 185 | 120 | 112 | 126 | 134
  NZ98/254 strain (Month 13) | 2.33 [1.92 to 2.83] | 1.93 [1.59 to 2.33] | 1.81 [1.44 to 2.27] | 2.57 [2.04 to 3.25] | 17.08 [14 to 21] | 2.82 [2.28 to 3.51]
  M14459 strain(Month 0): number analyzed (Participants) | 184 | 179 | 112 | 108 | 123 | 134
  M14459 strain(Month 0) | 1.37 [1.21 to 1.56] | 1.22 [1.08 to 1.39] | 1.22 [1.04 to 1.42] | 1.21 [1.04 to 1.41] | 1.34 [1.15 to 1.55] | 1.17 [1.02 to 1.35]
  M14459 strain (Month 2): number analyzed (Participants) | 184 | 179 | 112 | 108 | 123 | 134
  M14459 strain (Month 2) | 2.83 [2.31 to 3.46] | 2.55 [2.08 to 3.13] | 9.23 [7.21 to 12] | 2.34 [1.82 to 2.99] | 3.94 [3.11 to 4.98] | 2.40 [1.92 to 3.01]
  M14459 strain (Month 3): number analyzed (Participants) | 184 | 179 | 112 | 108 | 123 | 134
  M14459 strain (Month 3) | 18.29 [15 to 23] | 12.85 [10 to 16] | 5.30 [4.04 to 6.93] | 2.15 [1.64 to 2.82] | 3.11 [2.40 to 4.02] | 15.24 [12 to 20]
  M14459 strain (Month 7): number analyzed (Participants) | 184 | 179 | 112 | 108 | 123 | 134
  M14459 strain (Month 7) | 3.52 [2.91 to 4.26] | 3.24 [2.68 to 3.93] | 2.19 [1.74 to 2.77] | 27.47 [22 to 35] | 1.95 [1.56 to 2.43] | 28.56 [23 to 35]
  M14459 strain (Month 13): number analyzed (Participants) | 184 | 179 | 112 | 108 | 123 | 134
  M14459 strain (Month 13) | 2.46 [2.03 to 2.97] | 2.29 [1.89 to 2.78] | 1.95 [1.54 to 2.45] | 3.22 [2.55 to 4.06] | 29.01 [23 to 36] | 3.17 [2.57 to 3.92]
  M07-0241084 strain (Month 0): number analyzed (Participants) | 188 | 176 | 117 | 113 | 121 | 128
  M07-0241084 strain (Month 0) | 2.26 [1.81 to 2.82] | 2.07 [1.65 to 2.59] | 2.01 [1.53 to 2.63] | 2.06 [1.57 to 2.71] | 2.59 [1.99 to 3.37] | 1.83 [1.42 to 2.36]
  M07-0241084 strain (Month 2): number analyzed (Participants) | 188 | 176 | 117 | 113 | 121 | 128
  M07-0241084 strain (Month 2) | 5.09 [4.26 to 6.07] | 4.30 [3.59 to 5.14] | 6.73 [5.44 to 8.34] | 3.51 [2.83 to 4.35] | 4.90 [3.97 to 6.04] | 4.20 [3.43 to 5.15]
  M07-0241084 strain(Month 3): number analyzed (Participants) | 188 | 176 | 117 | 113 | 121 | 128
  M07-0241084 strain(Month 3) | 13.91 [12 to 17] | 8.82 [7.29 to 11] | 4.39 [3.49 to 5.50] | 3.30 [2.62 to 4.15] | 3.55 [2.84 to 4.43] | 9.29 [7.49 to 12]
  M07-0241084 strain (Month 7): number analyzed (Participants) | 188 | 176 | 117 | 113 | 121 | 128
  M07-0241084 strain (Month 7) | 5.42 [4.51 to 6.51] | 4.68 [3.88 to 5.63] | 3.36 [2.69 to 4.20] | 15.70 [13 to 20] | 2.96 [2.38 to 3.67] | 19.18 [16 to 24]
  M07-0241084 strain(Month 13): number analyzed (Participants) | 188 | 176 | 117 | 113 | 121 | 128
  M07-0241084 strain(Month 13) | 4.45 [3.71 to 5.35] | 4.01 [3.34 to 4.83] | 3.07 [2.46 to 3.83] | 5.42 [4.33 to 6.77] | 15.68 [13 to 19] | 5.80 [4.70 to 7.16]
  96217 strain (Month 0): number analyzed (Participants) | 186 | 178 | 120 | 112 | 128 | 121
  96217 strain (Month 0) | 2.32 [1.82 to 2.95] | 2.84 [2.23 to 3.62] | 2.88 [2.16 to 3.83] | 2.39 [1.78 to 3.21] | 2.78 [2.11 to 3.68] | 2.57 [1.94 to 3.40]
  96217 strain(Month 2): number analyzed (Participants) | 186 | 178 | 120 | 112 | 128 | 121
  96217 strain(Month 2) | 16.48 [13 to 21] | 11.62 [8.96 to 15] | 124.75 [92 to 169] | 11.61 [8.49 to 16] | 11.94 [8.87 to 16] | 8.54 [6.33 to 12]
  96217 strain(Month 3): number analyzed (Participants) | 186 | 178 | 120 | 112 | 128 | 121
  96217 strain(Month 3) | 263.56 [211 to 329] | 169.65 [136 to 212] | 82.23 [63 to 107] | 8.61 [6.57 to 11] | 7.72 [5.97 to 9.99] | 162.27 [125 to 210]
  96217 strain (Month 7): number analyzed (Participants) | 186 | 178 | 120 | 112 | 128 | 121
  96217 strain (Month 7) | 61.46 [50 to 75] | 43.01 [35 to 53] | 37.26 [29 to 47] | 264.85 [207 to 340] | 5.19 [4.10 to 6.58] | 306.14 [242 to 388]
  96217 strain (Month 13): number analyzed (Participants) | 186 | 178 | 120 | 112 | 128 | 121
  96217 strain (Month 13) | 33.07 [27 to 41] | 22.48 [18 to 28] | 24.00 [18 to 31] | 42.27 [32 to 55] | 264.32 [205 to 341] | 47.22 [37 to 61]
  Serogroup A (Month 0): number analyzed (Participants) | 172 | 178 | 107 | 105 | 120 | 127
  Serogroup A (Month 0) | 1.37 [1.18 to 1.59] | 1.17 [1.02 to 1.36] | 1.38 [1.15 to 1.65] | 1.08 [0.90 to 1.30] | 1.19 [1.00 to 1.41] | 1.06 [0.90 to 1.25]
  Serogroup A (Month 2): number analyzed (Participants) | 172 | 178 | 107 | 105 | 120 | 127
  Serogroup A (Month 2) | 4.05 [2.97 to 5.54] | 8.35 [6.14 to 11] | 85.49 [59 to 125] | 7.64 [5.22 to 11] | 22.54 [16 to 32] | 5.18 [3.65 to 7.34]
  Serogroup A (Month 3): number analyzed (Participants) | 172 | 178 | 107 | 105 | 120 | 127
  Serogroup A (Month 3) | 106.70 [82 to 139] | 68.85 [53 to 89] | 52.42 [38 to 72] | 5.31 [3.86 to 7.31] | 8.77 [6.49 to 12] | 78.30 [58 to 105]
  Serogroup A (Month 7): number analyzed (Participants) | 172 | 178 | 107 | 105 | 120 | 127
  Serogroup A (Month 7) | 14.15 [11 to 19] | 11.49 [8.71 to 15] | 9.88 [7.04 to 14] | 165.14 [117 to 233] | 3.25 [2.35 to 4.49] | 140.73 [103 to 193]
  Serogroup A (Month 13): number analyzed (Participants) | 172 | 178 | 107 | 105 | 120 | 127
  Serogroup A (Month 13) | 5.80 [4.30 to 7.82] | 4.64 [3.45 to 6.23] | 5.90 [4.11 to 8.46] | 15.20 [11 to 22] | 168.23 [119 to 238] | 13.32 [9.52 to 19]
  Serogroup C (Month 0): number analyzed (Participants) | 186 | 185 | 122 | 114 | 123 | 130
  Serogroup C (Month 0) | 3.46 [2.76 to 4.33] | 3.38 [2.71 to 4.23] | 3.87 [2.96 to 5.04] | 3.36 [2.56 to 4.40] | 3.80 [2.92 to 4.94] | 2.99 [2.32 to 3.87]
  Serogroup C (Month 2): number analyzed (Participants) | 186 | 185 | 122 | 114 | 123 | 130
  Serogroup C (Month 2) | 9.47 [7.18 to 13] | 31.56 [24 to 42] | 163.28 [118 to 227] | 37.24 [27 to 52] | 54.75 [40 to 76] | 40.29 [29 to 55]
  Serogroup C (Month 3): number analyzed (Participants) | 186 | 185 | 122 | 114 | 123 | 130
  Serogroup C (Month 3) | 41.25 [32 to 52] | 184.05 [145 to 234] | 119.71 [90 to 159] | 31.50 [24 to 42] | 41.15 [31 to 54] | 236.97 [180 to 312]
  Serogroup C (Month 7): number analyzed (Participants) | 186 | 185 | 122 | 114 | 123 | 130
  Serogroup C (Month 7) | 11.03 [8.81 to 14] | 80.70 [65 to 101] | 76.97 [59 to 100] | 260.57 [199 to 342] | 24.59 [19 to 32] | 476.44 [369 to 615]
  Serogroup C (Month 13): number analyzed (Participants) | 186 | 185 | 122 | 114 | 123 | 130
  Serogroup C (Month 13) | 8.45 [6.79 to 11] | 37.45 [30 to 47] | 38.42 [30 to 50] | 57.48 [44 to 75] | 303.63 [235 to 392] | 113.72 [89 to 146]
  Serogroup W (Month 0): number analyzed (Participants) | 162 | 180 | 119 | 108 | 123 | 123
  Serogroup W (Month 0) | 6.43 [4.46 to 9.27] | 4.75 [3.35 to 6.73] | 4.54 [2.98 to 6.90] | 4.29 [2.80 to 6.58] | 4.95 [3.30 to 7.44] | 4.46 [2.97 to 6.69]
  Serogroup W (Month 2): number analyzed (Participants) | 162 | 180 | 119 | 108 | 123 | 123
  Serogroup W (Month 2) | 17.43 [13 to 23] | 50.71 [39 to 66] | 175.57 [128 to 241] | 59.37 [43 to 82] | 94.34 [69 to 128] | 47.54 [35 to 65]
  Serogroup W (Month 3): number analyzed (Participants) | 162 | 180 | 119 | 108 | 123 | 123
  Serogroup W (Month 3) | 138.43 [111 to 173] | 214.70 [173 to 266] | 125.70 [97 to 162] | 59.26 [46 to 77] | 86.66 [68 to 111] | 200.91 [157 to 258]
  Serogroup W (Month 7): number analyzed (Participants) | 162 | 180 | 119 | 108 | 123 | 123
  Serogroup W (Month 7) | 22.53 [18 to 29] | 79.96 [63 to 101] | 74.84 [57 to 99] | 340.85 [256 to 453] | 58.19 [44 to 76] | 270.12 [206 to 354]
  Serogroup W (Month 13): number analyzed (Participants) | 162 | 180 | 119 | 108 | 123 | 123
  Serogroup W (Month 13) | 12.63 [9.86 to 16] | 45.63 [36 to 58] | 46.83 [35 to 62] | 96.43 [72 to 129] | 478.73 [363 to 631] | 95.90 [73 to 126]
  Serogroup Y (Month 0): number analyzed (Participants) | 188 | 180 | 120 | 110 | 127 | 137
  Serogroup Y (Month 0) | 1.72 [1.41 to 2.10] | 1.40 [1.14 to 1.71] | 1.68 [1.32 to 2.13] | 1.24 [0.97 to 1.59] | 1.79 [1.42 to 2.25] | 1.34 [1.07 to 1.67]
  Serogroup Y (Month 2): number analyzed (Participants) | 188 | 180 | 120 | 110 | 127 | 137
  Serogroup Y (Month 2) | 2.36 [1.72 to 3.23] | 19.43 [14 to 27] | 63.45 [44 to 93] | 16.41 [11 to 24] | 27.00 [19 to 39] | 19.82 [14 to 28]
  Serogroup Y (Month 3): number analyzed (Participants) | 188 | 180 | 120 | 110 | 127 | 137
  Serogroup Y (Month 3) | 3.12 [2.34 to 4.17] | 90.61 [68 to 121] | 42.97 [30 to 61] | 15.95 [11 to 23] | 18.76 [13 to 26] | 97.12 [70 to 134]
  Serogroup Y (Month 7): number analyzed (Participants) | 188 | 180 | 120 | 110 | 127 | 137
  Serogroup Y (Month 7) | 2.44 [1.87 to 3.17] | 34.27 [26 to 45] | 27.86 [20 to 38] | 152.73 [111 to 211] | 14.29 [11 to 19] | 180.33 [135 to 242]
  Serogroup Y (Month 13): number analyzed (Participants) | 188 | 180 | 120 | 110 | 127 | 137
  Serogroup Y (Month 13) | 2.28 [1.75 to 2.96] | 18.13 [14 to 24] | 15.19 [11 to 21] | 42.14 [31 to 58] | 231.39 [171 to 313] | 53.78 [40 to 72]

10. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥LLQ, ≥5, ≥8, ≥16, ≥32, ≥64, ≥128 Against NZ98/254 B Strain for All Schedules.
Description: The kinetic of immune response (at Months 0, 2, 3, 7 and 13) following different vaccination schedules as measured by the percentages of subjects with hSBA titers ≥LLQ, ≥5, ≥8, ≥16, ≥32, ≥64, ≥128 against NZ98/254 B strain was assessed.
Time Frame: At Month 0, Month 2, Month 3, Month 7 and Month 13.
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB_0_2 Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group | ABCWY_0_2_6 Group
Number analyzed (Participants) | 188 | 185 | 120 | 112 | 126 | 134
Percentages of subjects
  NZ98/254 Strain (At Month 0) ≥ LLQ (8.2) | 7 [3.73 to 11.53] | 6 [3.40 to 11.06] | 6 [2.38 to 11.65] | 5 [1.99 to 11.30] | 4 [1.30 to 9.02] | 2 [0.46 to 6.40]
  NZ98/254 Strain (At Month 0) ≥ 5 | 9 [4.94 to 13.45] | 7 [3.79 to 11.72] | 7 [2.92 to 12.71] | 5 [1.99 to 11.30] | 6 [2.26 to 11.11] | 3 [0.82 to 7.47]
  NZ98/254 Strain (At Month 0) ≥ 8 | 7 [4.13 to 12.18] | 6 [3.40 to 11.06] | 6 [2.38 to 11.65] | 5 [1.99 to 11.30] | 4 [1.30 to 9.02] | 2 [0.46 to 6.40]
  NZ98/254 Strain (At Month 0) ≥ 16 | 4 [1.85 to 8.21] | 5 [2.62 to 9.72] | 4 [1.37 to 9.46] | 4 [0.98 to 8.89] | 2 [0.19 to 5.62] | 1 [0.02 to 4.09]
  NZ98/254 Strain (At Month 0) ≥ 32 | 2 [0.33 to 4.59] | 3 [0.88 to 6.19] | 3 [0.52 to 7.13] | 1 [0.02 to 4.87] | 0 [0 to 2.89] | 0 [0 to 2.72]
  NZ98/254 Strain (At Month 0) ≥ 64 | 0 [0 to 1.94] | 3 [0.34 to 4.67] | 0 [0 to 3.03] | 1 [0.02 to 4.87] | 0 [0 to 2.89] | 0 [0 to 2.72]
  NZ98/254 Strain (At Month 0) ≥ 128 | 0 [0 to 1.94] | 0 [0 to 1.97] | 0 [0 to 3.03] | 0 [0 to 3.24] | 0 [0 to 2.89] | 0 [0 to 2.72]
  NZ98/254 Strain (At Month 2) ≥ LLQ (8.2) | 23 [17.55 to 30.12] | 20 [14.49 to 26.50] | 43 [33.53 to 51.85] | 17 [10.53 to 25.22] | 27 [19.47 to 35.62] | 18 [11.83 to 25.47]
  NZ98/254 Strain (At Month 2) ≥ 5 | 29 [22.86 to 36.32] | 24 [18.33 to 31.16] | 58 [48.98 to 67.26] | 18 [11.26 to 26.22] | 36 [27.38 to 44.74] | 20 [13.72 to 27.95]
  NZ98/254 Strain (At Month 2) ≥ 8 | 23 [17.55 to 30.12] | 20 [14.49 to 26.50] | 43 [33.53 to 51.85] | 17 [10.53 to 25.22] | 28 [20.17 to 36.46] | 18 [11.83 to 25.47]
  NZ98/254 Strain (At Month 2) ≥ 16 | 19 [13.79 to 25.51] | 15 [10.30 to 21.13] | 28 [20.49 to 37.28] | 11 [5.66 to 17.97] | 23 [15.99 to 31.35] | 13 [7.57 to 19.53]
  NZ98/254 Strain (At Month 2) ≥ 32 | 15 [10.13 to 20.80] | 10 [5.87 to 14.94] | 20 [13.25 to 28.28] | 9 [4.36 to 15.81] | 17 [10.62 to 24.34] | 7 [3.64 to 13.30]
  NZ98/254 Strain (At Month 2) ≥ 64 | 9 [4.94 to 13.45] | 7 [3.79 to 11.72] | 12 [6.53 to 18.80] | 4 [0.98 to 8.89] | 13 [7.44 to 19.80] | 2 [0.46 to 6.40]
  NZ98/254 Strain (At Month 2) ≥ 128 | 2 [0.33 to 4.59] | 5 [2.25 to 9.03] | 5 [1.86 to 10.57] | 3 [0.56 to 7.63] | 6 [2.78 to 12.13] | 1 [0.18 to 5.29]
  NZ98/254 Strain (At Month 3) ≥ LLQ (8.2) | 88 [82.82 to 92.52] | 61 [53.65 to 68.15] | 30 [21.98 to 39.04] | 14 [8.39 to 22.16] | 20 [13.27 to 27.88] | 68 [59.30 to 75.71]
  NZ98/254 Strain (At Month 3) ≥ 5 | 94 [89.12 to 96.66] | 76 [68.84 to 81.67] | 38 [29.61 to 47.65] | 17 [10.53 to 25.22] | 27 [19.47 to 35.62] | 78 [70.42 to 85.00]
  NZ98/254 Strain (At Month 3) ≥ 8 | 88 [82.82 to 92.52] | 63 [55.30 to 69.69] | 30 [21.98 to 39.04] | 14 [8.39 to 22.16] | 21 [13.94 to 28.75] | 69 [60.86 to 77.07]
  NZ98/254 Strain (At Month 3) ≥ 16 | 74 [67.05 to 80.05] | 44 [37.04 to 51.79] | 18 [11.86 to 26.43] | 11 [5.66 to 17.97] | 14 [8.69 to 21.63] | 46 [37.62 to 55.08]
  NZ98/254 Strain (At Month 3) ≥ 32 | 50 [42.64 to 57.36] | 23 [17.36 to 30.00] | 13 [7.17 to 19.78] | 5 [1.99 to 11.30] | 10 [5.02 to 16.05] | 19 [12.45 to 26.30]
  NZ98/254 Strain (At Month 3) ≥ 64 | 29 [22.86 to 36.32] | 12 [7.60 to 17.45] | 6 [2.38 to 11.65] | 4 [0.98 to 8.89] | 6 [2.26 to 11.11] | 14 [8.76 to 21.25]
  NZ98/254 Strain (At Month 3) ≥ 128 | 12 [7.48 to 17.18] | 6 [3.40 to 11.06] | 4 [1.37 to 9.46] | 2 [0.22 to 6.30] | 4 [1.30 to 9.02] | 4 [1.66 to 9.49]
  NZ98/254 Strain (At Month 7) ≥ LLQ (8.2) | 27 [20.43 to 33.52] | 19 [14.02 to 25.91] | 14 [8.47 to 21.71] | 63 [53.76 to 72.29] | 13 [7.44 to 19.80] | 72 [64.00 to 79.76]
  NZ98/254 Strain (At Month 7) ≥ 5 | 33 [26.31 to 40.19] | 27 [20.77 to 34.03] | 18 [11.86 to 26.43] | 80 [71.78 to 87.26] | 17 [11.28 to 25.23] | 82 [74.53 to 88.17]
  NZ98/254 Strain (At Month 7) ≥ 8 | 27 [20.43 to 33.52] | 20 [14.49 to 26.50] | 14 [8.47 to 21.71] | 69 [59.30 to 77.17] | 13 [7.44 to 19.80] | 74 [65.59 to 81.08]
  NZ98/254 Strain (At Month 7) ≥ 16 | 21 [15.19 to 27.25] | 14 [9.39 to 19.91] | 12 [6.53 to 18.80] | 46 [36.10 to 55.22] | 10 [5.02 to 16.05] | 55 [46.40 to 63.82]
  NZ98/254 Strain (At Month 7) ≥ 32 | 12 [7.92 to 17.79] | 10 [6.30 to 15.57] | 9 [4.67 to 15.81] | 26 [18.08 to 35.03] | 4 [1.30 to 9.02] | 34 [25.66 to 42.25]
  NZ98/254 Strain (At Month 7) ≥ 64 | 6 [3.34 to 10.88] | 6 [3.40 to 11.06] | 6 [2.38 to 11.65] | 13 [7.69 to 21.13] | 2 [0.19 to 5.62] | 16 [10.58 to 23.80]
  NZ98/254 Strain (At Month 7) ≥ 128 | 2 [0.33 to 4.59] | 4 [1.53 to 7.64] | 5 [1.86 to 10.57] | 7 [3.13 to 13.59] | 1 [0.02 to 4.34] | 5 [2.13 to 10.47]
  NZ98/254 Strain (At Month 13) ≥ LLQ (8.2) | 21 [15.19 to 27.25] | 16 [11.22 to 22.33] | 15 [9.14 to 22.67] | 18 [11.26 to 26.22] | 73 [64.38 to 80.53] | 19 [13.08 to 27.12]
  NZ98/254 Strain (At Month 13) ≥ 5 | 27 [20.43 to 33.52] | 19 [14.02 to 25.91] | 16 [9.81 to 23.62] | 28 [19.64 to 36.93] | 85 [77.46 to 90.67] | 25 [17.60 to 32.81]
  NZ98/254 Strain (At Month 13) ≥ 8 | 21 [15.19 to 27.25] | 16 [11.22 to 22.33] | 15 [9.14 to 22.67] | 18 [11.26 to 26.22] | 74 [65.23 to 81.24] | 19 [13.08 to 27.12]
  NZ98/254 Strain (At Month 13) ≥ 16 | 15 [10.13 to 20.80] | 12 [8.05 to 18.07] | 8 [4.07 to 14.79] | 12 [6.33 to 19.03] | 49 [40.19 to 58.26] | 14 [8.76 to 21.25]
  NZ98/254 Strain (At Month 13) ≥ 32 | 7 [4.13 to 12.18] | 7 [3.79 to 11.72] | 8 [3.49 to 13.76] | 8 [3.74 to 14.71] | 30 [22.31 to 38.97] | 4 [1.66 to 9.49]
  NZ98/254 Strain (At Month 13) ≥ 64 | 3 [0.87 to 6.10] | 5 [2.25 to 9.03] | 5 [1.86 to 10.57] | 5 [1.99 to 11.30] | 13 [8.06 to 20.72] | 3 [0.82 to 7.47]
  NZ98/254 Strain (At Month 13) ≥ 128 | 2 [0.33 to 4.59] | 3 [0.88 to 6.19] | 3 [0.92 to 8.31] | 3 [0.56 to 7.63] | 6 [2.78 to 12.13] | 2 [0.46 to 6.40]

11. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥LLQ, ≥5, ≥8, ≥16, ≥32, ≥64, ≥128 Against M14459 B Strain for All Schedules.
Description: The kinetic of immune response (at Months 0, 2, 3, 7 and 13) following different vaccination schedules as measured by the percentages of subjects with hSBA titers ≥LLQ, ≥5, ≥8, ≥16, ≥32, ≥64, ≥128 against M14459 B strain was assessed.
Time Frame: At Month 0, Month 2, Month 3, Month 7 and Month 13.
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB_0_2 Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group | ABCWY_0_2_6 Group
Number analyzed (Participants) | 184 | 179 | 112 | 108 | 123 | 134
Percentages of subjects
  M14459 Strain (At Month 0) ≥ LLQ (8.0) | 7 [3.41 to 11.11] | 5 [2.32 to 9.33] | 6 [2.55 to 12.45] | 4 [1.02 to 9.21] | 7 [2.85 to 12.41] | 2 [0.46 to 6.40]
  M14459 Strain (At Month 0) ≥ 5 | 12 [7.65 to 17.54] | 7 [3.92 to 12.10] | 6 [2.55 to 12.45] | 6 [2.65 to 12.90] | 11 [6.36 to 18.36] | 4 [1.22 to 8.49]
  M14459 Strain (At Month 0) ≥ 8 | 7 [3.41 to 11.11] | 5 [2.32 to 9.33] | 6 [2.55 to 12.45] | 4 [1.02 to 9.21] | 7 [2.85 to 12.41] | 2 [0.46 to 6.40]
  M14459 Strain (At Month 0) ≥ 16 | 3 [0.89 to 6.23] | 2 [0.35 to 4.82] | 2 [0.22 to 6.30] | 3 [0.58 to 7.90] | 2 [0.51 to 6.96] | 1 [0.18 to 5.29]
  M14459 Strain (At Month 0) ≥ 32 | 2 [0.34 to 4.69] | 0 [0 to 2.04] | 1 [0.02 to 4.87] | 1 [0.02 to 5.05] | 0 [0 to 2.95] | 1 [0.02 to 4.09]
  M14459 Strain (At Month 0) ≥ 64 | 1 [0.13 to 3.87] | 0 [0 to 2.04] | 0 [0 to 3.24] | 0 [0 to 3.36] | 0 [0 to 2.95] | 1 [0.02 to 4.09]
  M14459 Strain (At Month 0) ≥ 128 | 0 [0 to 1.98] | 0 [0 to 2.04] | 0 [0 to 3.24] | 0 [0 to 3.36] | 0 [0 to 2.95] | 0 [0 to 2.72]
  M14459 Strain (At Month 2) ≥ LLQ (8.0) | 28 [21.88 to 35.35] | 24 [17.96 to 30.96] | 61 [51.04 to 69.81] | 17 [10.19 to 25.06] | 34 [25.84 to 43.24] | 17 [11.20 to 24.63]
  M14459 Strain (At Month 2) ≥ 5 | 38 [30.49 to 44.92] | 30 [23.03 to 36.88] | 75 [65.93 to 82.70] | 26 [17.97 to 35.25] | 42 [33.42 to 51.51] | 22 [15.64 to 30.39]
  M14459 Strain (At Month 2) ≥ 8 | 28 [21.88 to 35.35] | 24 [17.96 to 30.96] | 61 [51.04 to 69.81] | 17 [10.19 to 25.06] | 34 [25.84 to 43.24] | 17 [11.20 to 24.63]
  M14459 Strain (At Month 2) ≥ 16 | 17 [11.74 to 23.05] | 13 [8.32 to 18.65] | 34 [25.25 to 43.48] | 11 [5.87 to 18.06] | 25 [17.81 to 33.83] | 12 [6.98 to 18.67]
  M14459 Strain (At Month 2) ≥ 32 | 9 [5.05 to 13.74] | 6 [3.11 to 10.73] | 19 [12.00 to 27.22] | 6 [2.07 to 11.70] | 13 [7.62 to 20.26] | 5 [2.13 to 10.47]
  M14459 Strain (At Month 2) ≥ 64 | 4 [1.90 to 8.39] | 2 [0.61 to 5.62] | 4 [0.98 to 8.89] | 2 [0.23 to 6.53] | 8 [3.97 to 14.44] | 2 [0.46 to 6.40]
  M14459 Strain (At Month 2) ≥ 128 | 1 [0.01 to 2.99] | 2 [0.35 to 4.82] | 2 [0.22 to 6.30] | 1 [0.02 to 5.05] | 5 [1.81 to 10.32] | 1 [0.18 to 5.29]
  M14459 Strain (At Month 3) ≥ LLQ (8.0) | 82 [75.75 to 87.32] | 68 [60.21 to 74.39] | 44 [34.39 to 53.44] | 16 [9.45 to 24.00] | 28 [20.69 to 37.29] | 73 [64.80 to 80.42]
  M14459 Strain (At Month 3) ≥ 5 | 84 [78.16 to 89.18] | 74 [66.66 to 80.03] | 54 [44.78 to 63.90] | 20 [13.23 to 29.20] | 35 [26.58 to 44.08] | 80 [72.05 to 86.28]
  M14459 Strain (At Month 3) ≥ 8 | 82 [75.75 to 87.32] | 68 [60.21 to 74.39] | 44 [34.39 to 53.44] | 16 [9.45 to 24.00] | 28 [20.69 to 37.29] | 73 [64.80 to 80.42]
  M14459 Strain (At Month 3) ≥ 16 | 66 [58.98 to 73.09] | 51 [43.83 to 58.92] | 24 [16.53 to 33.10] | 9 [4.53 to 16.37] | 18 [11.56 to 25.82] | 51 [41.98 to 59.48]
  M14459 Strain (At Month 3) ≥ 32 | 39 [32.03 to 46.58] | 30 [23.54 to 37.46] | 6 [2.55 to 12.45] | 4 [1.02 to 9.21] | 9 [4.55 to 15.44] | 28 [20.91 to 36.79]
  M14459 Strain (At Month 3) ≥ 64 | 18 [12.68 to 24.25] | 11 [6.51 to 16.08] | 3 [0.56 to 7.63] | 1 [0.02 to 5.05] | 4 [1.33 to 9.23] | 10 [5.83 to 16.91]
  M14459 Strain (At Month 3) ≥ 128 | 7 [3.41 to 11.11] | 2 [0.61 to 5.62] | 2 [0.22 to 6.30] | 1 [0.02 to 5.05] | 3 [0.89 to 8.12] | 3 [0.82 to 7.47]
  M14459 Strain (At Month 7) ≥ LLQ (8.0) | 34 [26.91 to 41.02] | 30 [23.03 to 36.88] | 17 [10.53 to 25.22] | 86 [78.13 to 92.01] | 15 [9.56 to 23.07] | 89 [82.21 to 93.60]
  M14459 Strain (At Month 7) ≥ 5 | 44 [36.73 to 51.51] | 35 [28.22 to 42.67] | 21 [14.24 to 30.19] | 92 [84.77 to 96.12] | 20 [12.92 to 27.63] | 93 [87.63 to 96.88]
  M14459 Strain (At Month 7) ≥ 8 | 34 [26.91 to 41.02] | 30 [23.03 to 36.88] | 17 [10.53 to 25.22] | 86 [78.13 to 92.01] | 15 [9.56 to 23.07] | 89 [82.21 to 93.60]
  M14459 Strain (At Month 7) ≥ 16 | 19 [13.62 to 25.45] | 14 [9.25 to 19.92] | 10 [5.01 to 16.89] | 69 [59.84 to 77.95] | 8 [3.97 to 14.44] | 72 [63.21 to 79.09]
  M14459 Strain (At Month 7) ≥ 32 | 11 [7.21 to 16.92] | 7 [3.51 to 11.42] | 5 [1.99 to 11.30] | 50 [40.22 to 59.78] | 6 [2.32 to 11.37] | 49 [40.52 to 58.02]
  M14459 Strain (At Month 7) ≥ 64 | 3 [1.21 to 6.96] | 4 [1.59 to 7.89] | 3 [0.56 to 7.63] | 23 [15.57 to 32.25] | 4 [1.33 to 9.23] | 22 [15.64 to 30.39]
  M14459 Strain (At Month 7) ≥ 128 | 0 [0 to 1.98] | 1 [0.01 to 3.07] | 1 [0.02 to 4.87] | 10 [5.20 to 17.49] | 2 [0.20 to 5.75] | 7 [3.12 to 12.37]
  M14459 Strain (At Month 13) ≥ LLQ (8.0) | 23 [17.46 to 30.16] | 20 [14.01 to 26.13] | 13 [7.01 to 20.08] | 23 [15.57 to 32.25] | 89 [81.64 to 93.64] | 27 [19.58 to 35.20]
  M14459 Strain (At Month 13) ≥ 5 | 30 [23.88 to 37.63] | 26 [19.47 to 32.75] | 20 [12.74 to 28.22] | 37 [27.94 to 46.86] | 93 [86.56 to 96.60] | 38 [29.82 to 46.84]
  M14459 Strain (At Month 13) ≥ 8 | 23 [17.46 to 30.16] | 20 [14.01 to 26.13] | 13 [7.01 to 20.08] | 23 [15.57 to 32.25] | 89 [81.64 to 93.64] | 27 [19.58 to 35.20]
  M14459 Strain (At Month 13) ≥ 16 | 15 [9.90 to 20.63] | 9 [5.63 to 14.77] | 7 [3.13 to 13.59] | 13 [7.27 to 20.79] | 76 [67.05 to 82.90] | 13 [7.57 to 19.53]
  M14459 Strain (At Month 13) ≥ 32 | 5 [2.64 to 9.77] | 4 [1.95 to 8.62] | 4 [0.98 to 8.89] | 7 [3.25 to 14.07] | 54 [45.25 to 63.47] | 6 [2.61 to 11.42]
  M14459 Strain (At Month 13) ≥ 64 | 2 [0.34 to 4.69] | 2 [0.61 to 5.62] | 3 [0.56 to 7.63] | 1 [0.02 to 5.05] | 29 [21.41 to 38.15] | 1 [0.18 to 5.29]
  M14459 Strain (At Month 13) ≥ 128 | 0 [0 to 1.98] | 1 [0.01 to 3.07] | 2 [0.22 to 6.30] | 1 [0.02 to 5.05] | 11 [5.75 to 17.40] | 1 [0.02 to 4.09]

12. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥LLQ, ≥5, ≥8, ≥16, ≥32, ≥64, ≥128 Against M07-0241084 B Strain for All Schedules.
Description: The kinetic of immune response (at Months 0, 2, 3, 7 and 13) following different vaccination schedules as measured by the percentages of subjects with hSBA titers ≥LLQ, ≥5, ≥8, ≥16, ≥32, ≥64, ≥128 against M07-0241084 B strain was assessed.
Time Frame: At Month 0, Month 2, Month 3, Month 7 and Month 13.
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB_0_2 Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group | ABCWY_0_2_6 Group
Number analyzed (Participants) | 188 | 176 | 117 | 113 | 121 | 128
Percentages of subjects
  M07-0241084 Strain (At Month 0) ≥ LLQ (8.9) | 21 [15.19 to 27.25] | 18 [12.78 to 24.69] | 17 [10.77 to 25.16] | 14 [8.32 to 21.97] | 21 [14.54 to 29.88] | 19 [12.40 to 26.60]
  M07-0241084 Strain (At Month 0) ≥ 5 | 30 [23.35 to 36.87] | 28 [21.36 to 35.08] | 25 [17.27 to 33.62] | 27 [19.46 to 36.63] | 30 [21.79 to 38.74] | 21 [14.38 to 29.19]
  M07-0241084 Strain (At Month 0) ≥ 8 | 22 [16.13 to 28.40] | 20 [14.26 to 26.56] | 18 [11.47 to 26.12] | 19 [12.62 to 27.98] | 24 [16.68 to 32.57] | 20 [13.72 to 28.33]
  M07-0241084 Strain (At Month 0) ≥ 16 | 13 [8.79 to 19.00] | 14 [9.41 to 20.25] | 12 [6.70 to 19.26] | 6 [2.53 to 12.35] | 16 [9.73 to 23.43] | 15 [9.18 to 22.21]
  M07-0241084 Strain (At Month 0) ≥ 32 | 8 [4.53 to 12.82] | 6 [3.16 to 10.91] | 7 [3.00 to 13.03] | 4 [0.97 to 8.82] | 9 [4.63 to 15.68] | 6 [2.74 to 11.94]
  M07-0241084 Strain (At Month 0) ≥ 64 | 3 [1.18 to 6.82] | 2 [0.35 to 4.90] | 3 [0.53 to 7.31] | 2 [0.22 to 6.25] | 3 [0.91 to 8.25] | 3 [0.86 to 7.81]
  M07-0241084 Strain (At Month 0) ≥ 128 | 0 [0 to 1.94] | 0 [0 to 2.07] | 0 [0 to 3.10] | 2 [0.22 to 6.25] | 1 [0.02 to 4.52] | 1 [0.02 to 4.28]
  M07-0241084 Strain (At Month 2) ≥ LLQ (8.9) | 38 [30.81 to 45.11] | 29 [22.40 to 36.28] | 37 [28.03 to 46.16] | 28 [20.24 to 37.57] | 39 [30.12 to 48.13] | 30 [22.65 to 39.22]
  M07-0241084 Strain (At Month 2) ≥ 5 | 47 [40.03 to 54.74] | 43 [35.75 to 50.85] | 54 [44.39 to 63.10] | 40 [30.73 to 49.46] | 54 [44.43 to 62.83] | 41 [32.04 to 49.66]
  M07-0241084 Strain (At Month 2) ≥ 8 | 42 [34.88 to 49.42] | 32 [25.54 to 39.84] | 43 [33.63 to 52.21] | 31 [22.61 to 40.36] | 43 [34.01 to 52.29] | 35 [26.93 to 44.09]
  M07-0241084 Strain (At Month 2) ≥ 16 | 31 [24.33 to 37.98] | 22 [16.26 to 29.02] | 29 [21.04 to 38.17] | 16 [9.72 to 24.00] | 30 [21.79 to 38.74] | 19 [12.40 to 26.60]
  M07-0241084 Strain (At Month 2) ≥ 32 | 20 [14.72 to 26.67] | 15 [10.36 to 21.53] | 17 [10.77 to 25.16] | 7 [3.11 to 13.47] | 19 [12.45 to 27.14] | 9 [4.37 to 14.86]
  M07-0241084 Strain (At Month 2) ≥ 64 | 10 [5.77 to 14.71] | 7 [3.99 to 12.30] | 9 [4.17 to 15.16] | 2 [0.22 to 6.25] | 9 [4.63 to 15.68] | 5 [1.74 to 9.92]
  M07-0241084 Strain (At Month 2) ≥ 128 | 3 [1.18 to 6.82] | 2 [0.35 to 4.90] | 3 [0.53 to 7.31] | 1 [0.02 to 4.83] | 5 [1.84 to 10.48] | 0 [0 to 2.84]
  M07-0241084 Strain (At Month 3) ≥ LLQ (8.9) | 66 [59.26 to 73.19] | 47 [39.60 to 54.81] | 28 [20.28 to 37.27] | 28 [20.24 to 37.57] | 30 [21.79 to 38.74] | 53 [44.11 to 62.00]
  M07-0241084 Strain (At Month 3) ≥ 5 | 79 [72.75 to 84.81] | 69 [61.94 to 76.04] | 43 [33.63 to 52.21] | 40 [30.73 to 49.46] | 43 [34.01 to 52.29] | 62 [52.72 to 70.17]
  M07-0241084 Strain (At Month 3) ≥ 8 | 69 [62.02 to 75.67] | 55 [47.45 to 62.60] | 34 [25.67 to 43.53] | 31 [22.61 to 40.36] | 34 [25.53 to 43.05] | 56 [47.21 to 65.00]
  M07-0241084 Strain (At Month 3) ≥ 16 | 52 [44.74 to 59.45] | 33 [26.07 to 40.43] | 21 [14.33 to 29.91] | 12 [6.27 to 18.87] | 21 [14.54 to 29.88] | 40 [31.30 to 48.87]
  M07-0241084 Strain (At Month 3) ≥ 32 | 33 [26.31 to 40.19] | 18 [12.78 to 24.69] | 15 [9.38 to 23.22] | 5 [1.97 to 11.20] | 15 [9.06 to 22.49] | 23 [15.73 to 30.89]
  M07-0241084 Strain (At Month 3) ≥ 64 | 18 [12.40 to 23.76] | 11 [7.08 to 17.00] | 5 [1.90 to 10.83] | 1 [0.02 to 4.83] | 4 [1.36 to 9.38] | 13 [7.32 to 19.50]
  M07-0241084 Strain (At Month 3) ≥ 128 | 5 [2.21 to 8.89] | 3 [0.93 to 6.50] | 3 [0.53 to 7.31] | 1 [0.02 to 4.83] | 2 [0.51 to 7.07] | 2 [0.49 to 6.70]
  M07-0241084 Strain (At Month 7) ≥ LLQ (8.9) | 40 [32.84 to 47.27] | 30 [22.92 to 36.88] | 26 [18.02 to 34.54] | 66 [56.88 to 74.99] | 26 [18.12 to 34.35] | 70 [61.60 to 78.06]
  M07-0241084 Strain (At Month 7) ≥ 5 | 50 [42.64 to 57.36] | 44 [36.30 to 51.42] | 32 [24.11 to 41.76] | 83 [74.99 to 89.56] | 36 [27.81 to 45.60] | 80 [72.53 to 86.94]
  M07-0241084 Strain (At Month 7) ≥ 8 | 42 [34.88 to 49.42] | 32 [25.54 to 39.84] | 27 [19.52 to 36.36] | 70 [60.57 to 78.18] | 28 [20.31 to 36.99] | 77 [68.26 to 83.59]
  M07-0241084 Strain (At Month 7) ≥ 16 | 29 [22.37 to 35.76] | 24 [18.28 to 31.47] | 19 [12.18 to 27.07] | 53 [43.48 to 62.55] | 18 [11.76 to 26.22] | 58 [48.77 to 66.49]
  M07-0241084 Strain (At Month 7) ≥ 32 | 21 [15.19 to 27.25] | 14 [8.94 to 19.61] | 9 [4.79 to 16.20] | 28 [20.24 to 37.57] | 8 [4.03 to 14.67] | 34 [25.49 to 42.48]
  M07-0241084 Strain (At Month 7) ≥ 64 | 6 [2.96 to 10.23] | 8 [4.42 to 12.99] | 6 [2.44 to 11.94] | 10 [4.96 to 16.75] | 4 [1.36 to 9.38] | 17 [11.10 to 24.86]
  M07-0241084 Strain (At Month 7) ≥ 128 | 1 [0.01 to 2.93] | 2 [0.35 to 4.90] | 1 [0.02 to 4.67] | 3 [0.55 to 7.56] | 1 [0.02 to 4.52] | 4 [1.28 to 8.88]
  M07-0241084 Strain (At Month 13) ≥ LLQ (8.9) | 34 [26.81 to 40.74] | 27 [20.84 to 34.48] | 23 [15.79 to 31.77] | 34 [25.01 to 43.12] | 69 [59.53 to 76.73] | 37 [28.38 to 45.69]
  M07-0241084 Strain (At Month 13) ≥ 5 | 46 [38.48 to 53.15] | 39 [31.95 to 46.83] | 36 [27.24 to 45.29] | 57 [46.99 to 65.93] | 82 [73.78 to 88.24] | 51 [41.80 to 59.72]
  M07-0241084 Strain (At Month 13) ≥ 8 | 37 [29.81 to 44.02] | 34 [26.60 to 41.01] | 27 [19.52 to 36.36] | 39 [29.91 to 48.56] | 74 [64.76 to 81.16] | 42 [33.51 to 51.23]
  M07-0241084 Strain (At Month 13) ≥ 16 | 26 [19.46 to 32.39] | 23 [16.76 to 29.64] | 17 [10.77 to 25.16] | 19 [12.62 to 27.98] | 55 [45.24 to 63.62] | 26 [18.46 to 34.26]
  M07-0241084 Strain (At Month 13) ≥ 32 | 16 [11.03 to 21.99] | 13 [8.47 to 18.96] | 11 [6.05 to 18.25] | 12 [6.27 to 18.87] | 35 [26.29 to 43.90] | 12 [6.71 to 18.59]
  M07-0241084 Strain (At Month 13) ≥ 64 | 6 [3.34 to 10.88] | 3 [1.26 to 7.27] | 4 [1.40 to 9.69] | 5 [1.97 to 11.20] | 20 [13.14 to 28.06] | 5 [1.74 to 9.92]
  M07-0241084 Strain (At Month 13) ≥ 128 | 2 [0.58 to 5.36] | 1 [0.01 to 3.12] | 2 [0.21 to 6.04] | 1 [0.02 to 4.83] | 9 [4.63 to 15.68] | 1 [0.02 to 4.28]

13. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥LLQ, ≥5, ≥8, ≥16, ≥32, ≥64, ≥128 Against 96217 B Strain for All Schedules.
Description: The kinetic of immune response (at Months 0, 2, 3, 7 and 13) following different vaccination schedules as measured by the percentages of subjects with hSBA titers ≥LLQ, ≥5, ≥8, ≥16, ≥32, ≥64, ≥128 against 96217 B strain was assessed.
Time Frame: At Month 0, Month 2, Month 3, Month 7 and Month 13.
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB_0_2 Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group | ABCWY_0_2_6 Group
Number analyzed (Participants) | 186 | 178 | 120 | 112 | 128 | 121
Percentages of subjects
  96217 Strain (At Month 0) ≥ LLQ (8.6) | 23 [17.26 to 29.85] | 29 [22.14 to 35.89] | 29 [21.23 to 38.16] | 28 [19.64 to 36.93] | 25 [17.77 to 33.42] | 27 [19.57 to 36.12]
  96217 Strain (At Month 0) ≥ 5 | 26 [19.68 to 32.72] | 35 [28.38 to 42.90] | 35 [26.52 to 44.24] | 29 [21.23 to 38.82] | 35 [26.93 to 44.09] | 29 [21.05 to 37.87]
  96217 Strain (At Month 0) ≥ 8 | 24 [18.23 to 31.00] | 30 [23.68 to 37.66] | 31 [22.73 to 39.91] | 28 [19.64 to 36.93] | 25 [17.77 to 33.42] | 27 [19.57 to 36.12]
  96217 Strain (At Month 0) ≥ 16 | 16 [11.15 to 22.22] | 17 [11.67 to 23.18] | 22 [14.67 to 30.11] | 19 [12.00 to 27.22] | 18 [11.74 to 25.73] | 16 [9.73 to 23.43]
  96217 Strain (At Month 0) ≥ 32 | 6 [3.38 to 11.00] | 8 [4.37 to 12.84] | 8 [4.07 to 14.79] | 4 [1.47 to 10.11] | 8 [3.81 to 13.90] | 7 [2.90 to 12.61]
  96217 Strain (At Month 0) ≥ 64 | 2 [0.33 to 4.64] | 2 [0.62 to 5.65] | 3 [0.52 to 7.13] | 0 [0 to 3.24] | 2 [0.49 to 6.70] | 5 [1.84 to 10.48]
  96217 Strain (At Month 0) ≥ 128 | 1 [0.01 to 2.96] | 1 [0.14 to 4.00] | 0 [0 to 3.03] | 0 [0 to 3.24] | 1 [0.02 to 4.28] | 2 [0.20 to 5.84]
  96217 Strain (At Month 2) ≥ LLQ (8.6) | 69 [61.63 to 75.39] | 64 [56.53 to 71.09] | 97 [91.69 to 99.08] | 62 [51.94 to 70.64] | 58 [48.77 to 66.49] | 50 [40.37 to 58.82]
  96217 Strain (At Month 2) ≥ 5 | 75 [68.42 to 81.29] | 67 [60.00 to 74.24] | 97 [91.69 to 99.08] | 66 [56.52 to 74.75] | 66 [56.72 to 73.79] | 53 [43.61 to 62.03]
  96217 Strain (At Month 2) ≥ 8 | 70 [63.31 to 76.88] | 64 [56.53 to 71.09] | 97 [91.69 to 99.08] | 63 [53.76 to 72.29] | 59 [50.34 to 67.96] | 51 [41.99 to 60.43]
  96217 Strain (At Month 2) ≥ 16 | 48 [41.01 to 55.81] | 48 [40.78 to 55.91] | 94 [88.35 to 97.62] | 48 [38.67 to 57.85] | 42 [33.51 to 51.23] | 39 [30.12 to 48.13]
  96217 Strain (At Month 2) ≥ 32 | 27 [21.15 to 34.43] | 21 [15.57 to 28.10] | 84 [76.38 to 90.19] | 20 [12.74 to 28.22] | 26 [18.46 to 34.26] | 24 [16.68 to 32.57]
  96217 Strain (At Month 2) ≥ 64 | 11 [6.69 to 16.12] | 15 [9.77 to 20.67] | 73 [63.60 to 80.25] | 9 [4.36 to 15.81] | 14 [8.55 to 21.31] | 12 [6.47 to 18.65]
  96217 Strain (At Month 2) ≥ 128 | 7 [3.77 to 11.66] | 4 [1.96 to 8.66] | 45 [35.91 to 54.35] | 4 [1.47 to 10.11] | 9 [4.94 to 15.80] | 7 [3.46 to 13.65]
  96217 Strain (At Month 3) ≥ LLQ (8.6) | 99 [97.04 to 99.99] | 97 [92.81 to 98.75] | 94 [88.35 to 97.62] | 58 [48.34 to 67.30] | 47 [38.00 to 55.89] | 97 [91.75 to 99.09]
  96217 Strain (At Month 3) ≥ 5 | 99 [97.04 to 99.99] | 97 [93.57 to 99.08] | 96 [90.54 to 98.53] | 61 [51.04 to 69.81] | 56 [47.21 to 65.00] | 98 [92.93 to 99.49]
  96217 Strain (At Month 3) ≥ 8 | 99 [97.04 to 99.99] | 97 [92.81 to 98.75] | 95 [89.43 to 98.14] | 58 [48.34 to 67.30] | 52 [43.34 to 61.24] | 97 [91.75 to 99.09]
  96217 Strain (At Month 3) ≥ 16 | 99 [97.04 to 99.99] | 95 [90.62 to 97.66] | 91 [84.19 to 95.33] | 40 [31.03 to 49.86] | 36 [27.65 to 44.89] | 95 [89.52 to 98.16]
  96217 Strain (At Month 3) ≥ 32 | 98 [95.36 to 99.67] | 89 [83.83 to 93.45] | 83 [75.44 to 89.51] | 21 [13.49 to 29.20] | 23 [15.73 to 30.89] | 92 [85.33 to 95.97]
  96217 Strain (At Month 3) ≥ 64 | 90 [84.51 to 93.74] | 81 [74.34 to 86.39] | 62 [52.35 to 70.39] | 6 [2.55 to 12.45] | 11 [6.11 to 17.67] | 84 [76.57 to 90.27]
  96217 Strain (At Month 3) ≥ 128 | 74 [67.28 to 80.32] | 63 [55.38 to 70.03] | 34 [25.76 to 43.38] | 4 [1.47 to 10.11] | 4 [1.28 to 8.88] | 60 [51.04 to 69.11]
  96217 Strain (At Month 7) ≥ LLQ (8.6) | 95 [91.01 to 97.76] | 91 [85.81 to 94.77] | 88 [80.22 to 92.83] | 97 [92.37 to 99.44] | 39 [30.56 to 48.08] | 99 [95.48 to 99.98]
  96217 Strain (At Month 7) ≥ 5 | 96 [92.40 to 98.47] | 93 [87.83 to 96.05] | 91 [84.19 to 95.33] | 97 [92.37 to 99.44] | 44 [35.00 to 52.79] | 99 [95.48 to 99.98]
  96217 Strain (At Month 7) ≥ 8 | 95 [91.01 to 97.76] | 91 [85.81 to 94.77] | 88 [80.22 to 92.83] | 97 [92.37 to 99.44] | 40 [31.30 to 48.87] | 99 [95.48 to 99.98]
  96217 Strain (At Month 7) ≥ 16 | 93 [88.34 to 96.23] | 85 [79.33 to 90.23] | 76 [67.17 to 83.18] | 96 [91.11 to 99.02] | 30 [22.65 to 39.22] | 99 [95.48 to 99.98]
  96217 Strain (At Month 7) ≥ 32 | 75 [67.85 to 80.80] | 65 [57.68 to 72.14] | 57 [47.31 to 65.68] | 96 [89.89 to 98.53] | 18 [11.74 to 25.73] | 98 [94.16 to 99.80]
  96217 Strain (At Month 7) ≥ 64 | 43 [35.79 to 50.46] | 34 [26.81 to 41.16] | 32 [23.48 to 40.78] | 87 [78.87 to 92.31] | 7 [3.27 to 12.93] | 98 [92.93 to 99.49]
  96217 Strain (At Month 7) ≥ 128 | 11 [7.13 to 16.74] | 7 [3.53 to 11.48] | 12 [6.53 to 18.80] | 73 [64.02 to 81.14] | 2 [0.49 to 6.70] | 85 [77.51 to 90.94]
  96217 Strain (At Month 13) ≥ LLQ (8.6) | 87 [81.41 to 91.55] | 83 [76.20 to 87.85] | 81 [72.64 to 87.44] | 90 [83.11 to 94.99] | 98 [93.30 to 99.51] | 93 [87.39 to 97.10]
  96217 Strain (At Month 13) ≥ 5 | 90 [85.14 to 94.16] | 85 [78.70 to 89.76] | 83 [75.44 to 89.51] | 92 [85.29 to 96.26] | 98 [94.47 to 99.81] | 93 [87.39 to 97.10]
  96217 Strain (At Month 13) ≥ 8 | 88 [82.03 to 92.00] | 83 [76.82 to 88.33] | 81 [72.64 to 87.44] | 90 [83.11 to 94.99] | 98 [94.47 to 99.81] | 93 [87.39 to 97.10]
  96217 Strain (At Month 13) ≥ 16 | 76 [69.00 to 81.77] | 69 [61.75 to 75.80] | 66 [56.62 to 74.24] | 79 [70.80 to 86.51] | 98 [93.30 to 99.51] | 88 [80.38 to 92.89]
  96217 Strain (At Month 13) ≥ 32 | 52 [44.72 to 59.51] | 40 [32.64 to 47.48] | 41 [31.95 to 50.18] | 57 [47.45 to 66.45] | 96 [91.12 to 98.72] | 64 [55.25 to 72.95]
  96217 Strain (At Month 13) ≥ 64 | 23 [17.26 to 29.85] | 13 [8.37 to 18.76] | 23 [15.38 to 31.02] | 30 [22.02 to 39.76] | 85 [77.79 to 90.82] | 36 [27.81 to 45.60]
  96217 Strain (At Month 13) ≥ 128 | 4 [1.87 to 8.30] | 3 [0.92 to 6.43] | 8 [3.49 to 13.76] | 13 [7.69 to 21.13] | 73 [64.08 to 80.16] | 12 [7.11 to 19.62]

14. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥LLQ, ≥5, ≥8, ≥16, ≥32, ≥64, ≥128 Against A Human Serogroup for All Schedules.
Description: The kinetic of immune response (at Months 0, 2, 3, 7 and 13) following different vaccination schedules as measured by the percentages of subjects with hSBA titers ≥LLQ, ≥5, ≥8, ≥16, ≥32, ≥64, ≥128 against A human serogroup was assessed.
Time Frame: At Month 0, Month 2, Month 3, Month 7 and Month 13.
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB_0_2 Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group | ABCWY_0_2_6 Group
Number analyzed (Participants) | 172 | 178 | 107 | 105 | 120 | 127
Percentages of subjects
  A human Serogroup (At Month 0) ≥ LLQ (22.7) | 6 [2.82 to 10.43] | 3 [1.25 to 7.19] | 5 [1.53 to 10.57] | 2 [0.23 to 6.71] | 3 [0.52 to 7.13] | 1 [0.02 to 4.31]
  A human Serogroup (At Month 0) ≥ 5 | 10 [6.32 to 16.03] | 6 [3.12 to 10.79] | 10 [5.24 to 17.65] | 4 [1.05 to 9.47] | 8 [3.49 to 13.76] | 3 [0.86 to 7.87]
  A human Serogroup (At Month 0) ≥ 8 | 10 [5.86 to 15.35] | 6 [2.73 to 10.09] | 10 [5.24 to 17.65] | 3 [0.59 to 8.12] | 5 [1.86 to 10.57] | 2 [0.49 to 6.75]
  A human Serogroup (At Month 0) ≥ 16 | 7 [3.66 to 11.87] | 4 [1.96 to 8.66] | 7 [3.28 to 14.20] | 2 [0.23 to 6.71] | 4 [1.37 to 9.46] | 2 [0.19 to 5.57]
  A human Serogroup (At Month 0) ≥ 32 | 4 [1.65 to 8.21] | 2 [0.62 to 5.65] | 3 [0.58 to 7.98] | 1 [0.02 to 5.19] | 2 [0.20 to 5.89] | 1 [0.02 to 4.31]
  A human Serogroup (At Month 0) ≥ 64 | 1 [0.14 to 4.14] | 1 [0.14 to 4.00] | 2 [0.23 to 6.59] | 1 [0.02 to 5.19] | 0 [0 to 3.03] | 1 [0.02 to 4.31]
  A human Serogroup (At Month 0) ≥ 128 | 1 [0.01 to 3.20] | 1 [0.01 to 3.09] | 1 [0.02 to 5.10] | 0 [0 to 3.45] | 0 [0 to 3.03] | 1 [0.02 to 4.31]
  A human Serogroup (At Month 2) ≥ LLQ (22.7) | 22 [16.13 to 29.04] | 35 [27.86 to 42.32] | 93 [85.80 to 96.72] | 33 [24.43 to 43.20] | 54 [44.83 to 63.29] | 28 [20.01 to 36.19]
  A human Serogroup (At Month 2) ≥ 5 | 37 [29.97 to 44.89] | 53 [45.76 to 60.87] | 95 [89.43 to 98.47] | 48 [37.78 to 57.59] | 75 [66.27 to 82.45] | 39 [30.08 to 47.63]
  A human Serogroup (At Month 2) ≥ 8 | 37 [29.43 to 44.30] | 51 [42.98 to 58.12] | 94 [88.19 to 97.91] | 46 [35.96 to 55.72] | 74 [65.38 to 81.72] | 38 [29.35 to 46.83]
  A human Serogroup (At Month 2) ≥ 16 | 28 [21.35 to 35.24] | 44 [36.41 to 51.44] | 93 [86.98 to 97.33] | 41 [31.45 to 50.98] | 67 [57.48 to 75.01] | 31 [22.83 to 39.51]
  A human Serogroup (At Month 2) ≥ 32 | 19 [13.09 to 25.24] | 33 [26.28 to 40.58] | 88 [80.12 to 93.37] | 30 [21.02 to 39.22] | 42 [32.74 to 51.02] | 22 [15.18 to 30.26]
  A human Serogroup (At Month 2) ≥ 64 | 12 [7.72 to 18.06] | 19 [13.12 to 25.04] | 69 [59.50 to 77.73] | 18 [11.26 to 26.81] | 33 [24.23 to 41.65] | 14 [8.62 to 21.47]
  A human Serogroup (At Month 2) ≥ 128 | 4 [1.65 to 8.21] | 10 [5.66 to 14.85] | 34 [24.80 to 43.42] | 9 [3.99 to 15.65] | 14 [8.47 to 21.71] | 6 [2.76 to 12.03]
  A human Serogroup (At Month 3) ≥ LLQ (22.7) | 94 [89.57 to 97.18] | 87 [80.61 to 91.17] | 80 [71.58 to 87.42] | 30 [21.02 to 39.22] | 38 [28.83 to 46.80] | 92 [86.00 to 96.16]
  A human Serogroup (At Month 3) ≥ 5 | 97 [93.35 to 99.05] | 94 [89.21 to 96.88] | 92 [84.63 to 96.08] | 40 [30.56 to 50.02] | 55 [45.65 to 64.09] | 94 [88.97 to 97.76]
  A human Serogroup (At Month 3) ≥ 8 | 97 [93.35 to 99.05] | 93 [87.83 to 96.05] | 91 [83.48 to 95.43] | 39 [29.67 to 49.06] | 53 [43.18 to 61.69] | 94 [87.97 to 97.24]
  A human Serogroup (At Month 3) ≥ 16 | 95 [90.30 to 97.58] | 91 [85.81 to 94.77] | 86 [77.93 to 91.94] | 33 [24.43 to 43.20] | 42 [32.74 to 51.02] | 92 [86.00 to 96.16]
  A human Serogroup (At Month 3) ≥ 32 | 91 [85.33 to 94.59] | 83 [76.20 to 87.85] | 74 [64.45 to 81.85] | 27 [18.51 to 36.19] | 31 [22.73 to 39.91] | 90 [83.13 to 94.44]
  A human Serogroup (At Month 3) ≥ 64 | 71 [63.53 to 77.59] | 57 [49.69 to 64.67] | 46 [36.12 to 55.70] | 12 [6.76 to 20.24] | 19 [12.56 to 27.36] | 61 [51.57 to 69.18]
  A human Serogroup (At Month 3) ≥ 128 | 45 [37.76 to 53.10] | 30 [23.17 to 37.07] | 21 [14.14 to 30.49] | 6 [2.13 to 12.02] | 10 [5.27 to 16.82] | 29 [21.41 to 37.85]
  A human Serogroup (At Month 7) ≥ LLQ (22.7) | 53 [45.74 to 61.12] | 46 [38.04 to 53.12] | 41 [31.70 to 51.05] | 95 [89.24 to 98.44] | 21 [13.96 to 29.20] | 94 [87.97 to 97.24]
  A human Serogroup (At Month 7) ≥ 5 | 70 [62.31 to 76.53] | 62 [54.80 to 69.50] | 60 [49.89 to 69.18] | 97 [91.88 to 99.41] | 29 [21.23 to 38.16] | 98 [93.25 to 99.51]
  A human Serogroup (At Month 7) ≥ 8 | 68 [60.50 to 74.92] | 58 [50.82 to 65.75] | 58 [48.01 to 67.42] | 97 [91.88 to 99.41] | 28 [19.75 to 36.40] | 98 [93.25 to 99.51]
  A human Serogroup (At Month 7) ≥ 16 | 61 [53.33 to 68.38] | 51 [43.53 to 58.67] | 49 [38.82 to 58.46] | 97 [91.88 to 99.41] | 22 [14.67 to 30.11] | 97 [92.13 to 99.14]
  A human Serogroup (At Month 7) ≥ 32 | 42 [34.95 to 50.20] | 37 [29.44 to 44.05] | 35 [25.65 to 44.39] | 91 [84.35 to 96.01] | 14 [8.47 to 21.71] | 93 [86.97 to 96.71]
  A human Serogroup (At Month 7) ≥ 64 | 19 [13.59 to 25.88] | 19 [13.61 to 25.66] | 18 [11.04 to 26.33] | 76 [66.89 to 83.96] | 7 [2.92 to 12.71] | 80 [72.33 to 86.84]
  A human Serogroup (At Month 7) ≥ 128 | 5 [2.42 to 9.70] | 6 [2.73 to 10.09] | 10 [5.24 to 17.65] | 63 [52.88 to 72.09] | 3 [0.52 to 7.13] | 54 [44.48 to 62.44]
  A human Serogroup (At Month 13) ≥ LLQ (22.7) | 33 [26.16 to 40.71] | 26 [20.09 to 33.52] | 34 [24.80 to 43.42] | 51 [41.47 to 61.30] | 93 [87.29 to 97.08] | 54 [45.26 to 63.19]
  A human Serogroup (At Month 13) ≥ 5 | 51 [42.87 to 58.28] | 42 [34.25 to 49.18] | 48 [37.92 to 57.54] | 68 [57.79 to 76.43] | 98 [92.87 to 99.48] | 65 [55.59 to 72.85]
  A human Serogroup (At Month 13) ≥ 8 | 48 [40.59 to 55.99] | 39 [31.57 to 46.34] | 47 [37.02 to 56.62] | 66 [55.81 to 74.70] | 98 [92.87 to 99.48] | 64 [54.78 to 72.12]
  A human Serogroup (At Month 13) ≥ 16 | 38 [30.52 to 45.49] | 30 [23.68 to 37.66] | 41 [31.70 to 51.05] | 59 [49.02 to 68.55] | 95 [89.43 to 98.14] | 60 [50.78 to 68.44]
  A human Serogroup (At Month 13) ≥ 32 | 24 [17.68 to 30.92] | 20 [14.09 to 26.27] | 27 [18.96 to 36.55] | 44 [34.14 to 53.83] | 88 [81.20 to 93.47] | 41 [32.30 to 50.02]
  A human Serogroup (At Month 13) ≥ 64 | 13 [8.67 to 19.39] | 8 [4.79 to 13.52] | 13 [7.34 to 20.98] | 27 [18.51 to 36.19] | 81 [72.64 to 87.44] | 16 [9.89 to 23.27]
  A human Serogroup (At Month 13) ≥ 128 | 4 [1.65 to 8.21] | 2 [0.35 to 4.85] | 6 [2.09 to 11.81] | 8 [3.35 to 14.46] | 61 [51.50 to 69.61] | 6 [2.24 to 11.03]

15. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥LLQ, ≥5, ≥8, ≥16, ≥32, ≥64, ≥128 Against C Human Serogroup for All Schedules.
Description: The kinetic of immune response (at Months 0, 2, 3, 7 and 13) following different vaccination schedules as measured by the percentages of subjects with hSBA titers ≥LLQ, ≥5, ≥8, ≥16, ≥32, ≥64, ≥128 against C human serogroup was assessed.
Time Frame: At Month 0, Month 2, Month 3, Month 7 and Month 13.
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB_0_2 Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group | ABCWY_0_2_6 Group
Number analyzed (Participants) | 186 | 185 | 122 | 114 | 123 | 130
Percentages of subjects
  C human Serogroup (At Month 0) ≥ LLQ (5.2) | 43 [35.79 to 50.46] | 45 [38.09 to 52.87] | 48 [38.43 to 56.78] | 41 [32.09 to 50.83] | 48 [38.88 to 57.16] | 41 [32.24 to 49.73]
  C human Serogroup (At Month 0) ≥ 5 | 46 [38.91 to 53.68] | 45 [38.09 to 52.87] | 49 [40.02 to 58.38] | 43 [33.75 to 52.59] | 49 [39.67 to 57.95] | 42 [32.97 to 50.51]
  C human Serogroup (At Month 0) ≥ 8 | 34 [27.61 to 41.71] | 30 [23.75 to 37.44] | 36 [27.57 to 45.25] | 30 [21.62 to 39.11] | 36 [27.33 to 44.91] | 30 [22.28 to 38.66]
  C human Serogroup (At Month 0) ≥ 16 | 19 [13.47 to 25.19] | 14 [8.94 to 19.30] | 20 [13.03 to 27.84] | 14 [8.24 to 21.79] | 24 [17.10 to 32.95] | 8 [3.75 to 13.69]
  C human Serogroup (At Month 0) ≥ 32 | 5 [2.61 to 9.66] | 6 [3.40 to 11.06] | 9 [4.59 to 15.56] | 4 [0.96 to 8.74] | 7 [3.40 to 13.44] | 3 [0.84 to 7.69]
  C human Serogroup (At Month 0) ≥ 64 | 2 [0.59 to 5.41] | 2 [0.34 to 4.67] | 2 [0.20 to 5.80] | 3 [0.55 to 7.50] | 3 [0.89 to 8.12] | 1 [0.02 to 4.21]
  C human Serogroup (At Month 0) ≥ 128 | 1 [0.01 to 2.96] | 2 [0.34 to 4.67] | 0 [0 to 2.98] | 1 [0.02 to 4.79] | 1 [0.02 to 4.45] | 0 [0 to 2.80]
  C human Serogroup (At Month 2) ≥ LLQ (5.2) | 61 [53.89 to 68.33] | 84 [78.27 to 89.24] | 100 [97.02 to 100] | 84 [76.20 to 90.37] | 89 [82.60 to 94.25] | 88 [80.78 to 92.80]
  C human Serogroup (At Month 2) ≥ 5 | 62 [54.98 to 69.35] | 84 [78.27 to 89.24] | 100 [97.02 to 100] | 84 [76.20 to 90.37] | 89 [82.60 to 94.25] | 88 [80.78 to 92.80]
  C human Serogroup (At Month 2) ≥ 8 | 53 [45.25 to 60.04] | 78 [71.16 to 83.60] | 98 [94.20 to 99.80] | 80 [71.28 to 86.76] | 86 [78.80 to 91.74] | 78 [69.56 to 84.52]
  C human Serogroup (At Month 2) ≥ 16 | 35 [28.62 to 42.82] | 65 [57.52 to 71.73] | 95 [89.60 to 98.17] | 64 [54.51 to 72.81] | 72 [62.71 to 79.31] | 61 [51.82 to 69.21]
  C human Serogroup (At Month 2) ≥ 32 | 18 [13.00 to 24.60] | 40 [32.88 to 47.44] | 89 [81.50 to 93.58] | 44 [34.58 to 53.46] | 55 [46.06 to 64.25] | 44 [35.16 to 52.82]
  C human Serogroup (At Month 2) ≥ 64 | 8 [4.58 to 12.95] | 23 [17.36 to 30.00] | 79 [70.35 to 85.58] | 29 [20.84 to 38.19] | 39 [30.36 to 48.23] | 25 [17.49 to 32.94]
  C human Serogroup (At Month 2) ≥ 128 | 3 [0.88 to 6.16] | 16 [10.76 to 21.73] | 53 [44.03 to 62.36] | 17 [10.34 to 24.80] | 26 [18.52 to 34.70] | 19 [12.85 to 27.07]
  C human Serogroup (At Month 3) ≥ LLQ (5.2) | 97 [93.84 to 99.12] | 99 [96.15 to 99.87] | 98 [94.20 to 99.80] | 81 [72.25 to 87.49] | 88 [80.68 to 93.01] | 99 [95.79 to 99.98]
  C human Serogroup (At Month 3) ≥ 5 | 97 [93.84 to 99.12] | 99 [96.15 to 99.87] | 98 [94.20 to 99.80] | 81 [72.25 to 87.49] | 88 [80.68 to 93.01] | 100 [97.20 to 100]
  C human Serogroup (At Month 3) ≥ 8 | 94 [89.00 to 96.62] | 98 [94.56 to 99.41] | 98 [92.98 to 99.49] | 77 [68.40 to 84.53] | 84 [76.01 to 89.78] | 99 [95.79 to 99.98]
  C human Serogroup (At Month 3) ≥ 16 | 78 [71.89 to 84.17] | 96 [92.36 to 98.47] | 95 [89.60 to 98.17] | 62 [52.72 to 71.19] | 63 [54.25 to 71.91] | 98 [93.40 to 99.52]
  C human Serogroup (At Month 3) ≥ 32 | 56 [48.46 to 63.17] | 90 [84.43 to 93.70] | 86 [78.63 to 91.67] | 43 [33.75 to 52.59] | 46 [36.53 to 54.75] | 94 [88.23 to 97.31]
  C human Serogroup (At Month 3) ≥ 64 | 26 [19.68 to 32.72] | 78 [71.16 to 83.60] | 67 [58.13 to 75.44] | 25 [17.75 to 34.45] | 30 [22.14 to 39.00] | 85 [77.24 to 90.34]
  C human Serogroup (At Month 3) ≥ 128 | 11 [6.69 to 16.12] | 58 [50.92 to 65.57] | 40 [31.39 to 49.42] | 18 [11.06 to 25.79] | 21 [14.30 to 29.42] | 60 [51.05 to 68.49]
  C human Serogroup (At Month 7) ≥ LLQ (5.2) | 69 [61.63 to 75.39] | 96 [92.36 to 98.47] | 97 [91.82 to 99.10] | 99 [95.21 to 99.98] | 82 [74.18 to 88.44] | 100 [97.20 to 100]
  C human Serogroup (At Month 7) ≥ 5 | 69 [62.19 to 75.89] | 96 [92.36 to 98.47] | 97 [91.82 to 99.10] | 99 [95.21 to 99.98] | 82 [74.18 to 88.44] | 100 [97.20 to 100]
  C human Serogroup (At Month 7) ≥ 8 | 58 [50.62 to 65.24] | 96 [92.36 to 98.47] | 96 [90.69 to 98.66] | 99 [95.21 to 99.98] | 73 [64.43 to 80.76] | 99 [95.79 to 99.98]
  C human Serogroup (At Month 7) ≥ 16 | 38 [30.65 to 45.02] | 90 [85.06 to 94.13] | 91 [84.44 to 95.41] | 98 [93.81 to 99.79] | 55 [46.06 to 64.25] | 99 [95.79 to 99.98]
  C human Serogroup (At Month 7) ≥ 32 | 23 [16.79 to 29.27] | 74 [66.54 to 79.72] | 77 [68.57 to 84.18] | 95 [88.90 to 98.04] | 35 [26.58 to 44.08] | 98 [94.55 to 99.81]
  C human Serogroup (At Month 7) ≥ 64 | 9 [5.00 to 13.59] | 53 [45.51 to 60.34] | 53 [44.03 to 62.36] | 86 [78.21 to 91.76] | 26 [18.52 to 34.70] | 96 [91.25 to 98.74]
  C human Serogroup (At Month 7) ≥ 128 | 3 [0.88 to 6.16] | 30 [23.75 to 37.44] | 25 [17.96 to 34.09] | 74 [64.61 to 81.49] | 16 [10.22 to 23.99] | 85 [78.12 to 90.97]
  C human Serogroup (At Month 13) ≥ LLQ (5.2) | 60 [52.25 to 66.79] | 92 [87.63 to 95.80] | 94 [88.54 to 97.66] | 97 [92.50 to 99.45] | 100 [97.05 to 100] | 99 [95.79 to 99.98]
  C human Serogroup (At Month 13) ≥ 5 | 61 [53.34 to 67.82] | 92 [87.63 to 95.80] | 94 [88.54 to 97.66] | 98 [93.81 to 99.79] | 100 [97.05 to 100] | 99 [95.79 to 99.98]
  C human Serogroup (At Month 13) ≥ 8 | 48 [41.01 to 55.81] | 88 [82.55 to 92.40] | 89 [82.47 to 94.20] | 91 [84.46 to 95.71] | 98 [94.25 to 99.80] | 98 [93.40 to 99.52]
  C human Serogroup (At Month 13) ≥ 16 | 30 [23.61 to 37.25] | 78 [71.26 to 83.60] | 79 [70.35 to 85.58] | 83 [75.20 to 89.66] | 98 [93.04 to 99.49] | 94 [88.23 to 97.31]
  C human Serogroup (At Month 13) ≥ 32 | 15 [10.24 to 21.02] | 51 [43.37 to 58.22] | 57 [48.10 to 66.28] | 61 [51.83 to 70.37] | 97 [91.88 to 99.11] | 81 [72.93 to 87.15]
  C human Serogroup (At Month 13) ≥ 64 | 9 [5.00 to 13.59] | 28 [21.76 to 35.17] | 25 [17.25 to 33.21] | 38 [28.81 to 47.28] | 93 [87.59 to 97.15] | 58 [49.49 to 67.03]
  C human Serogroup (At Month 13) ≥ 128 | 2 [0.59 to 5.41] | 16 [10.76 to 21.73] | 16 [10.31 to 24.18] | 25 [16.98 to 33.51] | 85 [76.93 to 90.44] | 40 [31.51 to 48.95]

16. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥LLQ, ≥5, ≥8, ≥16, ≥32, ≥64, ≥128 Against W Human Serogroup for All Schedules.
Description: The kinetic of immune response (at Months 0, 2, 3, 7 and 13) following different vaccination schedules as measured by the percentages of subjects with hSBA titers ≥LLQ, ≥5, ≥8, ≥16, ≥32, ≥64, ≥128 against W human serogroup was assessed.
Time Frame: At Month 0, Month 2, Month 3, Month 7 and Month 13.
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB_0_2 Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group | ABCWY_0_2_6 Group
Number analyzed (Participants) | 162 | 180 | 119 | 108 | 123 | 123
Percentages of subjects
  W human Serogroup (At Month 0) ≥ LLQ (39.6) | 30 [23.29 to 37.95] | 26 [19.86 to 33.17] | 29 [21.42 to 38.46] | 20 [13.23 to 29.20] | 29 [21.41 to 38.15] | 22 [14.99 to 30.31]
  W human Serogroup (At Month 0) ≥ 5 | 51 [43.27 to 59.15] | 43 [35.98 to 50.91] | 41 [32.24 to 50.57] | 42 [32.25 to 51.55] | 45 [35.75 to 53.94] | 45 [35.75 to 53.94]
  W human Serogroup (At Month 0) ≥ 8 | 49 [41.45 to 57.34] | 41 [33.85 to 48.67] | 40 [31.45 to 49.72] | 41 [31.38 to 50.62] | 45 [35.75 to 53.94] | 43 [34.20 to 52.32]
  W human Serogroup (At Month 0) ≥ 16 | 44 [36.05 to 51.83] | 39 [31.73 to 46.42] | 39 [30.66 to 48.87] | 34 [25.40 to 44.01] | 41 [31.89 to 49.88] | 38 [29.60 to 47.41]
  W human Serogroup (At Month 0) ≥ 32 | 35 [27.86 to 43.07] | 31 [24.43 to 38.42] | 31 [22.93 to 40.23] | 24 [16.37 to 33.25] | 33 [25.09 to 42.40] | 26 [18.52 to 34.70]
  W human Serogroup (At Month 0) ≥ 64 | 21 [14.99 to 28.07] | 19 [13.45 to 25.38] | 20 [13.37 to 28.51] | 13 [7.27 to 20.79] | 21 [14.30 to 29.42] | 12 [6.99 to 19.32]
  W human Serogroup (At Month 0) ≥ 128 | 8 [4.34 to 13.33] | 9 [5.17 to 14.03] | 10 [5.32 to 16.95] | 10 [5.20 to 17.49] | 7 [2.85 to 12.41] | 4 [1.33 to 9.23]
  W human Serogroup (At Month 2) ≥ LLQ (39.6) | 48 [40.24 to 56.12] | 65 [57.55 to 71.95] | 96 [90.47 to 98.62] | 67 [56.95 to 75.45] | 77 [68.81 to 84.31] | 60 [50.95 to 68.88]
  W human Serogroup (At Month 2) ≥ 5 | 66 [58.21 to 73.29] | 90 [84.66 to 93.96] | 99 [95.41 to 99.98] | 92 [84.77 to 96.12] | 93 [86.56 to 96.60] | 93 [86.56 to 96.60]
  W human Serogroup (At Month 2) ≥ 8 | 64 [56.30 to 71.57] | 86 [80.18 to 90.81] | 99 [95.41 to 99.98] | 92 [84.77 to 96.12] | 93 [86.56 to 96.60] | 89 [81.64 to 93.64]
  W human Serogroup (At Month 2) ≥ 16 | 60 [52.52 to 68.07] | 82 [75.84 to 87.51] | 99 [95.41 to 99.98] | 81 [72.86 to 88.31] | 89 [82.60 to 94.25] | 80 [72.37 to 87.08]
  W human Serogroup (At Month 2) ≥ 32 | 52 [44.49 to 60.36] | 69 [62.16 to 76.08] | 98 [94.06 to 99.80] | 72 [62.78 to 80.41] | 78 [69.69 to 85.01] | 65 [55.92 to 73.42]
  W human Serogroup (At Month 2) ≥ 64 | 44 [36.05 to 51.83] | 50 [42.47 to 57.53] | 84 [76.19 to 90.10] | 52 [42.03 to 61.57] | 67 [58.45 to 75.65] | 44 [34.97 to 53.13]
  W human Serogroup (At Month 2) ≥ 128 | 29 [22.16 to 36.65] | 31 [23.92 to 37.84] | 62 [52.84 to 70.91] | 33 [24.55 to 43.05] | 49 [39.67 to 57.95] | 27 [19.24 to 35.57]
  W human Serogroup (At Month 3) ≥ LLQ (39.6) | 89 [83.01 to 93.28] | 97 [92.89 to 98.77] | 85 [77.15 to 90.78] | 68 [57.91 to 76.28] | 77 [68.81 to 84.31] | 97 [91.88 to 99.11]
  W human Serogroup (At Month 3) ≥ 5 | 96 [92.11 to 98.63] | 99 [96.04 to 99.87] | 98 [94.06 to 99.80] | 94 [87.10 to 97.35] | 92 [85.56 to 96.03] | 100 [97.05 to 100]
  W human Serogroup (At Month 3) ≥ 8 | 96 [92.11 to 98.63] | 99 [96.04 to 99.87] | 97 [92.81 to 99.48] | 90 [82.51 to 94.80] | 90 [83.58 to 94.86] | 100 [97.05 to 100]
  W human Serogroup (At Month 3) ≥ 16 | 96 [91.30 to 98.25] | 99 [96.04 to 99.87] | 96 [90.47 to 98.62] | 81 [71.83 to 87.54] | 86 [78.80 to 91.74] | 99 [95.55 to 99.98]
  W human Serogroup (At Month 3) ≥ 32 | 91 [85.19 to 94.72] | 98 [94.41 to 99.39] | 91 [84.06 to 95.29] | 73 [63.76 to 81.22] | 78 [69.69 to 85.01] | 98 [93.04 to 99.49]
  W human Serogroup (At Month 3) ≥ 64 | 80 [73.27 to 86.08] | 93 [88.64 to 96.51] | 77 [68.73 to 84.48] | 50 [40.22 to 59.78] | 64 [55.09 to 72.67] | 91 [84.56 to 95.45]
  W human Serogroup (At Month 3) ≥ 128 | 61 [53.15 to 68.66] | 74 [66.83 to 80.14] | 50 [41.11 to 59.71] | 33 [24.55 to 43.05] | 44 [34.97 to 53.13] | 70 [61.00 to 77.86]
  W human Serogroup (At Month 7) ≥ LLQ (39.6) | 60 [51.90 to 67.49] | 82 [75.23 to 87.03] | 79 [70.57 to 85.92] | 99 [94.95 to 99.98] | 74 [65.30 to 81.48] | 99 [95.55 to 99.98]
  W human Serogroup (At Month 7) ≥ 5 | 71 [63.35 to 77.84] | 97 [92.89 to 98.77] | 96 [90.47 to 98.62] | 100 [96.64 to 100] | 93 [86.56 to 96.60] | 100 [97.05 to 100]
  W human Serogroup (At Month 7) ≥ 8 | 70 [62.70 to 77.28] | 95 [90.72 to 97.69] | 95 [89.35 to 98.13] | 100 [96.64 to 100] | 91 [84.56 to 95.45] | 100 [97.05 to 100]
  W human Serogroup (At Month 7) ≥ 16 | 69 [61.41 to 76.15] | 92 [87.29 to 95.68] | 91 [84.06 to 95.29] | 100 [96.64 to 100] | 87 [79.74 to 92.38] | 100 [97.05 to 100]
  W human Serogroup (At Month 7) ≥ 32 | 63 [55.03 to 70.41] | 84 [78.31 to 89.41] | 84 [76.19 to 90.10] | 100 [96.64 to 100] | 76 [67.93 to 83.61] | 99 [95.55 to 99.98]
  W human Serogroup (At Month 7) ≥ 64 | 49 [40.85 to 56.73] | 68 [60.42 to 74.54] | 67 [58.02 to 75.55] | 97 [92.10 to 99.42] | 59 [49.31 to 67.35] | 98 [93.04 to 99.49]
  W human Serogroup (At Month 7) ≥ 128 | 31 [23.85 to 38.59] | 41 [33.31 to 48.11] | 34 [25.98 to 43.72] | 87 [79.21 to 92.73] | 34 [25.84 to 43.24] | 82 [74.18 to 88.44]
  W human Serogroup (At Month 13) ≥ LLQ (39.6) | 47 [39.04 to 54.90] | 64 [56.41 to 70.90] | 66 [56.28 to 74.02] | 82 [73.90 to 89.06] | 98 [93.04 to 99.49] | 84 [76.01 to 89.78]
  W human Serogroup (At Month 13) ≥ 5 | 62 [54.40 to 69.83] | 93 [87.97 to 96.10] | 90 [83.05 to 94.68] | 99 [94.95 to 99.98] | 99 [95.55 to 99.98] | 98 [94.25 to 99.80]
  W human Serogroup (At Month 13) ≥ 8 | 60 [52.52 to 68.07] | 90 [84.66 to 93.96] | 90 [83.05 to 94.68] | 98 [93.47 to 99.77] | 99 [95.55 to 99.98] | 98 [94.25 to 99.80]
  W human Serogroup (At Month 13) ≥ 16 | 57 [48.79 to 64.54] | 84 [77.69 to 88.94] | 81 [72.42 to 87.34] | 94 [87.10 to 97.35] | 99 [95.55 to 99.98] | 96 [90.77 to 98.67]
  W human Serogroup (At Month 13) ≥ 32 | 50 [42.05 to 57.95] | 71 [63.90 to 77.61] | 72 [63.32 to 80.08] | 85 [77.06 to 91.29] | 98 [94.25 to 99.80] | 89 [82.60 to 94.25]
  W human Serogroup (At Month 13) ≥ 64 | 35 [27.28 to 42.43] | 44 [36.52 to 51.47] | 48 [38.66 to 57.25] | 73 [63.76 to 81.22] | 98 [93.04 to 99.49] | 68 [59.29 to 76.39]
  W human Serogroup (At Month 13) ≥ 128 | 21 [14.99 to 28.07] | 22 [16.38 to 29.01] | 28 [19.92 to 36.68] | 43 [33.13 to 52.47] | 94 [88.63 to 97.68] | 45 [35.75 to 53.94]

17. Secondary Outcome: Percentages of Subjects With hSBA Titers ≥LLQ, ≥5, ≥8, ≥16, ≥32, ≥64, ≥128 Against Y Human Serogroup for All Schedules.
Description: The kinetic of immune response (at Months 0, 2, 3, 7 and 13) following different vaccination schedules as measured by the percentages of subjects with hSBA titers ≥LLQ, ≥5, ≥8, ≥16, ≥32, ≥64, ≥128 against Y human serogroup was assessed.
Time Frame: At Month 0, Month 2, Month 3, Month 7 and Month 13.
Population: Analysis was done on the FAS Month 13 which included all screened subjects who received a study vaccination & provided evaluable serum samples at month 0 and atleast from month 2 to 13 and provided results for at least one serogroup or serogroup B test strain.
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB_0_2 Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group | ABCWY_0_2_6 Group
Number analyzed (Participants) | 188 | 180 | 120 | 110 | 127 | 137
Percentages of subjects
  Y human Serogroup (At Month 0) ≥ LLQ (14.7) | 15 [10.13 to 20.80] | 10 [6.04 to 15.34] | 13 [7.82 to 20.75] | 6 [2.60 to 12.67] | 13 [7.38 to 19.65] | 7 [3.05 to 12.10]
  Y human Serogroup (At Month 0) ≥ 5 | 16 [11.03 to 21.99] | 11 [6.92 to 16.64] | 15 [9.14 to 22.67] | 7 [3.19 to 13.83] | 17 [10.54 to 24.16] | 9 [4.61 to 14.80]
  Y human Serogroup (At Month 0) ≥ 8 | 16 [11.03 to 21.99] | 11 [6.92 to 16.64] | 14 [8.47 to 21.71] | 7 [3.19 to 13.83] | 16 [9.89 to 23.27] | 9 [4.61 to 14.80]
  Y human Serogroup (At Month 0) ≥ 16 | 15 [10.13 to 20.80] | 10 [6.04 to 15.34] | 13 [7.17 to 19.78] | 6 [2.60 to 12.67] | 12 [6.76 to 18.73] | 6 [2.55 to 11.18]
  Y human Serogroup (At Month 0) ≥ 32 | 9 [5.36 to 14.08] | 3 [0.91 to 6.36] | 8 [4.07 to 14.79] | 3 [0.57 to 7.76] | 8 [3.84 to 14.00] | 4 [1.62 to 9.29]
  Y human Serogroup (At Month 0) ≥ 64 | 2 [0.58 to 5.36] | 2 [0.35 to 4.79] | 4 [1.37 to 9.46] | 0 [0 to 3.30] | 5 [1.75 to 10.00] | 3 [0.80 to 7.31]
  Y human Serogroup (At Month 0) ≥ 128 | 0 [0 to 1.94] | 1 [0.01 to 3.06] | 1 [0.02 to 4.56] | 0 [0 to 3.30] | 1 [0.02 to 4.31] | 1 [0.02 to 4.00]
  Y human Serogroup (At Month 2) ≥ LLQ (14.7) | 21 [15.19 to 27.25] | 66 [58.70 to 72.99] | 85 [77.33 to 90.86] | 60 [50.22 to 69.22] | 72 [62.98 to 79.29] | 61 [52.62 to 69.51]
  Y human Serogroup (At Month 2) ≥ 5 | 27 [20.91 to 34.08] | 72 [64.48 to 78.12] | 90 [83.18 to 94.73] | 65 [55.79 to 74.26] | 78 [69.74 to 84.82] | 65 [56.35 to 72.91]
  Y human Serogroup (At Month 2) ≥ 8 | 26 [19.95 to 32.95] | 70 [62.74 to 76.59] | 89 [82.19 to 94.10] | 62 [52.07 to 70.92] | 76 [68.03 to 83.46] | 64 [54.85 to 71.56]
  Y human Serogroup (At Month 2) ≥ 16 | 20 [14.72 to 26.67] | 64 [56.41 to 70.90] | 85 [77.33 to 90.86] | 58 [48.39 to 67.52] | 69 [60.49 to 77.17] | 60 [51.14 to 68.13]
  Y human Serogroup (At Month 2) ≥ 32 | 13 [8.35 to 18.40] | 47 [39.75 to 54.79] | 75 [66.27 to 82.45] | 47 [37.68 to 57.02] | 54 [44.48 to 62.44] | 50 [41.70 to 59.01]
  Y human Serogroup (At Month 2) ≥ 64 | 5 [2.21 to 8.89] | 31 [23.92 to 37.84] | 59 [49.82 to 68.05] | 30 [21.63 to 39.48] | 39 [30.08 to 47.63] | 39 [31.18 to 48.12]
  Y human Serogroup (At Month 2) ≥ 128 | 1 [0.13 to 3.79] | 14 [9.19 to 19.82] | 39 [30.39 to 48.50] | 12 [6.45 to 19.36] | 23 [15.86 to 31.12] | 23 [16.56 to 31.34]
  Y human Serogroup (At Month 3) ≥ LLQ (14.7) | 27 [20.43 to 33.52] | 92 [87.29 to 95.68] | 80 [71.72 to 86.75] | 58 [48.39 to 67.52] | 62 [53.17 to 70.65] | 90 [83.45 to 94.30]
  Y human Serogroup (At Month 3) ≥ 5 | 33 [26.31 to 40.19] | 94 [89.33 to 96.91] | 84 [76.38 to 90.19] | 65 [54.85 to 73.43] | 70 [61.32 to 77.88] | 93 [86.99 to 96.44]
  Y human Serogroup (At Month 3) ≥ 8 | 30 [23.84 to 37.43] | 93 [88.64 to 96.51] | 83 [75.44 to 89.51] | 60 [50.22 to 69.22] | 67 [58.03 to 75.02] | 93 [86.99 to 96.44]
  Y human Serogroup (At Month 3) ≥ 16 | 26 [19.95 to 32.95] | 92 [86.63 to 95.26] | 79 [70.80 to 86.04] | 57 [47.48 to 66.66] | 59 [49.98 to 67.70] | 90 [83.45 to 94.30]
  Y human Serogroup (At Month 3) ≥ 32 | 18 [12.86 to 24.34] | 84 [77.69 to 88.94] | 68 [58.35 to 75.77] | 44 [34.20 to 53.42] | 44 [35.30 to 53.17] | 83 [75.88 to 89.05]
  Y human Serogroup (At Month 3) ≥ 64 | 9 [4.94 to 13.45] | 68 [61.00 to 75.05] | 47 [37.51 to 55.99] | 24 [16.06 to 32.68] | 31 [23.55 to 40.33] | 65 [56.35 to 72.91]
  Y human Serogroup (At Month 3) ≥ 128 | 2 [0.58 to 5.36] | 39 [32.25 to 46.99] | 28 [19.75 to 36.40] | 16 [10.00 to 24.62] | 23 [15.86 to 31.12] | 47 [38.15 to 55.43]
  Y human Serogroup (At Month 7) ≥ LLQ (14.7) | 23 [17.07 to 29.55] | 78 [70.99 to 83.62] | 72 [62.72 to 79.51] | 95 [88.51 to 97.97] | 54 [44.48 to 62.44] | 97 [92.69 to 99.20]
  Y human Serogroup (At Month 7) ≥ 5 | 26 [19.95 to 32.95] | 86 [79.56 to 90.34] | 80 [71.72 to 86.75] | 95 [89.71 to 98.51] | 69 [59.67 to 76.45] | 99 [94.83 to 99.82]
  Y human Serogroup (At Month 7) ≥ 8 | 26 [19.46 to 32.39] | 84 [77.69 to 88.94] | 77 [68.07 to 83.90] | 95 [89.71 to 98.51] | 64 [54.78 to 72.12] | 98 [93.73 to 99.55]
  Y human Serogroup (At Month 7) ≥ 16 | 22 [16.13 to 28.40] | 74 [66.83 to 80.14] | 69 [60.09 to 77.27] | 94 [87.33 to 97.40] | 52 [42.93 to 60.91] | 97 [92.69 to 99.20]
  Y human Serogroup (At Month 7) ≥ 32 | 13 [8.35 to 18.40] | 63 [55.27 to 69.85] | 54 [44.83 to 63.29] | 87 [79.57 to 92.86] | 40 [31.56 to 49.22] | 91 [85.20 to 95.39]
  Y human Serogroup (At Month 7) ≥ 64 | 3 [0.87 to 6.10] | 37 [30.15 to 44.73] | 35 [26.52 to 44.24] | 79 [70.30 to 86.26] | 27 [19.31 to 35.35] | 75 [67.08 to 82.16]
  Y human Serogroup (At Month 7) ≥ 128 | 1 [0.01 to 2.93] | 14 [9.66 to 20.44] | 22 [14.67 to 30.11] | 57 [47.48 to 66.66] | 13 [8.00 to 20.56] | 57 [48.20 to 65.36]
  Y human Serogroup (At Month 13) ≥ LLQ (14.7) | 19 [13.32 to 24.93] | 64 [56.41 to 70.90] | 58 [48.15 to 66.47] | 78 [69.30 to 85.49] | 97 [92.13 to 99.14] | 82 [75.06 to 88.44]
  Y human Serogroup (At Month 13) ≥ 5 | 25 [18.98 to 31.82] | 76 [68.61 to 81.64] | 73 [64.49 to 80.99] | 91 [83.92 to 95.55] | 97 [92.13 to 99.14] | 91 [85.20 to 95.39]
  Y human Serogroup (At Month 13) ≥ 8 | 24 [18.03 to 30.69] | 71 [63.90 to 77.61] | 63 [54.05 to 71.94] | 84 [75.38 to 90.00] | 97 [92.13 to 99.14] | 87 [80.03 to 92.02]
  Y human Serogroup (At Month 13) ≥ 16 | 18 [12.40 to 23.76] | 61 [53.58 to 68.27] | 55 [45.65 to 64.09] | 76 [67.32 to 83.94] | 97 [92.13 to 99.14] | 81 [73.44 to 87.21]
  Y human Serogroup (At Month 13) ≥ 32 | 10 [5.77 to 14.71] | 43 [35.45 to 50.35] | 40 [31.17 to 49.34] | 60 [50.22 to 69.22] | 93 [86.97 to 96.71] | 69 [60.13 to 76.27]
  Y human Serogroup (At Month 13) ≥ 64 | 3 [1.18 to 6.82] | 21 [15.39 to 27.81] | 23 [15.38 to 31.02] | 41 [31.63 to 50.69] | 92 [86.00 to 96.16] | 46 [37.44 to 54.70]
  Y human Serogroup (At Month 13) ≥ 128 | 1 [0.13 to 3.79] | 9 [5.17 to 14.03] | 11 [5.90 to 17.81] | 21 [13.74 to 29.70] | 73 [64.65 to 80.69] | 28 [21.09 to 36.80]

18. Secondary Outcome: Percentages of Subjects With Two-, Three- and Four-fold Titer Rise Against Serogroups A, C, W and Y and Serogroup B Test Strains for All Schedules.
Description: The kinetic of immune response (at Months 2, 3, 7 and 13) following different vaccination schedules as measured by the percentages of subjects with two-, three- and four-fold titer rise against serogroups A, C, W and Y and serogroup B test strains was assessed. The two/three/four fold titer rise is defined as: a) for subjects with prevaccination hSBA titers ≤ LLQ, a postvaccination hSBA ≥ 2/3/4 LLQ; b) for subjects with a prevaccination hSBA titers ≥ LLQ, an increase of at least 2/3/4 times of the prevaccination hSBA titer.
Time Frame: At Month 2, Month 3, Month 7 and Month 13
Population: as for outcome 9
Measure: Number (95% Confidence Interval); unit: Percentages of subjects
Arm/Group | rMenB_0_2 Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group | ABCWY_0_2_6 Group
Number analyzed (Participants) | 188 | 185 | 122 | 114 | 128 | 137
Percentages of subjects
  NZ98/254 Strain ≥ 2-fold (At Month 2) | 18 [12.86 to 24.34] | 13 [8.49 to 18.69] | 28 [19.75 to 36.40] | 9 [4.36 to 15.81] | 21 [14.62 to 29.62] | 12 [6.98 to 18.67]
  NZ98/254 Strain ≥ 3-fold (At Month 2) | 14 [9.24 to 19.60] | 9 [5.44 to 14.30] | 19 [12.56 to 27.36] | 9 [4.36 to 15.81] | 17 [11.28 to 25.23] | 7 [3.64 to 13.30]
  NZ98/254 Strain ≥ 4-fold (At Month 2) | 11 [7.05 to 16.57] | 8 [4.61 to 13.02] | 17 [10.49 to 24.56] | 7 [3.13 to 13.59] | 17 [10.62 to 24.34] | 7 [3.12 to 12.37]
  NZ98/254 Strain ≥ 2-fold (At Month 3) | 73 [66.48 to 79.57] | 42 [34.43 to 49.08] | 18 [11.17 to 25.50] | 9 [4.36 to 15.81] | 13 [8.06 to 20.72] | 43 [34.76 to 52.11]
  NZ98/254 Strain ≥ 3-fold (At Month 3) | 61 [53.81 to 68.18] | 32 [25.25 to 39.13] | 13 [7.17 to 19.78] | 5 [1.99 to 11.30] | 10 [5.61 to 17.00] | 28 [20.91 to 36.79]
  NZ98/254 Strain ≥ 4-fold (At Month 3) | 47 [39.51 to 54.21] | 22 [15.92 to 28.26] | 9 [4.67 to 15.81] | 4 [0.98 to 8.89] | 9 [4.44 to 15.08] | 19 [12.45 to 26.30]
  NZ98/254 Strain ≥ 2-fold (At Month 7) | 19 [13.32 to 24.93] | 12 [8.05 to 18.07] | 11 [5.90 to 17.81] | 45 [35.24 to 54.33] | 7 [3.32 to 13.13] | 54 [44.92 to 62.38]
  NZ98/254 Strain ≥ 3-fold (At Month 7) | 11 [7.05 to 16.57] | 10 [6.30 to 15.57] | 7 [2.92 to 12.71] | 33 [24.44 to 42.56] | 6 [2.78 to 12.13] | 43 [34.76 to 52.11]
  NZ98/254 Strain ≥ 4-fold (At Month 7) | 9 [5.36 to 14.08] | 8 [4.61 to 13.02] | 6 [2.38 to 11.65] | 24 [16.53 to 33.10] | 4 [1.30 to 9.02] | 33 [24.97 to 41.47]
  NZ98/254 Strain ≥ 2-fold (At Month 13) | 11 [6.62 to 15.95] | 9 [5.44 to 14.30] | 7 [2.92 to 12.71] | 10 [5.01 to 16.89] | 49 [40.19 to 58.26] | 14 [8.76 to 21.25]
  NZ98/254 Strain ≥ 3-fold (At Month 13) | 5 [2.58 to 9.56] | 7 [3.79 to 11.72] | 6 [2.38 to 11.65] | 9 [4.36 to 15.81] | 37 [28.12 to 45.55] | 7 [3.64 to 13.30]
  NZ98/254 Strain ≥ 4-fold (At Month 13) | 4 [1.85 to 8.21] | 5 [2.62 to 9.72] | 5 [1.86 to 10.57] | 6 [2.55 to 12.45] | 26 [18.76 to 34.77] | 4 [1.66 to 9.49]
  M14459 Strain ≥ 2-fold (At Month 2): number analyzed (Participants) | 184 | 179 | 112 | 108 | 123 | 137
  M14459 Strain ≥ 2-fold (At Month 2) | 14 [9.44 to 20.02] | 13 [8.32 to 18.65] | 34 [25.25 to 43.48] | 8 [3.88 to 15.23] | 23 [15.69 to 31.19] | 11 [6.40 to 17.79]
  M14459 Strain ≥ 3-fold (At Month 2): number analyzed (Participants) | 184 | 179 | 112 | 108 | 123 | 137
  M14459 Strain ≥ 3-fold (At Month 2) | 10 [5.90 to 15.02] | 10 [6.07 to 15.43] | 23 [15.76 to 32.14] | 6 [2.07 to 11.70] | 15 [9.56 to 23.07] | 6 [2.61 to 11.42]
  M14459 Strain ≥ 4-fold (At Month 2): number analyzed (Participants) | 184 | 179 | 112 | 108 | 123 | 137
  M14459 Strain ≥ 4-fold (At Month 2) | 7 [3.82 to 11.78] | 6 [2.71 to 10.03] | 15 [9.10 to 23.19] | 4 [1.02 to 9.21] | 12 [6.99 to 19.32] | 4 [1.22 to 8.49]
  M14459 Strain ≥ 2-fold (At Month 3): number analyzed (Participants) | 184 | 179 | 112 | 108 | 123 | 137
  M14459 Strain ≥ 2-fold (At Month 3) | 65 [57.86 to 72.07] | 50 [42.72 to 57.82] | 24 [16.53 to 33.10] | 6 [2.65 to 12.90] | 14 [8.26 to 21.20] | 50 [41.25 to 58.75]
  M14459 Strain ≥ 3-fold (At Month 3): number analyzed (Participants) | 184 | 179 | 112 | 108 | 123 | 137
  M14459 Strain ≥ 3-fold (At Month 3) | 49 [41.49 to 56.37] | 39 [31.38 to 46.10] | 10 [5.01 to 16.89] | 3 [0.58 to 7.90] | 11 [5.75 to 17.40] | 39 [30.52 to 47.60]
  M14459 Strain ≥ 4-fold (At Month 3): number analyzed (Participants) | 184 | 179 | 112 | 108 | 123 | 137
  M14459 Strain ≥ 4-fold (At Month 3) | 38 [30.49 to 44.92] | 28 [22.01 to 35.70] | 4 [1.47 to 10.11] | 3 [0.58 to 7.90] | 7 [3.40 to 13.44] | 28 [20.24 to 36.00]
  M14459 Strain ≥ 2-fold (At Month 7): number analyzed (Participants) | 184 | 179 | 112 | 108 | 123 | 137
  M14459 Strain ≥ 2-fold (At Month 7) | 16 [11.28 to 22.45] | 14 [9.25 to 19.92] | 9 [4.36 to 15.81] | 69 [58.88 to 77.12] | 7 [2.85 to 12.41] | 72 [63.21 to 79.09]
  M14459 Strain ≥ 3-fold (At Month 7): number analyzed (Participants) | 184 | 179 | 112 | 108 | 123 | 137
  M14459 Strain ≥ 3-fold (At Month 7) | 12 [7.65 to 17.54] | 7 [3.92 to 12.10] | 6 [2.55 to 12.45] | 55 [44.76 to 64.24] | 6 [2.32 to 11.37] | 54 [45.65 to 63.10]
  M14459 Strain ≥ 4-fold (At Month 7): number analyzed (Participants) | 184 | 179 | 112 | 108 | 123 | 137
  M14459 Strain ≥ 4-fold (At Month 7) | 8 [4.22 to 12.44] | 6 [3.11 to 10.73] | 4 [0.98 to 8.89] | 48 [38.43 to 57.97] | 5 [1.81 to 10.32] | 49 [39.79 to 57.29]
  M14459 Strain ≥ 2-fold (At Month 13): number analyzed (Participants) | 184 | 179 | 112 | 108 | 123 | 137
  M14459 Strain ≥ 2-fold (At Month 13) | 11 [7.21 to 16.92] | 9 [5.63 to 14.77] | 6 [2.55 to 12.45] | 10 [5.20 to 17.49] | 74 [65.30 to 81.48] | 12 [6.98 to 18.67]
  M14459 Strain ≥ 3-fold (At Month 13): number analyzed (Participants) | 184 | 179 | 112 | 108 | 123 | 137
  M14459 Strain ≥ 3-fold (At Month 13) | 8 [4.22 to 12.44] | 4 [1.95 to 8.62] | 4 [1.47 to 10.11] | 7 [3.25 to 14.07] | 59 [50.12 to 68.11] | 6 [2.61 to 11.42]
  M14459 Strain ≥ 4-fold (At Month 13): number analyzed (Participants) | 184 | 179 | 112 | 108 | 123 | 137
  M14459 Strain ≥ 4-fold (At Month 13) | 3 [1.21 to 6.96] | 4 [1.59 to 7.89] | 3 [0.56 to 7.63] | 6 [2.07 to 11.70] | 51 [42.05 to 60.33] | 4 [1.66 to 9.49]
  M07-0241084 Strain ≥ 2-fold (At Month 2): number analyzed (Participants) | 188 | 176 | 117 | 113 | 121 | 128
  M07-0241084 Strain ≥ 2-fold (At Month 2) | 16 [11.49 to 22.58] | 11 [6.63 to 16.34] | 20 [12.89 to 28.02] | 5 [1.97 to 11.20] | 19 [12.45 to 27.14] | 8 [3.81 to 13.90]
  M07-0241084 Strain ≥ 3-fold (At Month 2): number analyzed (Participants) | 188 | 176 | 117 | 113 | 121 | 128
  M07-0241084 Strain ≥ 3-fold (At Month 2) | 12 [7.92 to 17.79] | 7 [3.57 to 11.61] | 9 [4.79 to 16.20] | 2 [0.22 to 6.25] | 12 [6.47 to 18.65] | 4 [1.28 to 8.88]
  M07-0241084 Strain ≥ 4-fold (At Month 2): number analyzed (Participants) | 188 | 176 | 117 | 113 | 121 | 128
  M07-0241084 Strain ≥ 4-fold (At Month 2) | 8 [4.53 to 12.82] | 5 [1.98 to 8.76] | 7 [3.00 to 13.03] | 2 [0.22 to 6.25] | 9 [4.63 to 15.68] | 1 [0.02 to 4.28]
  M07-0241084 Strain ≥ 2-fold (At Month 3): number analyzed (Participants) | 188 | 176 | 117 | 113 | 121 | 128
  M07-0241084 Strain ≥ 2-fold (At Month 3) | 37 [29.81 to 44.02] | 22 [16.26 to 29.02] | 11 [6.05 to 18.25] | 2 [0.22 to 6.25] | 8 [4.03 to 14.67] | 21 [14.38 to 29.19]
  M07-0241084 Strain ≥ 3-fold (At Month 3): number analyzed (Participants) | 188 | 176 | 117 | 113 | 121 | 128
  M07-0241084 Strain ≥ 3-fold (At Month 3) | 28 [21.40 to 34.64] | 12 [7.54 to 17.66] | 7 [3.00 to 13.03] | 1 [0.02 to 4.83] | 5 [1.84 to 10.48] | 17 [11.10 to 24.86]
  M07-0241084 Strain ≥ 4-fold (At Month 3): number analyzed (Participants) | 188 | 176 | 117 | 113 | 121 | 128
  M07-0241084 Strain ≥ 4-fold (At Month 3) | 19 [13.32 to 24.93] | 9 [5.29 to 14.34] | 4 [1.40 to 9.69] | 0 [0 to 3.21] | 4 [1.36 to 9.38] | 13 [7.93 to 20.41]
  M07-0241084 Strain ≥ 2-fold (At Month 7): number analyzed (Participants) | 188 | 176 | 117 | 113 | 121 | 128
  M07-0241084 Strain ≥ 2-fold (At Month 7) | 19 [13.32 to 24.93] | 13 [8.00 to 18.31] | 8 [3.58 to 14.10] | 43 [34.07 to 53.01] | 4 [1.36 to 9.38] | 42 [33.51 to 51.23]
  M07-0241084 Strain ≥ 3-fold (At Month 7): number analyzed (Participants) | 188 | 176 | 117 | 113 | 121 | 128
  M07-0241084 Strain ≥ 3-fold (At Month 7) | 11 [7.05 to 16.57] | 7 [3.99 to 12.30] | 6 [2.44 to 11.94] | 31 [22.61 to 40.36] | 1 [0.02 to 4.52] | 32 [24.06 to 40.85]
  M07-0241084 Strain ≥ 4-fold (At Month 7): number analyzed (Participants) | 188 | 176 | 117 | 113 | 121 | 128
  M07-0241084 Strain ≥ 4-fold (At Month 7) | 7 [4.13 to 12.18] | 6 [2.76 to 10.20] | 3 [0.94 to 8.52] | 19 [12.62 to 27.98] | 1 [0.02 to 4.52] | 22 [15.05 to 30.04]
  M07-0241084 Strain ≥ 2-fold (At Month 13): number analyzed (Participants) | 188 | 176 | 117 | 113 | 121 | 128
  M07-0241084 Strain ≥ 2-fold (At Month 13) | 13 [8.35 to 18.40] | 11 [7.08 to 17.00] | 8 [3.58 to 14.10] | 13 [7.62 to 20.95] | 41 [32.45 to 50.63] | 15 [9.18 to 22.21]
  M07-0241084 Strain ≥ 3-fold (At Month 13): number analyzed (Participants) | 188 | 176 | 117 | 113 | 121 | 128
  M07-0241084 Strain ≥ 3-fold (At Month 13) | 9 [4.94 to 13.45] | 7 [3.99 to 12.30] | 5 [1.90 to 10.83] | 9 [4.33 to 15.67] | 34 [25.53 to 43.05] | 10 [5.52 to 16.74]
  M07-0241084 Strain ≥ 4-fold (At Month 13): number analyzed (Participants) | 188 | 176 | 117 | 113 | 121 | 128
  M07-0241084 Strain ≥ 4-fold (At Month 13) | 5 [2.58 to 9.56] | 6 [2.76 to 10.20] | 4 [1.40 to 9.69] | 6 [2.53 to 12.35] | 21 [13.84 to 28.97] | 6 [2.74 to 11.94]
  96217 Strain ≥ 2-fold (At Month 2): number analyzed (Participants) | 186 | 178 | 120 | 112 | 128 | 121
  96217 Strain ≥ 2-fold (At Month 2) | 34 [27.61 to 41.71] | 29 [22.65 to 36.48] | 88 [81.20 to 93.47] | 32 [23.63 to 41.63] | 31 [23.35 to 40.04] | 26 [18.84 to 35.24]
  96217 Strain ≥ 3-fold (At Month 2): number analyzed (Participants) | 186 | 178 | 120 | 112 | 128 | 121
  96217 Strain ≥ 3-fold (At Month 2) | 26 [19.68 to 32.72] | 20 [14.09 to 26.27] | 81 [72.64 to 87.44] | 19 [12.00 to 27.22] | 18 [11.74 to 25.73] | 19 [12.45 to 27.14]
  96217 Strain ≥ 4-fold (At Month 2): number analyzed (Participants) | 186 | 178 | 120 | 112 | 128 | 121
  96217 Strain ≥ 4-fold (At Month 2) | 18 [12.54 to 24.00] | 13 [8.37 to 18.76] | 76 [67.17 to 83.18] | 12 [6.33 to 19.03] | 14 [8.55 to 21.31] | 16 [9.73 to 23.43]
  96217 Strain ≥ 2-fold (At Month 3): number analyzed (Participants) | 186 | 178 | 120 | 112 | 128 | 121
  96217 Strain ≥ 2-fold (At Month 3) | 97 [93.84 to 99.12] | 92 [87.16 to 95.63] | 85 [77.33 to 90.86] | 28 [19.64 to 36.93] | 23 [16.41 to 31.74] | 91 [84.32 to 95.37]
  96217 Strain ≥ 3-fold (At Month 3): number analyzed (Participants) | 186 | 178 | 120 | 112 | 128 | 121
  96217 Strain ≥ 3-fold (At Month 3) | 96 [92.40 to 98.47] | 89 [83.18 to 93.00] | 76 [67.17 to 83.18] | 14 [8.39 to 22.16] | 17 [11.10 to 24.86] | 88 [81.35 to 93.53]
  96217 Strain ≥ 4-fold (At Month 3): number analyzed (Participants) | 186 | 178 | 120 | 112 | 128 | 121
  96217 Strain ≥ 4-fold (At Month 3) | 94 [89.66 to 97.01] | 83 [76.20 to 87.85] | 69 [60.09 to 77.27] | 11 [5.66 to 17.97] | 13 [7.93 to 20.41] | 83 [75.63 to 89.60]
  96217 Strain ≥ 2-fold (At Month 7): number analyzed (Participants) | 186 | 178 | 120 | 112 | 128 | 121
  96217 Strain ≥ 2-fold (At Month 7) | 81 [74.81 to 86.53] | 74 [66.48 to 79.91] | 64 [54.90 to 72.71] | 96 [91.11 to 99.02] | 16 [10.45 to 23.98] | 97 [91.75 to 99.09]
  96217 Strain ≥ 3-fold (At Month 7): number analyzed (Participants) | 186 | 178 | 120 | 112 | 128 | 121
  96217 Strain ≥ 3-fold (At Month 7) | 73 [65.57 to 78.85] | 63 [55.38 to 70.03] | 52 [42.37 to 60.88] | 96 [91.11 to 99.02] | 9 [4.94 to 15.80] | 96 [90.62 to 98.64]
  96217 Strain ≥ 4-fold (At Month 7): number analyzed (Participants) | 186 | 178 | 120 | 112 | 128 | 121
  96217 Strain ≥ 4-fold (At Month 7) | 61 [53.89 to 68.33] | 50 [42.43 to 57.57] | 42 [32.74 to 51.02] | 95 [88.70 to 98.01] | 7 [3.27 to 12.93] | 94 [88.44 to 97.64]
  96217 Strain ≥ 2-fold (At Month 13): number analyzed (Participants) | 186 | 178 | 120 | 112 | 128 | 121
  96217 Strain ≥ 2-fold (At Month 13) | 65 [57.73 to 71.88] | 54 [46.32 to 61.42] | 52 [42.37 to 60.88] | 72 [63.07 to 80.36] | 96 [91.12 to 98.72] | 77 [68.32 to 84.04]
  96217 Strain ≥ 3-fold (At Month 13): number analyzed (Participants) | 186 | 178 | 120 | 112 | 128 | 121
  96217 Strain ≥ 3-fold (At Month 13) | 53 [45.78 to 60.56] | 39 [32.10 to 46.91] | 34 [25.76 to 43.38] | 54 [44.78 to 63.90] | 95 [89.06 to 97.77] | 62 [52.71 to 70.65]
  96217 Strain ≥ 4-fold (At Month 13): number analyzed (Participants) | 186 | 178 | 120 | 112 | 128 | 121
  96217 Strain ≥ 4-fold (At Month 13) | 35 [28.62 to 42.82] | 22 [16.57 to 29.32] | 28 [19.75 to 36.40] | 45 [35.24 to 54.33] | 93 [87.07 to 96.73] | 51 [41.99 to 60.43]
  A human Serogroup ≥ 2-fold (At Month 2): number analyzed (Participants) | 172 | 178 | 107 | 105 | 120 | 127
  A human Serogroup ≥ 2-fold (At Month 2) | 12 [7.72 to 18.06] | 23 [17.07 to 29.92] | 78 [68.49 to 85.07] | 21 [13.62 to 29.99] | 38 [28.83 to 46.80] | 17 [10.54 to 24.16]
  A human Serogroup ≥ 3-fold (At Month 2): number analyzed (Participants) | 172 | 178 | 107 | 105 | 120 | 127
  A human Serogroup ≥ 3-fold (At Month 2) | 9 [5.41 to 14.67] | 16 [11.19 to 22.55] | 64 [53.69 to 72.64] | 14 [8.22 to 22.47] | 30 [21.98 to 39.04] | 13 [7.38 to 19.65]
  A human Serogroup ≥ 4-fold (At Month 2): number analyzed (Participants) | 172 | 178 | 107 | 105 | 120 | 127
  A human Serogroup ≥ 4-fold (At Month 2) | 6 [2.82 to 10.43] | 11 [6.55 to 16.17] | 50 [39.72 to 59.37] | 11 [6.05 to 19.11] | 20 [13.25 to 28.28] | 7 [3.29 to 13.03]
  A human Serogroup ≥ 2-fold (At Month 3): number analyzed (Participants) | 172 | 178 | 107 | 105 | 120 | 127
  A human Serogroup ≥ 2-fold (At Month 3) | 80 [72.85 to 85.40] | 71 [63.52 to 77.35] | 61 [50.84 to 70.05] | 20 [12.83 to 28.93] | 24 [16.82 to 32.83] | 74 [65.49 to 81.39]
  A human Serogroup ≥ 3-fold (At Month 3): number analyzed (Participants) | 172 | 178 | 107 | 105 | 120 | 127
  A human Serogroup ≥ 3-fold (At Month 3) | 66 [58.09 to 72.76] | 52 [44.64 to 59.77] | 41 [31.70 to 51.05] | 12 [6.76 to 20.24] | 18 [11.86 to 26.43] | 56 [46.83 to 64.70]
  A human Serogroup ≥ 4-fold (At Month 3): number analyzed (Participants) | 172 | 178 | 107 | 105 | 120 | 127
  A human Serogroup ≥ 4-fold (At Month 3) | 56 [48.64 to 63.93] | 42 [34.79 to 49.75] | 31 [22.27 to 40.50] | 7 [2.72 to 13.25] | 14 [8.47 to 21.71] | 40 [31.56 to 49.22]
  A human Serogroup ≥ 2-fold (At Month 7): number analyzed (Participants) | 172 | 178 | 107 | 105 | 120 | 127
  A human Serogroup ≥ 2-fold (At Month 7) | 27 [20.82 to 34.63] | 28 [21.11 to 34.71] | 25 [17.33 to 34.55] | 87 [78.64 to 92.51] | 8 [3.49 to 13.76] | 88 [81.27 to 93.24]
  A human Serogroup ≥ 3-fold (At Month 7): number analyzed (Participants) | 172 | 178 | 107 | 105 | 120 | 127
  A human Serogroup ≥ 3-fold (At Month 7) | 17 [11.59 to 23.31] | 16 [11.19 to 22.55] | 16 [9.54 to 24.21] | 76 [66.89 to 83.96] | 6 [2.38 to 11.65] | 77 [68.88 to 84.14]
  A human Serogroup ≥ 4-fold (At Month 7): number analyzed (Participants) | 172 | 178 | 107 | 105 | 120 | 127
  A human Serogroup ≥ 4-fold (At Month 7) | 11 [6.78 to 16.71] | 10 [5.66 to 14.85] | 13 [7.34 to 20.98] | 70 [60.78 to 78.98] | 5 [1.86 to 10.57] | 70 [61.32 to 77.88]
  A human Serogroup ≥ 2-fold (At Month 13): number analyzed (Participants) | 172 | 178 | 107 | 105 | 120 | 127
  A human Serogroup ≥ 2-fold (At Month 13) | 16 [10.61 to 22.01] | 12 [7.91 to 18.11] | 18 [11.04 to 26.33] | 31 [22.72 to 41.22] | 85 [77.33 to 90.86] | 28 [20.71 to 37.02]
  A human Serogroup ≥ 3-fold (At Month 13): number analyzed (Participants) | 172 | 178 | 107 | 105 | 120 | 127
  A human Serogroup ≥ 3-fold (At Month 13) | 9 [5.41 to 14.67] | 8 [4.37 to 12.84] | 11 [5.93 to 18.77] | 25 [16.86 to 34.14] | 80 [71.72 to 86.75] | 15 [9.25 to 22.37]
  A human Serogroup ≥ 4-fold (At Month 13): number analyzed (Participants) | 172 | 178 | 107 | 105 | 120 | 127
  A human Serogroup ≥ 4-fold (At Month 13) | 5 [2.42 to 9.70] | 4 [1.60 to 7.93] | 9 [4.57 to 16.52] | 15 [8.97 to 23.56] | 78 [68.98 to 84.62] | 7 [3.29 to 13.03]
  C human Serogroup ≥ 2-fold (At Month 2): number analyzed (Participants) | 186 | 185 | 122 | 114 | 123 | 130
  C human Serogroup ≥ 2-fold (At Month 2) | 24 [18.23 to 31.00] | 64 [56.41 to 70.71] | 95 [89.60 to 98.17] | 55 [45.66 to 64.58] | 73 [64.43 to 80.76] | 62 [52.61 to 69.93]
  C human Serogroup ≥ 3-fold (At Month 2): number analyzed (Participants) | 186 | 185 | 122 | 114 | 123 | 130
  C human Serogroup ≥ 3-fold (At Month 2) | 15 [10.24 to 21.02] | 50 [42.84 to 57.69] | 91 [84.44 to 95.41] | 48 [38.79 to 57.80] | 59 [49.31 to 67.35] | 54 [44.89 to 62.62]
  C human Serogroup ≥ 4-fold (At Month 2): number analyzed (Participants) | 186 | 185 | 122 | 114 | 123 | 130
  C human Serogroup ≥ 4-fold (At Month 2) | 9 [5.00 to 13.59] | 42 [34.43 to 49.08] | 88 [80.53 to 92.95] | 44 [34.58 to 53.46] | 50 [40.46 to 58.75] | 42 [32.97 to 50.51]
  C human Serogroup ≥ 2-fold (At Month 3): number analyzed (Participants) | 186 | 185 | 122 | 114 | 123 | 130
  C human Serogroup ≥ 2-fold (At Month 3) | 80 [73.05 to 85.12] | 94 [89.61 to 96.99] | 93 [86.46 to 96.57] | 58 [48.29 to 67.08] | 65 [55.92 to 73.42] | 98 [93.40 to 99.52]
  C human Serogroup ≥ 3-fold (At Month 3): number analyzed (Participants) | 186 | 185 | 122 | 114 | 123 | 130
  C human Serogroup ≥ 3-fold (At Month 3) | 64 [56.63 to 70.87] | 90 [85.06 to 94.13] | 90 [83.45 to 94.81] | 47 [37.94 to 56.94] | 50 [40.46 to 58.75] | 96 [91.25 to 98.74]
  C human Serogroup ≥ 4-fold (At Month 3): number analyzed (Participants) | 186 | 185 | 122 | 114 | 123 | 130
  C human Serogroup ≥ 4-fold (At Month 3) | 49 [41.54 to 56.34] | 87 [81.31 to 91.51] | 83 [74.90 to 89.02] | 41 [32.09 to 50.83] | 42 [33.42 to 51.51] | 92 [85.36 to 95.70]
  C human Serogroup ≥ 2-fold (At Month 7): number analyzed (Participants) | 186 | 185 | 122 | 114 | 123 | 130
  C human Serogroup ≥ 2-fold (At Month 7) | 29 [22.62 to 36.12] | 86 [80.70 to 91.06] | 89 [81.50 to 93.58] | 97 [92.50 to 99.45] | 50 [40.46 to 58.75] | 98 [94.55 to 99.81]
  C human Serogroup ≥ 3-fold (At Month 7): number analyzed (Participants) | 186 | 185 | 122 | 114 | 123 | 130
  C human Serogroup ≥ 3-fold (At Month 7) | 16 [10.70 to 21.62] | 80 [73.50 to 85.51] | 79 [70.35 to 85.58] | 94 [87.76 to 97.50] | 37 [28.09 to 45.75] | 98 [94.55 to 99.81]
  C human Serogroup ≥ 4-fold (At Month 7): number analyzed (Participants) | 186 | 185 | 122 | 114 | 123 | 130
  C human Serogroup ≥ 4-fold (At Month 7) | 10 [6.26 to 15.49] | 71 [64.26 to 77.75] | 72 [63.29 to 79.87] | 92 [85.54 to 96.33] | 28 [19.96 to 36.43] | 98 [93.40 to 99.52]
  C human Serogroup ≥ 2-fold (At Month 13): number analyzed (Participants) | 186 | 185 | 122 | 114 | 123 | 130
  C human Serogroup ≥ 2-fold (At Month 13) | 19 [13.94 to 25.77] | 73 [65.97 to 79.23] | 74 [65.04 to 81.32] | 82 [73.23 to 88.22] | 97 [91.88 to 99.11] | 92 [86.31 to 96.25]
  C human Serogroup ≥ 3-fold (At Month 13): number analyzed (Participants) | 186 | 185 | 122 | 114 | 123 | 130
  C human Serogroup ≥ 3-fold (At Month 13) | 13 [8.89 to 19.20] | 64 [56.41 to 70.71] | 61 [52.24 to 70.14] | 70 [60.89 to 78.38] | 96 [90.77 to 98.67] | 89 [82.59 to 93.99]
  C human Serogroup ≥ 4-fold (At Month 13): number analyzed (Participants) | 186 | 185 | 122 | 114 | 123 | 130
  C human Serogroup ≥ 4-fold (At Month 13) | 10 [5.84 to 14.86] | 51 [43.91 to 58.75] | 53 [44.03 to 62.36] | 56 [46.54 to 65.42] | 93 [87.59 to 97.15] | 85 [77.24 to 90.34]
  W human Serogroup ≥ 2-fold (At Month 2): number analyzed (Participants) | 162 | 180 | 119 | 108 | 123 | 123
  W human Serogroup ≥ 2-fold (At Month 2) | 24 [17.71 to 31.41] | 32 [24.95 to 39.00] | 65 [55.42 to 73.24] | 35 [26.24 to 44.96] | 50 [41.25 to 59.54] | 33 [25.09 to 42.40]
  W human Serogroup ≥ 3-fold (At Month 2): number analyzed (Participants) | 162 | 180 | 119 | 108 | 123 | 123
  W human Serogroup ≥ 3-fold (At Month 2) | 17 [11.28 to 23.31] | 19 [13.93 to 25.99] | 52 [42.75 to 61.34] | 25 [17.17 to 34.25] | 40 [31.12 to 49.05] | 22 [14.99 to 30.31]
  W human Serogroup ≥ 4-fold (At Month 2): number analyzed (Participants) | 162 | 180 | 119 | 108 | 123 | 123
  W human Serogroup ≥ 4-fold (At Month 2) | 11 [6.72 to 16.99] | 16 [11.06 to 22.31] | 42 [33.03 to 51.41] | 18 [10.94 to 26.10] | 34 [25.84 to 43.24] | 18 [11.56 to 25.82]
  W human Serogroup ≥ 2-fold (At Month 3): number analyzed (Participants) | 162 | 180 | 119 | 108 | 123 | 123
  W human Serogroup ≥ 2-fold (At Month 3) | 67 [59.48 to 74.44] | 78 [71.59 to 84.12] | 55 [46.07 to 64.57] | 34 [25.40 to 44.01] | 46 [37.31 to 55.56] | 76 [67.93 to 83.61]
  W human Serogroup ≥ 3-fold (At Month 3): number analyzed (Participants) | 162 | 180 | 119 | 108 | 123 | 123
  W human Serogroup ≥ 3-fold (At Month 3) | 54 [46.32 to 62.16] | 65 [57.55 to 71.95] | 39 [29.87 to 48.02] | 23 [15.57 to 32.25] | 34 [25.84 to 43.24] | 67 [58.45 to 75.65]
  W human Serogroup ≥ 4-fold (At Month 3): number analyzed (Participants) | 162 | 180 | 119 | 108 | 123 | 123
  W human Serogroup ≥ 4-fold (At Month 3) | 43 [34.87 to 50.59] | 57 [49.09 to 64.02] | 30 [22.17 to 39.35] | 19 [12.46 to 28.17] | 28 [20.69 to 37.29] | 56 [46.87 to 65.03]
  W human Serogroup ≥ 2-fold (At Month 7): number analyzed (Participants) | 162 | 180 | 119 | 108 | 123 | 123
  W human Serogroup ≥ 2-fold (At Month 7) | 31 [24.42 to 39.23] | 51 [43.57 to 58.62] | 43 [33.83 to 52.25] | 90 [82.51 to 94.80] | 41 [31.89 to 49.88] | 89 [81.64 to 93.64]
  W human Serogroup ≥ 3-fold (At Month 7): number analyzed (Participants) | 162 | 180 | 119 | 108 | 123 | 123
  W human Serogroup ≥ 3-fold (At Month 7) | 22 [15.53 to 28.74] | 30 [23.41 to 37.26] | 29 [20.67 to 37.57] | 81 [71.83 to 87.54] | 28 [19.96 to 36.43] | 80 [72.37 to 87.08]
  W human Serogroup ≥ 4-fold (At Month 7): number analyzed (Participants) | 162 | 180 | 119 | 108 | 123 | 123
  W human Serogroup ≥ 4-fold (At Month 7) | 13 [8.21 to 19.13] | 21 [14.91 to 27.20] | 17 [10.58 to 24.76] | 73 [63.76 to 81.22] | 20 [13.61 to 28.52] | 73 [64.43 to 80.76]
  W human Serogroup ≥ 2-fold (At Month 13): number analyzed (Participants) | 162 | 180 | 119 | 108 | 123 | 123
  W human Serogroup ≥ 2-fold (At Month 13) | 20 [13.92 to 26.73] | 26 [19.36 to 32.58] | 32 [23.69 to 41.10] | 56 [46.60 to 66.00] | 94 [88.63 to 97.68] | 61 [51.77 to 69.64]
  W human Serogroup ≥ 3-fold (At Month 13): number analyzed (Participants) | 162 | 180 | 119 | 108 | 123 | 123
  W human Serogroup ≥ 3-fold (At Month 13) | 9 [4.81 to 14.07] | 13 [8.28 to 18.55] | 17 [10.58 to 24.76] | 38 [28.80 to 47.81] | 92 [85.56 to 96.03] | 46 [36.53 to 54.75]
  W human Serogroup ≥ 4-fold (At Month 13): number analyzed (Participants) | 162 | 180 | 119 | 108 | 123 | 123
  W human Serogroup ≥ 4-fold (At Month 13) | 7 [3.44 to 11.82] | 11 [6.48 to 15.99] | 13 [7.88 to 20.91] | 27 [18.78 to 36.24] | 89 [82.60 to 94.25] | 29 [21.41 to 38.15]
  Y human Serogroup ≥ 2-fold (At Month 2): number analyzed (Participants) | 188 | 180 | 120 | 110 | 127 | 137
  Y human Serogroup ≥ 2-fold (At Month 2) | 6 [2.96 to 10.23] | 49 [41.38 to 56.43] | 74 [65.38 to 81.72] | 47 [37.68 to 57.02] | 53 [43.70 to 61.68] | 51 [42.42 to 59.73]
  Y human Serogroup ≥ 3-fold (At Month 2): number analyzed (Participants) | 188 | 180 | 120 | 110 | 127 | 137
  Y human Serogroup ≥ 3-fold (At Month 2) | 4 [1.51 to 7.52] | 39 [32.25 to 46.99] | 64 [54.90 to 72.71] | 40 [30.78 to 49.78] | 41 [32.30 to 50.02] | 43 [34.64 to 51.80]
  Y human Serogroup ≥ 4-fold (At Month 2): number analyzed (Participants) | 188 | 180 | 120 | 110 | 127 | 137
  Y human Serogroup ≥ 4-fold (At Month 2) | 2 [0.58 to 5.36] | 32 [25.46 to 39.58] | 58 [48.15 to 66.47] | 33 [24.08 to 42.33] | 36 [27.88 to 45.22] | 37 [29.13 to 45.89]
  Y human Serogroup ≥ 2-fold (At Month 3): number analyzed (Participants) | 188 | 180 | 120 | 110 | 127 | 137
  Y human Serogroup ≥ 2-fold (At Month 3) | 10 [5.77 to 14.71] | 84 [78.31 to 89.41] | 66 [56.62 to 74.24] | 45 [35.93 to 55.23] | 46 [36.81 to 54.74] | 83 [75.88 to 89.05]
  Y human Serogroup ≥ 3-fold (At Month 3): number analyzed (Participants) | 188 | 180 | 120 | 110 | 127 | 137
  Y human Serogroup ≥ 3-fold (At Month 3) | 7 [3.73 to 11.53] | 80 [73.40 to 85.58] | 55 [45.65 to 64.09] | 35 [25.74 to 44.21] | 35 [26.43 to 43.60] | 75 [67.08 to 82.16]
  Y human Serogroup ≥ 4-fold (At Month 3): number analyzed (Participants) | 188 | 180 | 120 | 110 | 127 | 137
  Y human Serogroup ≥ 4-fold (At Month 3) | 4 [1.85 to 8.21] | 68 [61.00 to 75.05] | 48 [39.12 to 57.63] | 29 [20.82 to 38.52] | 31 [23.55 to 40.33] | 66 [57.86 to 74.26]
  Y human Serogroup ≥ 2-fold (At Month 7): number analyzed (Participants) | 188 | 180 | 120 | 110 | 127 | 137
  Y human Serogroup ≥ 2-fold (At Month 7) | 5 [2.21 to 8.89] | 60 [52.45 to 67.22] | 51 [41.55 to 60.07] | 90 [82.81 to 94.90] | 39 [30.08 to 47.63] | 92 [86.09 to 95.92]
  Y human Serogroup ≥ 3-fold (At Month 7): number analyzed (Participants) | 188 | 180 | 120 | 110 | 127 | 137
  Y human Serogroup ≥ 3-fold (At Month 7) | 3 [1.18 to 6.82] | 48 [40.29 to 55.34] | 44 [35.11 to 53.52] | 83 [74.35 to 89.27] | 28 [20.71 to 37.02] | 87 [80.03 to 92.02]
  Y human Serogroup ≥ 4-fold (At Month 7): number analyzed (Participants) | 188 | 180 | 120 | 110 | 127 | 137
  Y human Serogroup ≥ 4-fold (At Month 7) | 3 [0.87 to 6.10] | 41 [33.31 to 48.11] | 38 [29.61 to 47.65] | 79 [70.30 to 86.26] | 23 [15.86 to 31.12] | 76 [67.87 to 82.80]
  Y human Serogroup ≥ 2-fold (At Month 13): number analyzed (Participants) | 188 | 180 | 120 | 110 | 127 | 137
  Y human Serogroup ≥ 2-fold (At Month 13) | 5 [2.21 to 8.89] | 43 [35.45 to 50.35] | 38 [29.61 to 47.65] | 60 [50.22 to 69.22] | 94 [88.97 to 97.76] | 72 [63.20 to 78.91]
  Y human Serogroup ≥ 3-fold (At Month 13): number analyzed (Participants) | 188 | 180 | 120 | 110 | 127 | 137
  Y human Serogroup ≥ 3-fold (At Month 13) | 3 [1.18 to 6.82] | 34 [27.01 to 41.30] | 28 [20.49 to 37.28] | 48 [38.55 to 57.91] | 91 [84.08 to 95.02] | 54 [45.30 to 62.56]
  Y human Serogroup ≥ 4-fold (At Month 13): number analyzed (Participants) | 188 | 180 | 120 | 110 | 127 | 137
  Y human Serogroup ≥ 4-fold (At Month 13) | 2 [0.58 to 5.36] | 25 [18.86 to 31.99] | 23 [16.10 to 31.93] | 45 [35.93 to 55.23] | 89 [82.20 to 93.84] | 47 [38.15 to 55.43]

19. Secondary Outcome: The Area Under the Curve (AUC) for Percentage of Subjects With hSBA Titers ≥LLQ for All Serogroups and Strains.
Description: The area under the curve for percentage of subjects with hSBA titers ≥ LLQ for all serogroups (A, C, W and Y) and for all serogroup B test strains (M14459, 96217, NZ98/254 and M07-0241084) was summarized overall (from Month 0 to Month 13) and by period (from Month 0 to Month 2, Month 2 to Month 3, Month 3 to Month 7 and Month 7 to Month 13) by vaccine groups. It was computed as the sum of the trapezoidal areas and the time unit used was the month. AUC 0_13 = (r0+r2)(2-0)/2 + (r2+r3)(3-2)/2 + (r3+r7)(7-3)/2 + (r7+r13)(13-7)/2 with ri = percentages of subjects with both hSBA titers >= LLQ against N. meningitis for all serogroups A, C, W and Y and for all serogroup B test strains at Month 1.
Time Frame: From Month 0 to Month 13
Population: Analysis was done on the FAS Month 13 Over Time. All subjects in All Enrolled Set who received a study meningococcal vaccination & provided evaluable serum samples at one month after the last meningococcal vaccination whose result is available for at least one A,C,W,or Y serogroup or serogroup B test strain.
Measure: Number; unit: Percentage of subjects
Arm/Group | rMenB_0_2 Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group | ABCWY_0_2_6 Group
Number analyzed (Participants) | 200 | 196 | 131 | 118 | 132 | 140
Percentage of subjects
  Serogroup A- Month 0-2 (LLQ-22.7): number analyzed (Participants) | 191 | 189 | 129 | 113 | 126 | 140
  Serogroup A- Month 0-2 (LLQ-22.7) | 26.52 | 38.01 | 98.62 | 38.05 | 57.12 | 27.86
  Serogroup A- Month 2-3 (LLQ-22.7): number analyzed (Participants) | 197 | 193 | 125 | 118 | 130 | 135
  Serogroup A- Month 2-3 (LLQ-22.7) | 57.69 | 60.98 | 86.91 | 33.40 | 47.00 | 59.13
  Serogroup A- Month 3-7 (LLQ-22.7): number analyzed (Participants) | 191 | 194 | 124 | 118 | 127 | 136
  Serogroup A- Month 3-7 (LLQ-22.7) | 292.53 | 264.81 | 243.86 | 252.54 | 119.41 | 370.46
  Serogroup A- Month 7-13 (LLQ-22.7): number analyzed (Participants) | 194 | 191 | 127 | 113 | 132 | 136
  Serogroup A- Month 7-13 (LLQ-22.7) | 256.04 | 214.62 | 217.88 | 446.58 | 343.24 | 436.76
  B M14459- Month 0-2 (LLQ-8.0): number analyzed (Participants) | 196 | 194 | 127 | 113 | 130 | 140
  B M14459- Month 0-2 (LLQ-8.0) | 35.10 | 27.81 | 67.02 | 21.09 | 40.10 | 18.57
  B M14459- Month 2-3 (LLQ-8.0): number analyzed (Participants) | 198 | 193 | 127 | 117 | 129 | 139
  B M14459- Month 2-3 (LLQ-8.0) | 55.45 | 46.06 | 52.36 | 16.53 | 30.88 | 44.90
  B M14459- Month 3-7 (LLQ-8.0): number analyzed (Participants) | 197 | 192 | 129 | 117 | 132 | 140
  B M14459- Month 3-7 (LLQ-8.0) | 228.61 | 196.15 | 117.62 | 206.84 | 84.60 | 325.33
  B M14459- Month 7-13 (LLQ-8.0): number analyzed (Participants) | 197 | 188 | 125 | 115 | 132 | 135
  B M14459- Month 7-13 (LLQ-8.0) | 162.94 | 141.79 | 82.51 | 329.36 | 309.09 | 347.86
  B 96217- Month 0-2 (LLQ-8.6): number analyzed (Participants) | 197 | 190 | 130 | 117 | 130 | 134
  B 96217- Month 0-2 (LLQ-8.6) | 93.52 | 91.00 | 124.70 | 88.27 | 83.08 | 79.10
  B 96217- Month 2-3 (LLQ-8.6): number analyzed (Participants) | 197 | 192 | 130 | 117 | 132 | 134
  B 96217- Month 2-3 (LLQ-8.6) | 85.03 | 80.02 | 95.77 | 58.55 | 52.33 | 74.25
  B 96217- Month 3-7 (LLQ-8.6): number analyzed (Participants) | 199 | 193 | 131 | 116 | 132 | 139
  B 96217- Month 3-7 (LLQ-8.6) | 388.93 | 373.02 | 361.75 | 307.65 | 172.73 | 392.59
  B 96217- Month 7-13 (LLQ-8.6): number analyzed (Participants) | 200 | 191 | 127 | 117 | 132 | 139
  B 96217- Month 7-13 (LLQ-8.6) | 545.92 | 515.49 | 495.00 | 561.47 | 411.36 | 578.42
  B NZ98/254- Month 0-2 (LLQ-8.2): number analyzed (Participants) | 198 | 193 | 129 | 116 | 131 | 139
  B NZ98/254- Month 0-2 (LLQ-8.2) | 30.27 | 25.84 | 48.92 | 22.37 | 31.33 | 20.13
  B NZ98/254- Month 2-3 (LLQ-8.2): number analyzed (Participants) | 198 | 194 | 129 | 117 | 131 | 137
  B NZ98/254- Month 2-3 (LLQ-8.2) | 55.56 | 40.77 | 37.21 | 15.89 | 24.05 | 42.93
  B NZ98/254- Month 3-7 (LLQ-8.2): number analyzed (Participants) | 196 | 194 | 130 | 116 | 132 | 140
  B NZ98/254- Month 3-7 (LLQ-8.2) | 227.81 | 162.89 | 92.78 | 156.65 | 65.46 | 282.91
  B NZ98/254- Month 7-13 (LLQ-8.2): number analyzed (Participants) | 200 | 193 | 129 | 117 | 130 | 138
  B NZ98/254- Month 7-13 (LLQ-8.2) | 142.59 | 105.40 | 90.34 | 242.66 | 257.90 | 277.24
  B M07-0241084- Month 0-2 (LLQ-8.9): number analyzed (Participants) | 196 | 191 | 127 | 117 | 130 | 140
  B M07-0241084- Month 0-2 (LLQ-8.9) | 57.74 | 43.20 | 53.67 | 42.74 | 58.93 | 47.53
  B M07-0241084- Month 2-3 (LLQ-8.9): number analyzed (Participants) | 198 | 189 | 129 | 116 | 128 | 137
  B M07-0241084- Month 2-3 (LLQ-8.9) | 52.46 | 37.16 | 34.01 | 28.33 | 34.47 | 41.65
  B M07-0241084- Month 3-7 (LLQ-8.9): number analyzed (Participants) | 197 | 193 | 129 | 118 | 132 | 137
  B M07-0241084- Month 3-7 (LLQ-8.9) | 213.53 | 151.20 | 111.63 | 190.79 | 110.94 | 251.09
  B M07-0241084- Month 7-13 (LLQ-8.9): number analyzed (Participants) | 198 | 190 | 130 | 116 | 130 | 136
  B M07-0241084- Month 7-13 (LLQ-8.9) | 217.26 | 159.73 | 145.97 | 301.71 | 282.69 | 320.48
  Serogroup C- Month 0-2(LLQ-5.2): number analyzed (Participants) | 198 | 193 | 129 | 118 | 131 | 140
  Serogroup C- Month 0-2(LLQ-5.2) | 102.82 | 129.30 | 148.03 | 126.63 | 135.79 | 128.34
  Serogroup C- Month 2-3(LLQ-5.2): number analyzed (Participants) | 197 | 194 | 129 | 117 | 132 | 136
  Serogroup C- Month 2-3(LLQ-5.2) | 78.78 | 91.97 | 99.22 | 82.97 | 88.21 | 92.85
  Serogroup C- Month 3-7(LLQ-5.2): number analyzed (Participants) | 199 | 196 | 131 | 118 | 131 | 138
  Serogroup C- Month 3-7(LLQ-5.2) | 331.60 | 390.80 | 390.79 | 360.70 | 339.12 | 398.53
  Serogroup C- Month 7-13(LLQ-5.2): number analyzed (Participants) | 196 | 192 | 130 | 116 | 130 | 139
  Serogroup C- Month 7-13(LLQ-5.2) | 382.55 | 567.41 | 574.69 | 589.70 | 545.04 | 595.68
  Serogroup W-Month 0-2(LLQ-39.6): number analyzed (Participants) | 199 | 195 | 130 | 116 | 131 | 138
  Serogroup W-Month 0-2(LLQ-39.6) | 75.66 | 93.12 | 124.89 | 85.71 | 103.94 | 84.23
  Serogroup W-Month 2-3(LLQ-39.6): number analyzed (Participants) | 186 | 190 | 129 | 114 | 131 | 137
  Serogroup W-Month 2-3(LLQ-39.6) | 68.51 | 81.75 | 90.33 | 65.66 | 75.19 | 78.97
  Serogroup W-Month 3-7(LLQ-39.6): number analyzed (Participants) | 195 | 195 | 131 | 118 | 131 | 129
  Serogroup W-Month 3-7(LLQ-39.6) | 293.42 | 359.84 | 327.79 | 331.64 | 297.71 | 392.61
  Serogroup W-Month 7-13(LLQ-39.6): number analyzed (Participants) | 194 | 192 | 130 | 117 | 130 | 139
  Serogroup W-Month 7-13(LLQ-39.6) | 305.31 | 444.54 | 434.34 | 543.61 | 512.92 | 550.19
  Serogroup Y-Month 0-2(LLQ-14.7): number analyzed (Participants) | 199 | 193 | 129 | 115 | 131 | 139
  Serogroup Y-Month 0-2(LLQ-14.7) | 36.25 | 76.31 | 99.44 | 67.83 | 84.92 | 67.58
  Serogroup Y-Month 2-3(LLQ-14.7): number analyzed (Participants) | 197 | 195 | 128 | 116 | 132 | 138
  Serogroup Y-Month 2-3(LLQ-14.7) | 24.51 | 79.32 | 83.26 | 58.88 | 67.70 | 75.50
  Serogroup Y-Month 3-7(LLQ-14.7): number analyzed (Participants) | 199 | 194 | 131 | 118 | 132 | 139
  Serogroup Y-Month 3-7(LLQ-14.7) | 100.05 | 339.26 | 339.26 | 303.62 | 234.85 | 373.95
  Serogroup Y-Month 7-13(LLQ-14.7): number analyzed (Participants) | 199 | 191 | 129 | 117 | 131 | 139
  Serogroup Y-Month 7-13(LLQ-14.7) | 125.13 | 425.13 | 389.69 | 520.64 | 454.48 | 537.41

20. Secondary Outcome: Number of Participants Reporting Any Solicited Local or Systemic AEs and Other Indicators of Reactogenicity Within 30 Minutes After Vaccination.
Description: Number of participants reporting any solicited local or systemic AEs and other indicators of reactogenicity within 30 minutes after each vaccination. Assessed solicited symptoms were Pain, erythema and induration. Assessed solicited systemic symptoms were Fatigue, headache, myalgia, arthralgia, loss of appetite, nausea, chills, and fever (body temperature ≥38.0°C).
Time Frame: Within 30 minutes after vaccination
Population: Analysis was done on subjects in Solicited Safety Set - all screened subjects who provided informed consent & provided demographic &/or other baseline screening measurements, regardless of the subject's randomization & vaccination status in the trial, received a subject ID,provided post-vaccination reactogenicity data & received a study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | rMenB_0_2 Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group | ABCWY_0_2_6 Group
Number analyzed (Participants) | 228 | 232 | 155 | 134 | 151 | 159
Participants
  Any Induration(1st vaccination): number analyzed (Participants) | 217 | 219 | 146 | 128 | 143 | 151
  Any Induration(1st vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Induration(1st vaccination): number analyzed (Participants) | 217 | 219 | 146 | 128 | 143 | 151
  Grade 3 Induration(1st vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Induration(2nd vaccination): number analyzed (Participants) | 215 | 217 | 150 | 125 | 144 | 151
  Any Induration(2nd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Induration(2nd vaccination): number analyzed (Participants) | 215 | 217 | 150 | 125 | 144 | 151
  Grade 3 Induration(2nd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Induration(3rd vaccination): number analyzed (Participants) | 212 | 219 | 146 | 125 | 141 | 151
  Any Induration(3rd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Induration(3rd vaccination): number analyzed (Participants) | 212 | 219 | 146 | 125 | 141 | 151
  Grade 3 Induration(3rd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Induration(4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Any Induration(4th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Induration(4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Grade 3 Induration(4th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Induration(5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 134 | 149
  Any Induration(5th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Induration(5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 134 | 149
  Grade 3 Induration(5th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Erythema(1st vaccination): number analyzed (Participants) | 217 | 219 | 146 | 128 | 143 | 151
  Any Erythema(1st vaccination) | 1 | 0 | 0 | 0 | 1 | 0
  Grade 3 Erythema(1st vaccination): number analyzed (Participants) | 217 | 219 | 146 | 128 | 143 | 151
  Grade 3 Erythema(1st vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Erythema(2nd vaccination): number analyzed (Participants) | 215 | 217 | 150 | 125 | 144 | 151
  Any Erythema(2nd vaccination) | 2 | 0 | 0 | 1 | 0 | 0
  Grade 3 Erythema(2nd vaccination): number analyzed (Participants) | 215 | 217 | 150 | 125 | 144 | 151
  Grade 3 Erythema(2nd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Erythema(3rd vaccination): number analyzed (Participants) | 212 | 219 | 146 | 125 | 141 | 151
  Any Erythema(3rd vaccination) | 0 | 1 | 0 | 1 | 0 | 0
  Grade 3 Erythema(3rd vaccination): number analyzed (Participants) | 212 | 219 | 146 | 125 | 141 | 151
  Grade 3 Erythema(3rd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Erythema(4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Any Erythema(4th vaccination) | 0 | 1 | 0 | 0 | 0 | 1
  Grade 3 Erythema(4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Grade 3 Erythema(4th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Erythema(5th vaccination): number analyzed (Participants) | 206 | 206 | 141 | 122 | 133 | 149
  Any Erythema(5th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Erythema(5th vaccination): number analyzed (Participants) | 206 | 206 | 141 | 122 | 133 | 149
  Grade 3 Erythema(5th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain(1st vaccination): number analyzed (Participants) | 228 | 231 | 155 | 134 | 151 | 159
  Any Pain(1st vaccination) | 19 | 4 | 12 | 8 | 17 | 13
  Grade 3 Pain(1st vaccination): number analyzed (Participants) | 228 | 231 | 155 | 134 | 151 | 159
  Grade 3 Pain(1st vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain(2nd vaccination): number analyzed (Participants) | 216 | 221 | 150 | 129 | 145 | 153
  Any Pain(2nd vaccination) | 10 | 12 | 11 | 9 | 14 | 9
  Grade 3 Pain(2nd vaccination): number analyzed (Participants) | 216 | 221 | 150 | 129 | 145 | 153
  Grade 3 Pain(2nd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain(3rd vaccination): number analyzed (Participants) | 213 | 219 | 146 | 126 | 141 | 152
  Any Pain(3rd vaccination) | 10 | 11 | 8 | 7 | 5 | 13
  Grade 3 Pain(3rd vaccination): number analyzed (Participants) | 213 | 219 | 146 | 126 | 141 | 152
  Grade 3 Pain(3rd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain(4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Any Pain(4th vaccination) | 28 | 22 | 7 | 14 | 8 | 17
  Grade 3 Pain(4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Grade 3 Pain(4th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Pain(5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 133 | 149
  Any Pain(5th vaccination) | 19 | 16 | 12 | 15 | 13 | 12
  Grade 3 Pain(5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 133 | 149
  Grade 3 Pain(5th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Nausea(1st vaccination): number analyzed (Participants) | 228 | 231 | 155 | 134 | 151 | 158
  Any Nausea(1st vaccination) | 0 | 0 | 2 | 1 | 2 | 2
  Grade 3 Nausea(1st vaccination): number analyzed (Participants) | 228 | 231 | 155 | 134 | 151 | 158
  Grade 3 Nausea(1st vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Nausea(2nd vaccination): number analyzed (Participants) | 216 | 221 | 150 | 129 | 145 | 153
  Any Nausea(2nd vaccination) | 2 | 0 | 1 | 1 | 0 | 0
  Grade 3 Nausea(2nd vaccination): number analyzed (Participants) | 216 | 221 | 150 | 129 | 145 | 153
  Grade 3 Nausea(2nd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Nausea(3rd vaccination): number analyzed (Participants) | 213 | 219 | 146 | 126 | 141 | 152
  Any Nausea(3rd vaccination) | 2 | 0 | 2 | 0 | 0 | 1
  Grade 3 Nausea(3rd vaccination): number analyzed (Participants) | 213 | 219 | 146 | 126 | 141 | 152
  Grade 3 Nausea(3rd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Nausea(4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Any Nausea(4th vaccination) | 2 | 0 | 2 | 0 | 1 | 0
  Grade 3 Nausea(4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Grade 3 Nausea(4th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Nausea(5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 134 | 149
  Any Nausea(5th vaccination) | 1 | 0 | 3 | 1 | 0 | 1
  Grade 3 Nausea(5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 134 | 149
  Grade 3 Nausea(5th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Fatigue (1st vaccination): number analyzed (Participants) | 228 | 231 | 155 | 134 | 151 | 158
  Any Fatigue (1st vaccination) | 4 | 6 | 6 | 1 | 2 | 1
  Grade 3 Fatigue(1st vaccination): number analyzed (Participants) | 228 | 231 | 155 | 134 | 151 | 158
  Grade 3 Fatigue(1st vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Fatigue (2nd vaccination): number analyzed (Participants) | 216 | 221 | 150 | 129 | 145 | 153
  Any Fatigue (2nd vaccination) | 4 | 3 | 1 | 1 | 2 | 0
  Grade 3 Fatigue(2nd vaccination): number analyzed (Participants) | 216 | 221 | 150 | 129 | 145 | 153
  Grade 3 Fatigue(2nd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Fatigue (3rd vaccination): number analyzed (Participants) | 213 | 219 | 146 | 126 | 141 | 152
  Any Fatigue (3rd vaccination) | 2 | 4 | 0 | 1 | 1 | 2
  Grade 3 Fatigue(3rd vaccination): number analyzed (Participants) | 213 | 219 | 146 | 126 | 141 | 152
  Grade 3 Fatigue(3rd vaccination) | 0 | 0 | 0 | 1 | 0 | 0
  Any Fatigue (4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Any Fatigue (4th vaccination) | 2 | 1 | 1 | 0 | 1 | 3
  Grade 3 Fatigue(4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Grade 3 Fatigue(4th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Fatigue (5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 134 | 149
  Any Fatigue (5th vaccination) | 1 | 2 | 1 | 3 | 1 | 1
  Grade 3 Fatigue(5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 134 | 149
  Grade 3 Fatigue(5th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Myalgia(1st vaccination): number analyzed (Participants) | 228 | 231 | 155 | 134 | 151 | 158
  Any Myalgia(1st vaccination) | 0 | 1 | 0 | 0 | 0 | 0
  Grade 3 Myalgia(1st vaccination): number analyzed (Participants) | 228 | 231 | 155 | 134 | 151 | 158
  Grade 3 Myalgia(1st vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Myalgia(2nd vaccination): number analyzed (Participants) | 216 | 221 | 150 | 129 | 145 | 153
  Any Myalgia(2nd vaccination) | 0 | 0 | 1 | 0 | 3 | 1
  Grade 3 Myalgia(2nd vaccination): number analyzed (Participants) | 216 | 221 | 150 | 129 | 145 | 153
  Grade 3 Myalgia(2nd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Myalgia(3rd vaccination): number analyzed (Participants) | 213 | 219 | 146 | 126 | 141 | 152
  Any Myalgia(3rd vaccination) | 0 | 0 | 0 | 1 | 0 | 0
  Grade 3 Myalgia(3rd vaccination): number analyzed (Participants) | 213 | 219 | 146 | 126 | 141 | 152
  Grade 3 Myalgia(3rd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Myalgia(4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Any Myalgia(4th vaccination) | 0 | 0 | 0 | 0 | 1 | 0
  Grade 3 Myalgia(4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Grade 3 Myalgia(4th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Myalgia(5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 134 | 149
  Any Myalgia(5th vaccination) | 0 | 4 | 1 | 0 | 1 | 0
  Grade 3 Myalgia(5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 134 | 149
  Grade 3 Myalgia(5th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Arthralgia(1st vaccination): number analyzed (Participants) | 228 | 231 | 155 | 134 | 151 | 158
  Any Arthralgia(1st vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Arthralgia(1st vaccination): number analyzed (Participants) | 228 | 231 | 155 | 134 | 151 | 158
  Grade 3 Arthralgia(1st vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Arthralgia(2nd vaccination): number analyzed (Participants) | 216 | 221 | 150 | 129 | 145 | 153
  Any Arthralgia(2nd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Arthralgia(2nd vaccination): number analyzed (Participants) | 216 | 221 | 150 | 129 | 145 | 153
  Grade 3 Arthralgia(2nd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Arthralgia(3rd vaccination): number analyzed (Participants) | 213 | 219 | 146 | 126 | 141 | 152
  Any Arthralgia(3rd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Arthralgia(3rd vaccination): number analyzed (Participants) | 213 | 219 | 146 | 126 | 141 | 152
  Grade 3 Arthralgia(3rd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Arthralgia(4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Any Arthralgia(4th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Arthralgia(4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Grade 3 Arthralgia(4th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Arthralgia(5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 134 | 149
  Any Arthralgia(5th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Arthralgia(5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 134 | 149
  Grade 3 Arthralgia(5th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Headache(1st vaccination): number analyzed (Participants) | 228 | 231 | 155 | 134 | 151 | 158
  Any Headache(1st vaccination) | 2 | 3 | 1 | 1 | 1 | 0
  Grade 3 Headache(1st vaccination): number analyzed (Participants) | 228 | 231 | 155 | 134 | 151 | 158
  Grade 3 Headache(1st vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Headache(2nd vaccination): number analyzed (Participants) | 216 | 221 | 150 | 129 | 145 | 153
  Any Headache(2nd vaccination) | 3 | 1 | 2 | 1 | 1 | 1
  Grade 3 Headache(2nd vaccination): number analyzed (Participants) | 216 | 221 | 150 | 129 | 145 | 153
  Grade 3 Headache(2nd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Headache(3rd vaccination): number analyzed (Participants) | 213 | 219 | 146 | 126 | 141 | 152
  Any Headache(3rd vaccination) | 2 | 1 | 2 | 0 | 1 | 1
  Grade 3 Headache(3rd vaccination): number analyzed (Participants) | 213 | 219 | 146 | 126 | 141 | 152
  Grade 3 Headache(3rd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Headache(4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Any Headache(4th vaccination) | 3 | 2 | 0 | 0 | 1 | 1
  Grade 3 Headache(4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Grade 3 Headache(4th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Headache(5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 134 | 149
  Any Headache(5th vaccination) | 2 | 1 | 0 | 0 | 0 | 1
  Grade 3 Headache(5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 134 | 149
  Grade 3 Headache(5th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Chills(1st vaccination): number analyzed (Participants) | 228 | 231 | 155 | 134 | 151 | 158
  Any Chills(1st vaccination) | 0 | 1 | 1 | 0 | 2 | 2
  Grade 3 Chills(1st vaccination): number analyzed (Participants) | 228 | 231 | 155 | 134 | 151 | 158
  Grade 3 Chills(1st vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Chills(2nd vaccination): number analyzed (Participants) | 216 | 221 | 150 | 129 | 145 | 153
  Any Chills(2nd vaccination) | 1 | 1 | 1 | 1 | 0 | 0
  Gradec3 Chills(2nd vaccination): number analyzed (Participants) | 216 | 221 | 150 | 129 | 145 | 153
  Gradec3 Chills(2nd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Chills(3rd vaccination): number analyzed (Participants) | 213 | 219 | 146 | 126 | 141 | 152
  Any Chills(3rd vaccination) | 1 | 1 | 0 | 0 | 0 | 0
  Grade 3 Chills(3rd vaccination): number analyzed (Participants) | 213 | 219 | 146 | 126 | 141 | 152
  Grade 3 Chills(3rd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Chills(4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Any Chills(4th vaccination) | 1 | 1 | 0 | 0 | 0 | 0
  Grade 3 Chills(4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Grade 3 Chills(4th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Chills(5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 134 | 149
  Any Chills(5th vaccination) | 1 | 1 | 0 | 0 | 0 | 0
  Grade 3 Chills(5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 134 | 149
  Grade 3 Chills(5th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Appetite Loss(1st vaccination): number analyzed (Participants) | 228 | 231 | 155 | 134 | 151 | 158
  Any Appetite Loss(1st vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Appetite Loss(1st vaccination): number analyzed (Participants) | 228 | 231 | 155 | 134 | 151 | 158
  Grade 3 Appetite Loss(1st vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Appetite Loss(2nd vaccination): number analyzed (Participants) | 216 | 221 | 150 | 129 | 145 | 153
  Any Appetite Loss(2nd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Appetite Loss(2nd vaccination): number analyzed (Participants) | 216 | 221 | 150 | 129 | 145 | 153
  Grade 3 Appetite Loss(2nd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Appetite Loss(3rd vaccination): number analyzed (Participants) | 213 | 219 | 146 | 126 | 141 | 152
  Any Appetite Loss(3rd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Appetite Loss(3rd vaccination): number analyzed (Participants) | 213 | 219 | 146 | 126 | 141 | 152
  Grade 3 Appetite Loss(3rd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Any Appetite Loss(4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Any Appetite Loss(4th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Appetite Loss(4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Grade 3 Appetite Loss(4th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  AnyAppetiteLoss(5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 134 | 149
  AnyAppetiteLoss(5th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Grade 3 Appetite Loss(5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 134 | 149
  Grade 3 Appetite Loss(5th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Fever(1st vaccination): number analyzed (Participants) | 228 | 232 | 155 | 133 | 151 | 158
  Fever(1st vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Fever(2nd vaccination): number analyzed (Participants) | 216 | 221 | 150 | 128 | 145 | 153
  Fever(2nd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Fever(3rd vaccination): number analyzed (Participants) | 213 | 218 | 146 | 125 | 141 | 152
  Fever(3rd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Fever(4th vaccination): number analyzed (Participants) | 211 | 214 | 140 | 124 | 137 | 152
  Fever(4th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Fever(5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 134 | 149
  Fever(5th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Fever prevention(1st vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Fever prevention(2nd vaccination): number analyzed (Participants) | 216 | 221 | 150 | 129 | 145 | 153
  Pain/Fever prevention(2nd vaccination) | 0 | 2 | 0 | 0 | 0 | 0
  Pain/Fever prevention(3rd vaccination): number analyzed (Participants) | 213 | 219 | 146 | 126 | 141 | 152
  Pain/Fever prevention(3rd vaccination) | 1 | 0 | 0 | 0 | 0 | 0
  Pain/Fever prevention(4th vaccination): number analyzed (Participants) | 211 | 214 | 141 | 124 | 138 | 152
  Pain/Fever prevention(4th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Fever prevention(5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 134 | 149
  Pain/Fever prevention(5th vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Fever treatment(1st vaccination): number analyzed (Participants) | 227 | 232 | 155 | 134 | 151 | 159
  Pain/Fever treatment(1st vaccination) | 0 | 0 | 1 | 0 | 0 | 0
  Pain/Fever treatment(2nd vaccination): number analyzed (Participants) | 216 | 221 | 150 | 129 | 145 | 153
  Pain/Fever treatment(2nd vaccination) | 1 | 0 | 0 | 0 | 0 | 1
  Pain/Fever treatment(3rd vaccination): number analyzed (Participants) | 213 | 219 | 146 | 126 | 141 | 152
  Pain/Fever treatment(3rd vaccination) | 0 | 0 | 0 | 0 | 0 | 0
  Pain/Fever treatment(4th vaccination): number analyzed (Participants) | 212 | 214 | 141 | 124 | 138 | 152
  Pain/Fever treatment(4th vaccination) | 0 | 1 | 0 | 0 | 0 | 0
  Pain/Fever treatment(5th vaccination): number analyzed (Participants) | 207 | 206 | 141 | 122 | 134 | 149
  Pain/Fever treatment(5th vaccination) | 0 | 0 | 0 | 0 | 1 | 0

21. Secondary Outcome: Number of Participants Reporting Any Unsolicited AEs Within 30 Minutes After Vaccination.
Description: An unsolicited adverse event is an adverse event that was not solicited and that was spontaneously communicated by a participant and/or parent/legal guardian who has signed the informed consent. Number of participants reporting any unsolicited AE within 30 minutes after each vaccination.
Time Frame: Within 30 minutes after vaccination
Population: Analysis was done on subjects in the Unsolicited Safety Set-all screened subjects who provided informed consent & demographic &/or other baseline screening measurements, regardless of the subject's randomization & vaccination status, received a subject ID, received a study vaccination & have either post-vaccination reactogenicity data or records.
Measure: Count of Participants; unit: Participants
Arm/Group | rMenB_0_2 Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group | ABCWY_0_2_6 Group
Number analyzed (Participants) | 221 | 228 | 151 | 129 | 147 | 157
Participants
  Dizziness | 3 | 0 | 1 | 2 | 0 | 1
  Presyncope | 2 | 1 | 0 | 0 | 0 | 0
  Syncope | 0 | 1 | 1 | 0 | 1 | 0
  Injection site pain | 1 | 0 | 0 | 0 | 0 | 1
  Asthenia | 0 | 0 | 0 | 0 | 0 | 1
  Dyspnoea | 1 | 0 | 0 | 0 | 0 | 0
  Fatigue | 0 | 0 | 0 | 0 | 1 | 0
  Headache | 0 | 0 | 0 | 0 | 1 | 0
  Hypoaesthesia | 0 | 0 | 0 | 0 | 1 | 0
  Injection site bruising | 1 | 0 | 0 | 0 | 0 | 0
  Injection site warmth | 0 | 1 | 0 | 0 | 0 | 0
  Pain | 0 | 0 | 0 | 0 | 1 | 0
  Paraesthesia | 1 | 0 | 0 | 0 | 0 | 0
  Pruritus allergic | 0 | 0 | 1 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants Reporting Unsolicited AEs From Day 1 to Day 30 After Any Vaccination.
Description: The number of participants reporting unsolicited AEs and possibly or probably related unsolicited AEs were assessed.
Time Frame: Day 1 through Day 30 after any vaccination
Population: Analysis was done on subjects in the Unsolicited Safety Set -all screened subjects who provided informed consent & provided demographic &/or other baseline screening measurements, regardless of the subject's randomization & vaccination status, received a subject ID, received a study vaccination & have either post-vaccination reactogenicity records.
Measure: Count of Participants; unit: Participants
Arm/Group | rMenB_0_2 Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group | ABCWY_0_2_6 Group
Number analyzed (Participants) | 221 | 228 | 151 | 129 | 147 | 157
Participants
  Any AE(s) | 146 | 148 | 93 | 76 | 97 | 104
  Possibly or Probably Related AE(s) | 25 | 31 | 23 | 16 | 18 | 27

23. Secondary Outcome: Number of Participants Reporting Any Solicited Local or Systemic Adverse Events (AEs) and Other Indicators of Reactogenicity From Day 1 to Day 7.
Description: Number of participants reporting any solicited local or systemic AEs and other indicators of reactogenicity from Day 1 (6 hours) to Day 7 after any meningococcal vaccination is reported.
Time Frame: At Day 1 (6 hours) to Day 7 after vaccination
Population: Analysis was done on all subjects in the Solicited Safety Set-all screened subjects who provided informed consent & provided demographic &/ other baseline screening measurements,regardless of the subject's randomization & vaccination status in the trial,received a subject ID,provided post-vaccination reactogenicity data & received study vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | rMenB_0_2 Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group | ABCWY_0_2_6 Group
Number analyzed (Participants) | 228 | 231 | 155 | 134 | 151 | 159
Participants
  Any AE | 225 | 228 | 153 | 131 | 151 | 157
  Any Local AE | 224 | 227 | 148 | 129 | 148 | 156
  Any Systemic AE | 201 | 201 | 143 | 117 | 134 | 143
  Any Pain (1st vacc): number analyzed (Participants) | 227 | 231 | 154 | 134 | 151 | 159
  Any Pain (1st vacc) | 213 | 223 | 142 | 126 | 80 | 146
  Grade 3 Pain (1st vacc): number analyzed (Participants) | 227 | 231 | 154 | 134 | 151 | 159
  Grade 3 Pain (1st vacc) | 9 | 13 | 2 | 10 | 0 | 6
  Any Pain (2nd vacc): number analyzed (Participants) | 214 | 216 | 150 | 128 | 144 | 151
  Any Pain (2nd vacc) | 32 | 34 | 122 | 41 | 135 | 51
  Grade 3 Pain (2nd vacc): number analyzed (Participants) | 214 | 216 | 150 | 128 | 144 | 151
  Grade 3 Pain (2nd vacc) | 0 | 1 | 5 | 0 | 11 | 0
  Any Pain (3rd vacc): number analyzed (Participants) | 212 | 217 | 144 | 125 | 138 | 150
  Any Pain (3rd vacc) | 193 | 185 | 38 | 26 | 16 | 133
  Grade 3 Pain (3rd vacc): number analyzed (Participants) | 212 | 217 | 144 | 125 | 138 | 150
  Grade 3 Pain (3rd vacc) | 11 | 7 | 0 | 0 | 0 | 5
  Any Pain (4th vacc): number analyzed (Participants) | 206 | 211 | 139 | 120 | 136 | 152
  Any Pain (4th vacc) | 79 | 77 | 19 | 106 | 44 | 138
  Grade 3 Pain (4th vacc): number analyzed (Participants) | 206 | 211 | 139 | 120 | 136 | 152
  Grade 3 Pain (4th vacc) | 1 | 0 | 0 | 10 | 0 | 9
  Any Pain (5th vacc): number analyzed (Participants) | 206 | 206 | 140 | 121 | 132 | 147
  Any Pain (5th vacc) | 83 | 80 | 58 | 48 | 119 | 64
  Grade 3 Pain (5th vacc): number analyzed (Participants) | 206 | 206 | 140 | 121 | 132 | 147
  Grade 3 Pain (5th vacc) | 0 | 1 | 1 | 0 | 11 | 1
  Any Erythema (1st vacc): number analyzed (Participants) | 226 | 231 | 154 | 133 | 150 | 159
  Any Erythema (1st vacc) | 23 | 21 | 16 | 11 | 1 | 23
  Grade 3 Erythema (1st vacc): number analyzed (Participants) | 226 | 231 | 154 | 133 | 150 | 159
  Grade 3 Erythema (1st vacc) | 0 | 1 | 1 | 0 | 0 | 2
  Any Erythema (2nd vacc): number analyzed (Participants) | 213 | 215 | 150 | 128 | 144 | 121
  Any Erythema (2nd vacc) | 3 | 5 | 8 | 1 | 17 | 2
  Grade3Erythema(2ndvacc): number analyzed (Participants) | 213 | 215 | 150 | 128 | 144 | 121
  Grade3Erythema(2ndvacc) | 0 | 0 | 1 | 0 | 3 | 0
  Any Erythema (3rd vacc): number analyzed (Participants) | 211 | 216 | 144 | 121 | 136 | 150
  Any Erythema (3rd vacc) | 32 | 27 | 0 | 2 | 0 | 19
  Grade3Erythema(3rdvacc): number analyzed (Participants) | 211 | 216 | 144 | 121 | 136 | 150
  Grade3Erythema(3rdvacc) | 2 | 6 | 0 | 0 | 0 | 1
  Any Erythema (4th vacc): number analyzed (Participants) | 202 | 209 | 137 | 119 | 133 | 151
  Any Erythema (4th vacc) | 1 | 1 | 0 | 10 | 0 | 13
  Grade3Erythema(4thvacc): number analyzed (Participants) | 202 | 209 | 137 | 119 | 133 | 151
  Grade3Erythema(4thvacc) | 0 | 0 | 0 | 1 | 0 | 4
  Any Erythema (5th vacc): number analyzed (Participants) | 203 | 203 | 139 | 119 | 129 | 146
  Any Erythema (5th vacc) | 1 | 1 | 1 | 0 | 11 | 0
  Grade3Erythema(5thvacc): number analyzed (Participants) | 203 | 203 | 139 | 119 | 129 | 146
  Grade3Erythema(5thvacc) | 0 | 0 | 0 | 0 | 1 | 0
  AnyInduration(1st vacc): number analyzed (Participants) | 226 | 231 | 154 | 133 | 150 | 159
  AnyInduration(1st vacc) | 21 | 20 | 12 | 13 | 3 | 19
  Grade3Induration(1vacc): number analyzed (Participants) | 226 | 231 | 154 | 133 | 150 | 159
  Grade3Induration(1vacc) | 0 | 0 | 0 | 1 | 0 | 1
  AnyInduration(2nd vacc): number analyzed (Participants) | 213 | 215 | 150 | 128 | 144 | 151
  AnyInduration(2nd vacc) | 2 | 2 | 10 | 0 | 11 | 2
  Grade3Induration(2vacc): number analyzed (Participants) | 213 | 215 | 150 | 128 | 144 | 151
  Grade3Induration(2vacc) | 0 | 0 | 0 | 0 | 0 | 0
  AnyInduration(3rd vacc): number analyzed (Participants) | 211 | 216 | 144 | 121 | 136 | 150
  AnyInduration(3rd vacc) | 24 | 17 | 0 | 0 | 1 | 20
  Grade3Induration(3vacc): number analyzed (Participants) | 211 | 216 | 144 | 121 | 136 | 150
  Grade3Induration(3vacc) | 2 | 0 | 0 | 0 | 0 | 0
  AnyInduration(4th vacc): number analyzed (Participants) | 202 | 209 | 137 | 119 | 133 | 151
  AnyInduration(4th vacc) | 2 | 3 | 0 | 10 | 0 | 14
  Grade3Induration(4vacc): number analyzed (Participants) | 202 | 209 | 137 | 119 | 133 | 151
  Grade3Induration(4vacc) | 0 | 0 | 0 | 1 | 0 | 1
  AnyInduration(5th vacc): number analyzed (Participants) | 203 | 203 | 139 | 119 | 129 | 146
  AnyInduration(5th vacc) | 2 | 3 | 1 | 2 | 16 | 1
  Grade 3 Induration(5th vacc): number analyzed (Participants) | 203 | 203 | 139 | 119 | 129 | 146
  Grade 3 Induration(5th vacc) | 0 | 0 | 0 | 1 | 1 | 0
  Any Fatigue (1st vacc): number analyzed (Participants) | 227 | 231 | 154 | 134 | 151 | 159
  Any Fatigue (1st vacc) | 126 | 121 | 84 | 68 | 68 | 76
  Grade 3 Fatigue(1st vacc): number analyzed (Participants) | 227 | 231 | 154 | 134 | 151 | 159
  Grade 3 Fatigue(1st vacc) | 7 | 7 | 4 | 3 | 3 | 4
  Any Fatigue (2nd vacc): number analyzed (Participants) | 214 | 216 | 150 | 128 | 144 | 151
  Any Fatigue (2nd vacc) | 61 | 64 | 64 | 40 | 64 | 49
  Grade 3 Fatigue(2nd vacc): number analyzed (Participants) | 214 | 216 | 150 | 128 | 144 | 151
  Grade 3 Fatigue(2nd vacc) | 0 | 3 | 4 | 2 | 1 | 0
  Any Fatigue (3rd vacc): number analyzed (Participants) | 212 | 217 | 144 | 125 | 138 | 150
  Any Fatigue (3rd vacc) | 106 | 96 | 44 | 32 | 32 | 55
  Garde 3 Fatigue(3rd vacc): number analyzed (Participants) | 212 | 217 | 144 | 125 | 138 | 150
  Garde 3 Fatigue(3rd vacc) | 4 | 5 | 1 | 0 | 1 | 1
  Any Fatigue (4th vacc): number analyzed (Participants) | 206 | 211 | 139 | 120 | 136 | 152
  Any Fatigue (4th vacc) | 50 | 56 | 37 | 51 | 35 | 73
  Grade 3 Fatigue(4th vacc): number analyzed (Participants) | 206 | 211 | 139 | 120 | 136 | 152
  Grade 3 Fatigue(4th vacc) | 2 | 3 | 0 | 5 | 2 | 3
  Any Fatigue (5th vacc): number analyzed (Participants) | 206 | 206 | 140 | 121 | 132 | 147
  Any Fatigue (5th vacc) | 62 | 59 | 37 | 41 | 51 | 46
  Grade3Fatigue(5th vacc): number analyzed (Participants) | 206 | 206 | 140 | 121 | 132 | 147
  Grade3Fatigue(5th vacc) | 1 | 2 | 4 | 0 | 6 | 3
  Any Headache (1st vacc): number analyzed (Participants) | 227 | 231 | 154 | 134 | 151 | 159
  Any Headache (1st vacc) | 103 | 92 | 65 | 52 | 63 | 64
  Grade3Headache(1stvacc): number analyzed (Participants) | 227 | 231 | 154 | 134 | 151 | 159
  Grade3Headache(1stvacc) | 4 | 3 | 5 | 2 | 2 | 3
  Any Headache (2nd vacc): number analyzed (Participants) | 214 | 216 | 150 | 128 | 144 | 151
  Any Headache (2nd vacc) | 67 | 47 | 70 | 36 | 63 | 41
  Grade3Headache(2ndvacc): number analyzed (Participants) | 214 | 216 | 150 | 128 | 144 | 151
  Grade3Headache(2ndvacc) | 1 | 2 | 3 | 2 | 4 | 2
  Any Headache (3rd vacc): number analyzed (Participants) | 212 | 217 | 144 | 125 | 138 | 150
  Any Headache (3rd vacc) | 90 | 76 | 42 | 28 | 30 | 53
  Grade3Headache(3rdvacc): number analyzed (Participants) | 212 | 217 | 144 | 125 | 138 | 150
  Grade3Headache(3rdvacc) | 3 | 4 | 1 | 0 | 3 | 0
  Any Headache (4th vacc): number analyzed (Participants) | 206 | 211 | 139 | 120 | 136 | 152
  Any Headache (4th vacc) | 49 | 35 | 26 | 44 | 26 | 52
  Grade3Headache(4thvacc): number analyzed (Participants) | 206 | 211 | 139 | 120 | 136 | 152
  Grade3Headache(4thvacc) | 3 | 3 | 0 | 2 | 0 | 4
  Any Headache (5th vacc): number analyzed (Participants) | 206 | 206 | 140 | 121 | 132 | 147
  Any Headache (5th vacc) | 64 | 40 | 33 | 33 | 52 | 37
  Grade3Headache(5thvacc): number analyzed (Participants) | 206 | 206 | 140 | 121 | 132 | 147
  Grade3Headache(5thvacc) | 1 | 1 | 2 | 1 | 2 | 2
  Any Myalgia (1st vacc): number analyzed (Participants) | 227 | 231 | 154 | 134 | 151 | 159
  Any Myalgia (1st vacc) | 62 | 53 | 39 | 34 | 33 | 40
  Grade3Myalgia(1st vacc): number analyzed (Participants) | 227 | 231 | 154 | 134 | 151 | 159
  Grade3Myalgia(1st vacc) | 2 | 4 | 2 | 2 | 0 | 3
  Any Myalgia (2nd vacc): number analyzed (Participants) | 214 | 216 | 150 | 128 | 144 | 151
  Any Myalgia (2nd vacc) | 15 | 20 | 27 | 15 | 37 | 18
  Grade3Myalgia(2nd vacc): number analyzed (Participants) | 214 | 216 | 150 | 128 | 144 | 151
  Grade3Myalgia(2nd vacc) | 0 | 3 | 1 | 1 | 1 | 0
  Any Myalgia (3rd vacc): number analyzed (Participants) | 212 | 217 | 144 | 125 | 138 | 150
  Any Myalgia (3rd vacc) | 52 | 40 | 13 | 10 | 13 | 34
  Grade3Myalgia(3rd vacc): number analyzed (Participants) | 212 | 217 | 144 | 125 | 138 | 150
  Grade3Myalgia(3rd vacc) | 2 | 2 | 0 | 0 | 2 | 2
  Any Myalgia (4th vacc): number analyzed (Participants) | 206 | 211 | 139 | 120 | 136 | 152
  Any Myalgia (4th vacc) | 17 | 20 | 11 | 26 | 13 | 39
  Grade3Myalgia(4th vacc): number analyzed (Participants) | 206 | 211 | 139 | 120 | 136 | 152
  Grade3Myalgia(4th vacc) | 1 | 1 | 1 | 2 | 0 | 2
  Any Myalgia (5th vacc): number analyzed (Participants) | 206 | 206 | 140 | 121 | 132 | 147
  Any Myalgia (5th vacc) | 16 | 26 | 19 | 12 | 21 | 19
  Grade3Myalgia(5th vacc): number analyzed (Participants) | 206 | 206 | 140 | 121 | 132 | 147
  Grade3Myalgia(5th vacc) | 0 | 1 | 0 | 0 | 1 | 1
  AnyAppetite Loss(1vacc): number analyzed (Participants) | 227 | 231 | 154 | 134 | 151 | 159
  AnyAppetite Loss(1vacc) | 41 | 33 | 28 | 22 | 14 | 18
  Grade3AppetiteLoss(1vacc): number analyzed (Participants) | 227 | 231 | 154 | 134 | 151 | 159
  Grade3AppetiteLoss(1vacc) | 2 | 3 | 0 | 0 | 0 | 0
  AnyAppetiteLoss(2vacc): number analyzed (Participants) | 214 | 216 | 150 | 128 | 144 | 151
  AnyAppetiteLoss(2vacc) | 17 | 11 | 15 | 12 | 19 | 9
  Grade3AppetiteLoss(2vacc): number analyzed (Participants) | 214 | 216 | 150 | 128 | 144 | 151
  Grade3AppetiteLoss(2vacc) | 0 | 1 | 0 | 0 | 2 | 0
  AnyAppetiteLoss(3vacc): number analyzed (Participants) | 212 | 217 | 144 | 125 | 138 | 150
  AnyAppetiteLoss(3vacc) | 28 | 28 | 7 | 7 | 11 | 17
  Grade3AppetiteLoss(3vacc): number analyzed (Participants) | 212 | 217 | 144 | 125 | 138 | 150
  Grade3AppetiteLoss(3vacc) | 1 | 0 | 1 | 0 | 1 | 0
  AnyAppetiteLoss(4vacc): number analyzed (Participants) | 206 | 211 | 139 | 120 | 136 | 152
  AnyAppetiteLoss(4vacc) | 11 | 10 | 4 | 13 | 11 | 23
  Grade3AppetiteLoss(4vacc): number analyzed (Participants) | 206 | 211 | 139 | 120 | 136 | 152
  Grade3AppetiteLoss(4vacc) | 0 | 0 | 0 | 0 | 0 | 0
  AnyAppetiteLoss(5vacc): number analyzed (Participants) | 206 | 206 | 140 | 121 | 132 | 147
  AnyAppetiteLoss(5vacc) | 18 | 14 | 9 | 9 | 22 | 7
  Grade3AppetiteLoss(5vacc): number analyzed (Participants) | 206 | 206 | 140 | 121 | 132 | 147
  Grade3AppetiteLoss(5vacc) | 0 | 0 | 1 | 0 | 0 | 0
  Any Nausea (1st vacc): number analyzed (Participants) | 227 | 221 | 154 | 134 | 151 | 159
  Any Nausea (1st vacc) | 42 | 36 | 28 | 17 | 26 | 21
  Grade 3 Nausea(1stvacc): number analyzed (Participants) | 227 | 221 | 154 | 134 | 151 | 159
  Grade 3 Nausea(1stvacc) | 1 | 0 | 0 | 0 | 0 | 1
  Any Nausea (2nd vacc): number analyzed (Participants) | 214 | 216 | 150 | 128 | 144 | 151
  Any Nausea (2nd vacc) | 17 | 15 | 20 | 10 | 26 | 15
  Grade 3 Nausea(2nd vacc): number analyzed (Participants) | 214 | 216 | 150 | 128 | 144 | 151
  Grade 3 Nausea(2nd vacc) | 0 | 0 | 0 | 0 | 0 | 0
  Any Nausea (3rd vacc): number analyzed (Participants) | 212 | 217 | 144 | 125 | 138 | 150
  Any Nausea (3rd vacc) | 35 | 24 | 10 | 8 | 4 | 21
  Grade 3 Nausea(3rd vacc): number analyzed (Participants) | 212 | 217 | 144 | 125 | 138 | 150
  Grade 3 Nausea(3rd vacc) | 0 | 0 | 0 | 0 | 0 | 0
  Any Nausea (4th vacc): number analyzed (Participants) | 206 | 211 | 139 | 120 | 136 | 152
  Any Nausea (4th vacc) | 21 | 13 | 9 | 11 | 14 | 23
  Grade 3 Nausea(4th vacc): number analyzed (Participants) | 206 | 211 | 139 | 120 | 136 | 152
  Grade 3 Nausea(4th vacc) | 1 | 0 | 0 | 0 | 0 | 0
  Any Nausea (5th vacc): number analyzed (Participants) | 206 | 206 | 140 | 121 | 132 | 147
  Any Nausea (5th vacc) | 16 | 15 | 8 | 11 | 21 | 12
  Grade 3 Nausea(5th vacc): number analyzed (Participants) | 206 | 206 | 140 | 121 | 132 | 147
  Grade 3 Nausea(5th vacc) | 0 | 0 | 0 | 0 | 0 | 0
  Any Chills (1st vacc): number analyzed (Participants) | 226 | 231 | 154 | 133 | 150 | 159
  Any Chills (1st vacc) | 45 | 36 | 41 | 24 | 27 | 40
  Grade 3 Chills(1stvacc): number analyzed (Participants) | 226 | 231 | 154 | 133 | 150 | 159
  Grade 3 Chills(1stvacc) | 1 | 0 | 1 | 1 | 2 | 1
  Any Chills (2nd vacc): number analyzed (Participants) | 213 | 215 | 150 | 128 | 144 | 151
  Any Chills (2nd vacc) | 17 | 26 | 26 | 12 | 32 | 15
  Grade 3 Chills(2ndvacc): number analyzed (Participants) | 213 | 215 | 150 | 128 | 144 | 151
  Grade 3 Chills(2ndvacc) | 0 | 1 | 1 | 0 | 0 | 0
  Any Chills(3rd vacc): number analyzed (Participants) | 212 | 217 | 144 | 125 | 138 | 150
  Any Chills(3rd vacc) | 33 | 33 | 9 | 7 | 12 | 22
  Grade 3 Chills(3rdvacc): number analyzed (Participants) | 212 | 217 | 144 | 125 | 138 | 150
  Grade 3 Chills(3rdvacc) | 1 | 1 | 0 | 0 | 1 | 0
  Any Chills(4thvacc): number analyzed (Participants) | 206 | 211 | 139 | 120 | 136 | 152
  Any Chills(4thvacc) | 11 | 11 | 10 | 12 | 9 | 31
  Grade 3 Chills(4thvacc): number analyzed (Participants) | 206 | 211 | 139 | 120 | 136 | 152
  Grade 3 Chills(4thvacc) | 2 | 0 | 0 | 0 | 0 | 1
  Any Chills (5th vacc): number analyzed (Participants) | 212 | 217 | 144 | 125 | 138 | 150
  Any Chills (5th vacc) | 19 | 23 | 17 | 11 | 22 | 13
  Grade 3 Chills(5vacc): number analyzed (Participants) | 212 | 217 | 144 | 125 | 138 | 150
  Grade 3 Chills(5vacc) | 0 | 0 | 0 | 1 | 0 | 0
  Fever (1st vacc): number analyzed (Participants) | 227 | 231 | 154 | 133 | 151 | 158
  Fever (1st vacc) | 5 | 4 | 5 | 1 | 2 | 3
  Fever (2nd vacc): number analyzed (Participants) | 214 | 216 | 149 | 127 | 144 | 151
  Fever (2nd vacc) | 2 | 6 | 4 | 2 | 9 | 3
  Fever (3rd vacc): number analyzed (Participants) | 212 | 217 | 143 | 124 | 138 | 150
  Fever (3rd vacc) | 6 | 3 | 2 | 0 | 4 | 4
  Fever (4th vacc): number analyzed (Participants) | 206 | 211 | 138 | 119 | 136 | 151
  Fever (4th vacc) | 0 | 2 | 0 | 3 | 0 | 7
  Fever (5th vacc): number analyzed (Participants) | 206 | 206 | 139 | 120 | 132 | 147
  Fever (5th vacc) | 5 | 1 | 2 | 0 | 3 | 1
  Pain/Fever prevention(1): number analyzed (Participants) | 227 | 231 | 154 | 134 | 151 | 159
  Pain/Fever prevention(1) | 28 | 34 | 21 | 26 | 5 | 34
  Pain/Fever prevention(2): number analyzed (Participants) | 214 | 216 | 150 | 128 | 144 | 151
  Pain/Fever prevention(2) | 5 | 7 | 18 | 5 | 24 | 7
  Pain/Fever prevention(3): number analyzed (Participants) | 212 | 217 | 144 | 125 | 138 | 150
  Pain/Fever prevention(3) | 32 | 34 | 3 | 2 | 3 | 21
  Pain/Fever prevention(4) | 6 | 5 | 3 | 19 | 3 | 25
  Pain/Fever prevention(5): number analyzed (Participants) | 206 | 206 | 140 | 121 | 132 | 147
  Pain/Fever prevention(5) | 5 | 9 | 4 | 1 | 26 | 3
  Pain/Fever treatment(1): number analyzed (Participants) | 227 | 231 | 154 | 134 | 151 | 159
  Pain/Fever treatment(1) | 31 | 45 | 27 | 32 | 6 | 31
  Pain/Fever treatment(2): number analyzed (Participants) | 214 | 216 | 150 | 128 | 144 | 151
  Pain/Fever treatment(2) | 3 | 4 | 20 | 3 | 29 | 4
  Pain/Fever treatment(3): number analyzed (Participants) | 212 | 217 | 144 | 125 | 138 | 150
  Pain/Fever treatment(3) | 38 | 37 | 2 | 4 | 2 | 23
  Pain/Fever treatment(4): number analyzed (Participants) | 206 | 211 | 139 | 120 | 136 | 152
  Pain/Fever treatment(4) | 7 | 4 | 2 | 22 | 2 | 27
  Pain/Fever treatment(5): number analyzed (Participants) | 206 | 206 | 140 | 121 | 132 | 147
  Pain/Fever treatment(5) | 3 | 8 | 2 | 3 | 29 | 2
  Any Arthralgia(1st vacc): number analyzed (Participants) | 227 | 231 | 154 | 134 | 151 | 159
  Any Arthralgia(1st vacc) | 25 | 14 | 13 | 17 | 12 | 14
  Grade3Arthralgia(1stvacc): number analyzed (Participants) | 227 | 231 | 154 | 134 | 151 | 159
  Grade3Arthralgia(1stvacc) | 0 | 1 | 0 | 0 | 1 | 2
  Any Arthralgia (2nd vacc): number analyzed (Participants) | 214 | 216 | 150 | 128 | 144 | 151
  Any Arthralgia (2nd vacc) | 7 | 11 | 10 | 9 | 8 | 7
  Grade3Arthralgia(2ndvacc): number analyzed (Participants) | 214 | 216 | 150 | 128 | 144 | 151
  Grade3Arthralgia(2ndvacc) | 0 | 0 | 0 | 1 | 0 | 1
  Any Arthralgia(3rd vacc): number analyzed (Participants) | 212 | 217 | 144 | 125 | 138 | 150
  Any Arthralgia(3rd vacc) | 16 | 7 | 4 | 3 | 6 | 11
  Grade3Arthralgia(3rdvacc): number analyzed (Participants) | 212 | 217 | 144 | 125 | 138 | 150
  Grade3Arthralgia(3rdvacc) | 0 | 1 | 0 | 0 | 0 | 0
  Any Arthralgia(4th vacc): number analyzed (Participants) | 206 | 211 | 139 | 120 | 136 | 152
  Any Arthralgia(4th vacc) | 8 | 10 | 5 | 10 | 7 | 18
  Grade3Arthralgia(4thvacc): number analyzed (Participants) | 206 | 211 | 139 | 120 | 136 | 152
  Grade3Arthralgia(4thvacc) | 1 | 0 | 0 | 0 | 0 | 2
  Any Arthralgia(5th vacc): number analyzed (Participants) | 206 | 206 | 140 | 121 | 132 | 147
  Any Arthralgia(5th vacc) | 8 | 9 | 8 | 6 | 11 | 11
  Grade3Arthralgia(5thvacc): number analyzed (Participants) | 206 | 206 | 140 | 121 | 132 | 147
  Grade3Arthralgia(5thvacc) | 0 | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Number of Participants Reporting Any Serious AE (SAE), Medically Attended AEs (MAAEs), AEs Leading to Premature Withdrawal
Description: The number of participants reporting any SAE, possibly or probably related SAE(s), medically-attended AEs, AEs leading to premature withdrawal, AEs leading to death, AEs leading to hospitalization and AEs leading to dose reduction, interruption and delay in study vaccination during the entire study period is reported.
Time Frame: During the entire study period (Month 0 to Month 13)
Population: Analysis was done on all subjects in the Unsolicited Safety Set-all screened subjects who provided informed consent & provided demographic &/or other baseline screening measurements, regardless of the subject's randomization & vaccination status, received a subject ID, received a study vaccination and have post-vaccination unsolicited AE records.
Measure: Count of Participants; unit: Participants
Arm/Group | rMenB_0_2 Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group | ABCWY_0_2_6 Group
Number analyzed (Participants) | 221 | 228 | 151 | 129 | 147 | 157
Participants
  Any SAE(s) | 9 | 3 | 8 | 7 | 2 | 6
  Possibly or Probably Related SAE(s) | 0 | 1 | 1 | 0 | 0 | 0
  Medically Attended AE(s) | 103 | 97 | 68 | 57 | 67 | 79
  AE(s) leading to premature withdrawal | 2 | 6 | 4 | 2 | 1 | 3
  AE(s) leading to Death | 0 | 0 | 0 | 0 | 0 | 0
  AE(s) leading to Hospitalization | 9 | 1 | 7 | 6 | 1 | 6
  AE(s)leadingtodosereduction,interruption,vaccdelay | 8 | 8 | 7 | 2 | 4 | 5

ADVERSE EVENTS:
Time Frame: Solicited AEs were collected from day 1 to day 7, Unsolicited AEs were collected from day 1 to day 30, SAEs were collected throughout the entire study period.
Description: Solicited AEs were collected by Systematic assessment; Unsolicited AEs were collected by non-systematic assessment.
Arm/Group | rMenB_0_2 Group | ABCWY_ 0_2 Group | ABCWY_0_1 Group | ABCWY_0_6 Group | ABCWY_0_11 Group | ABCWY_0_2_6 Group
All-Cause Mortality (participants affected / at risk) | 0/228 | 0/231 | 0/155 | 0/134 | 0/151 | 0/159
Serious Adverse Events (participants affected / at risk) | 9/228 | 3/231 | 8/155 | 7/134 | 2/151 | 6/159
Other Adverse Events (participants affected / at risk) | 226/228 | 229/231 | 153/155 | 131/134 | 151/151 | 158/159
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | rMenB_0_2 Group (N=228) | ABCWY_ 0_2 Group (N=231) | ABCWY_0_1 Group (N=155) | ABCWY_0_6 Group (N=134) | ABCWY_0_11 Group (N=151) | ABCWY_0_2_6 Group (N=159)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0 | 0 | 0 | 0
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 1
Abdominal migraine (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0
Crohn's disease (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0
Chest pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 0 | 1 | 0 | 0
Appendicitis (Infections and infestations) | 1 | 0 | 2 | 0 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Infectious mononucleosis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Pelvic inflammatory disease (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 1
Peritonsillar abscess (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0
Carbon monoxide poisoning (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1
Failure to thrive (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0
Obesity (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1
Type 1 diabetes mellitus (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Connective tissue disorder (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0
Torticollis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1
Fibroadenoma of breast (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 1 | 0
Abortion incomplete (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0
Mental disorder (Psychiatric disorders) | 0 | 0 | 0 | 1 | 0 | 0
Suicidal ideation (Psychiatric disorders) | 0 | 1 | 1 | 0 | 0 | 0
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0 | 0
Testicular torsion (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1
Tooth extraction (Surgical and medical procedures) | 0 | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | rMenB_0_2 Group (N=228) | ABCWY_ 0_2 Group (N=231) | ABCWY_0_1 Group (N=155) | ABCWY_0_6 Group (N=134) | ABCWY_0_11 Group (N=151) | ABCWY_0_2_6 Group (N=159)
Abdominal pain upper (Gastrointestinal disorders) | 16 | 9 | 6 | 5 | 9 | 9
Nausea (Gastrointestinal disorders) | 74 | 68 | 51 | 47 | 56 | 62
Chills (General disorders) | 80 | 76 | 61 | 40 | 62 | 70
Fatigue (General disorders) | 169 | 165 | 119 | 98 | 105 | 120
Injection site erythema (General disorders) | 131 | 131 | 80 | 80 | 89 | 97
Injection site induration (General disorders) | 110 | 98 | 67 | 53 | 70 | 85
Injection site pain (General disorders) | 221 | 225 | 148 | 129 | 148 | 154
Pyrexia (General disorders) | 27 | 27 | 20 | 13 | 25 | 26
Gastroenteritis (Infections and infestations) | 15 | 11 | 13 | 9 | 10 | 10
Nasopharyngitis (Infections and infestations) | 37 | 30 | 28 | 21 | 24 | 25
Pharyngitis (Infections and infestations) | 16 | 21 | 7 | 8 | 11 | 15
Respiratory tract infection (Injury, poisoning and procedural complications) | 15 | 12 | 10 | 5 | 6 | 10
Rhinitis (Infections and infestations) | 15 | 18 | 7 | 6 | 5 | 11
Tonsillitis (Infections and infestations) | 7 | 10 | 3 | 6 | 9 | 5
Upper respiratory tract infection (Infections and infestations) | 53 | 58 | 37 | 31 | 35 | 37
Decreased appetite (Metabolism and nutrition disorders) | 69 | 64 | 45 | 43 | 45 | 52
Arthralgia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 48 | 48 | 28 | 31 | 27 | 38
Myalgia (Musculoskeletal and connective tissue disorders) | 103 | 99 | 69 | 54 | 65 | 81
Headache (Nervous system disorders) | 165 | 149 | 114 | 93 | 110 | 117
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 5 | 6 | 1 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 12 | 13 | 9 | 7 | 5 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.